CLINICAL TRIAL: NCT03000530
Title: A Phase 2, Two-Part (Open-Label Followed by Double-Blind) Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of SAGE-217 in the Treatment of Adult Subjects With Moderate to Severe Major Depressive Disorder
Brief Title: A Study to Evaluate SAGE-217 in Participants With Moderate to Severe Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 217-MDD-201
Record Dates: First submitted 2016-12-14; First posted 2016-12-22 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Major Depression
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — zuranolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A: SAGE-217 (Experimental): Participants received SAGE-217, 30 milligrams (mg), oral solution, once daily for 14 days, as tolerated.
  Interventions: Drug: SAGE-217
- Part B: Placebo (Placebo Comparator): Eligible participants received matching placebo capsules once daily for 14 days.
  Interventions: Drug: Placebo
- Part B: SAGE-217 (Experimental): Eligible participants received SAGE-217, 30 mg, oral capsules, once daily for 14 days.
  Interventions: Drug: SAGE-217

INTERVENTIONS:
Drug: SAGE-217
  Arms: Part A: SAGE-217; Part B: SAGE-217
Drug: Placebo
  Arms: Part B: Placebo

SUMMARY:
This is a two-part (open-label followed by double-blind) study evaluating the safety, tolerability, pharmacokinetics, and efficacy of SAGE-217 in 102 participants diagnosed with moderate to severe Major Depressive Disorder.

DETAILED DESCRIPTION:
Part A of the study is an open-label design with dosing of SAGE-217 for 14 days.

Part B of the study is a randomized, double-blind, parallel-group, placebo-controlled design. Eligible participants were randomized to SAGE-217 or placebo for 14 days.

This study was previously posted by Sage Therapeutics. In November 2023, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of Major Depressive Disorder that has been present for at least a 4-week period as diagnosed by Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I)

Exclusion Criteria:

* Participant has a history of suicide attempt
* Participant has a history of treatment-resistant depression, defined as persistent depressive symptoms despite treatment with adequate doses of antidepressants from two different classes for an adequate amount of time
* Participant has active psychosis
* Participant has a medical history of seizures
* Participant has a medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Sage Investigational Site, Garden Grove, California
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Lake Charles, Louisiana
  - Sage Investigational Site, Berlin, New Jersey
  - Sage Investigational Site, Dayton, Ohio
  - Sage Investigational Site, Austin, Texas
  - Sage Investigational Site, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Background] Gunduz-Bruce H, Silber C, Kaul I, Rothschild AJ, Riesenberg R, Sankoh AJ, Li H, Lasser R, Zorumski CF, Rubinow DR, Paul SM, Jonas J, Doherty JJ, Kanes SJ. Trial of SAGE-217 in Patients with Major Depressive Disorder. N Engl J Med. 2019 Sep 5;381(10):903-911. doi: 10.1056/NEJMoa1815981. PMID 31483961
- [Derived] Suthoff E, Kosinski M, Arnaud A, Hodgkins P, Gunduz-Bruce H, Lasser R, Silber C, Sankoh AJ, Li H, Werneburg B, Jonas J, Doherty J, Kanes SJ, Bonthapally V. Patient-reported health-related quality of life from a randomized, placebo-controlled phase 2 trial of zuranolone in adults with major depressive disorder. J Affect Disord. 2022 Jul 1;308:19-26. doi: 10.1016/j.jad.2022.03.068. Epub 2022 Apr 2. PMID 35378149
- See also: Related Info — http://www.sagerx.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Part A, 21 participants were screened; 13 received at least one dose of study drug. In Part B, 169 participants were screened; 89 received at least one dose of study drug.
Period: Overall Study
Arm/Group | Part A: SAGE-217 | Part B: Placebo | Part B: SAGE-217
Started | 13 | 44 | 45
Completed | 13 | 39 | 41
Not Completed | 0 | 5 | 4
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received at least one dose of the study drug.
Groups:
- Part A: SAGE-217: Participants received SAGE-217, 30 mg, oral solution, once daily for 14 days, as tolerated.
- Total: Total of all reporting groups
Arm/Group | Part A: SAGE-217 | Part B: Placebo | Part B: SAGE-217 | Total
Number analyzed (Participants) | 13 | 44 | 45 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (12.83) | 38.3 (12.15) | 49.1 (13.61) | 44.3 (13.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 30 | 25 | 64
  Male | 4 | 14 | 20 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 1
  Black or African American | 9 | 28 | 36 | 73
  White | 4 | 16 | 7 | 27
  Other | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 7 | 1 | 9
  Not Hispanic or Latino | 12 | 37 | 44 | 93
17-item Hamilton Rating Scale for Depression (HAM-D) Total Score - Part B [Mean (Standard Deviation); unit: score on a scale] — The HAM-D total score comprised a sum of 17 individual item scores. Items scored in a range of 0 to 2 included: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score could range from 0 to 52. Higher scores indicated a greater degree of depression. Population: The efficacy set included all participants who were randomized and received at least one dose of the double-blind study drug and had a baseline and at least 1 post-baseline efficacy evaluation in Part B.
  score on a scale
    number analyzed (Participants) | 0 | 44 | 45 | 89
    (all) |  | 25.7 (2.42) | 25.2 (2.58) | 25.5 (2.50)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) - Part A
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. A TEAE was defined as an adverse event with onset after the start of study drug, or any worsening of a pre-existing medical condition/adverse event with onset after the start of study drug and until 7 days after the last dose. The analysis was performed in participants included in Part A of the study.
Time Frame: Day 1 up to Day 21
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
percentage of participants | 92.3

2. Primary Outcome: Percentage of Participants With TEAEs, Graded by Severity - Part A
Description: Severity was assessed according to the following scale: mild (awareness of sign or symptom, but easily tolerated); moderate (discomfort sufficient to cause interference with normal activities); severe (incapacitating, with inability to perform normal activities). The analysis was performed in participants included in Part A of the study.
Time Frame: Day 1 up to Day 21
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
percentage of participants
  Mild | 69.2
  Moderate | 23.1
  Severe | 0

3. Primary Outcome: Change From Baseline in Basophils - Part A
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, hematocrit, hemoglobin, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets, erythrocytes, reticulocytes and leukocytes. The analysis was performed in participants included in Part A of the study. ET = Early Termination.
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (10^9 cells/L)
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
10^9 cells per liter (10^9 cells/L)
  Baseline | 0.032 (0.0286)
  Change from Baseline at Day 8 | -0.002 (0.0388)
  Change from Baseline at Day 15/ET | 0.005 (0.0445)
  Change from Baseline at Follow-up Day 21 | -0.003 (0.0273)
  Change from Baseline at Follow-up Day 28 | -0.007 (0.0244)

4. Primary Outcome: Change From Baseline in Basophils to Leukocytes Ratio [Percentage (%)] - Part A
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, hematocrit, hemoglobin, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets, erythrocytes, reticulocytes and leukocytes. The analysis was performed in participants included in Part A of the study. ET = Early Termination. The blood cell differential (ratio) data are presented as International System (SI) unit, percentage (%).
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
percentage
  Baseline | 0.56 (0.323)
  Change from Baseline at Day 8 | 0.38 (1.308)
  Change from Baseline at Day 15/ET | 0.13 (0.681)
  Change from Baseline at Follow-up Day 21 | 0.02 (0.453)
  Change from Baseline at Follow-up Day 28 | -0.05 (0.310)

5. Primary Outcome: Change From Baseline in Eosinophils - Part A
Description: as for outcome 3
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
10^9 cells/L
  Baseline | 0.155 (0.0990)
  Change from Baseline at Day 8 | 0.031 (0.0749)
  Change from Baseline at Day 15/ET | 0.044 (0.0906)
  Change from Baseline at Follow-up Day 21 | 0.018 (0.0796)
  Change from Baseline at Follow-up Day 28 | 0.011 (0.1030)

6. Primary Outcome: Change From Baseline in Eosinophils to Leukocytes Ratio (%) - Part A
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, hematocrit, hemoglobin, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets, erythrocytes, reticulocytes and leukocytes. The analysis was performed in participants included in Part A of the study. ET = Early Termination. The blood cell differential (ratio) data are presented as SI unit, percentage (%).
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
percentage
  Baseline | 2.20 (1.155)
  Change from Baseline at Day 8 | 0.68 (1.174)
  Change from Baseline at Day 15/ET | 0.98 (1.438)
  Change from Baseline at Follow-up Day 21 | 0.52 (1.382)
  Change from Baseline at Follow-up Day 28 | 0.43 (1.865)

7. Primary Outcome: Change From Baseline in Hematocrit - Part A
Description: as for outcome 3
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: fraction of one
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
fraction of one
  Baseline | 0.419 (0.0341)
  Change from Baseline at Day 8 | 0.001 (0.0123)
  Change from Baseline at Day 15/ET | -0.006 (0.0203)
  Change from Baseline at Follow-up Day 21 | -0.020 (0.0239)
  Change from Baseline at Follow-up Day 28 | -0.017 (0.0256)

8. Primary Outcome: Change From Baseline in Hemoglobin - Part A
Description: as for outcome 3
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
grams per liter (g/L)
  Baseline | 136.7 (11.28)
  Change from Baseline at Day 8 | 0.2 (4.30)
  Change from Baseline at Day 15/ET | -2.4 (5.25)
  Change from Baseline at Follow-up Day 21 | -5.7 (5.79)
  Change from Baseline at Follow-up Day 28 | -4.8 (6.21)

9. Primary Outcome: Change From Baseline in Lymphocytes - Part A
Description: as for outcome 3
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
10^9 cells/L
  Baseline | 2.356 (0.4184)
  Change from Baseline at Day 8 | -0.302 (0.3742)
  Change from Baseline at Day 15/ET | -0.339 (0.4330)
  Change from Baseline at Follow-up Day 21 | -0.260 (0.4550)
  Change from Baseline at Follow-up Day 28 | -0.204 (0.3183)

10. Primary Outcome: Change From Baseline in Lymphocytes to Leukocytes Ratio (%) - Part A
Description: as for outcome 6
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
percentage
  Baseline | 34.89 (9.321)
  Change from Baseline at Day 8 | -1.75 (4.741)
  Change from Baseline at Day 15/ET | -1.25 (7.573)
  Change from Baseline at Follow-up Day 21 | -1.11 (5.716)
  Change from Baseline at Follow-up Day 28 | -0.62 (7.047)

11. Primary Outcome: Change From Baseline in Monocytes - Part A
Description: as for outcome 3
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
10^9 cells/L
  Baseline | 0.485 (0.1785)
  Change from Baseline at Day 8 | -0.042 (0.1673)
  Change from Baseline at Day 15/ET | -0.074 (0.1373)
  Change from Baseline at Follow-up Day 21 | -0.090 (0.1513)
  Change from Baseline at Follow-up Day 28 | -0.103 (0.1369)

12. Primary Outcome: Change From Baseline in Monocytes to Leukocytes Ratio (%) - Part A
Description: as for outcome 6
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
percentage
  Baseline | 6.72 (1.263)
  Change from Baseline at Day 8 | 0.35 (1.805)
  Change from Baseline at Day 15/ET | -0.03 (1.625)
  Change from Baseline at Follow-up Day 21 | -0.67 (2.364)
  Change from Baseline at Follow-up Day 28 | -0.82 (2.403)

13. Primary Outcome: Change From Baseline in Neutrophils - Part A
Description: as for outcome 3
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
10^9 cells/L
  Baseline | 4.126 (1.7922)
  Change from Baseline at Day 8 | -0.485 (1.0690)
  Change from Baseline at Day 15/ET | -0.528 (1.1266)
  Change from Baseline at Follow-up Day 21 | -0.411 (1.1296)
  Change from Baseline at Follow-up Day 28 | -0.190 (1.2929)

14. Primary Outcome: Change From Baseline in Neutrophils to Leukocytes Ratio (%) - Part A
Description: as for outcome 6
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
percentage
  Baseline | 55.63 (8.925)
  Change from Baseline at Day 8 | 0.76 (5.123)
  Change from Baseline at Day 15/ET | 0.16 (8.428)
  Change from Baseline at Follow-up Day 21 | 1.23 (7.037)
  Change from Baseline at Follow-up Day 28 | 1.06 (8.908)

15. Primary Outcome: Change From Baseline in Platelets - Part A
Description: as for outcome 3
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
10^9 cells/L
  Baseline | 265.5 (50.99)
  Change from Baseline at Day 8 | -13.4 (26.77)
  Change from Baseline at Day 15/ET | -7.8 (25.00)
  Change from Baseline at Follow-up Day 21 | 8.8 (19.68)
  Change from Baseline at Follow-up Day 28 | -9.9 (34.29)

16. Primary Outcome: Change From Baseline in Erythrocytes - Part A
Description: as for outcome 3
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (10^12 cells/L)
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
10^12 cells per liter (10^12 cells/L)
  Baseline | 4.661 (0.4521)
  Change from Baseline at Day 8 | 0.021 (0.1406)
  Change from Baseline at Day 15/ET | -0.050 (0.1920)
  Change from Baseline at Follow-up Day 21 | -0.198 (0.2302)
  Change from Baseline at Follow-up Day 28 | -0.164 (0.2382)

17. Primary Outcome: Change From Baseline in Reticulocytes - Part A
Description: as for outcome 3
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
10^9 cells/L
  Baseline | 51.926 (21.8233)
  Change from Baseline at Day 8 | -3.694 (22.4664)
  Change from Baseline at Day 15/ET | -6.163 (24.9724)
  Change from Baseline at Follow-up Day 21 | 6.174 (27.1013)
  Change from Baseline at Follow-up Day 28 | 13.012 (24.3634)

18. Primary Outcome: Change From Baseline in Leukocytes - Part A
Description: as for outcome 3
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
10^9 cells/L
  Baseline | 7.16 (2.098)
  Change from Baseline at Day 8 | -0.82 (1.446)
  Change from Baseline at Day 15/ET | -0.91 (1.388)
  Change from Baseline at Follow-up Day 21 | -0.75 (1.331)
  Change from Baseline at Follow-up Day 28 | -0.49 (1.387)

19. Primary Outcome: Change From Baseline in Albumin - Part A
Description: Clinical chemistry measures included albumin, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, bilirubin, chloride, carbon dioxide, creatinine, potassium, protein, sodium, and urea nitrogen. The analysis was performed in participants included in Part A of the study. ET = Early Termination.
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
g/L
  Baseline | 42.8 (2.82)
  Change from Baseline at Day 8 | -1.5 (2.07)
  Change from Baseline at Day 15/ET | -1.0 (2.45)
  Change from Baseline at Follow-up Day 21 | -1.5 (2.57)
  Change from Baseline at Follow-up Day 28 | -0.8 (2.34)

20. Primary Outcome: Change From Baseline in Alkaline Phosphatase - Part A
Description: as for outcome 19
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 10
units per liter (U/L)
  Baseline | 84.3 (43.15)
  Change from Baseline at Day 8 | 6.1 (20.73)
  Change from Baseline at Day 15/ET | 16.5 (30.62)
  Change from Baseline at Follow-up Day 21 | 2.3 (9.93)
  Change from Baseline at Follow-up Day 28 | 2.5 (10.34)

21. Primary Outcome: Change From Baseline in Alanine Aminotransferase - Part A
Description: as for outcome 19
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
U/L
  Baseline | 18.8 (10.85)
  Change from Baseline at Day 8 | 8.8 (11.31)
  Change from Baseline at Day 15/ET | 11.0 (21.63)
  Change from Baseline at Follow-up Day 21 | 2.8 (7.73)
  Change from Baseline at Follow-up Day 28 | -1.7 (9.39)

22. Primary Outcome: Change From Baseline in Aspartate Aminotransferase - Part A
Description: as for outcome 19
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
U/L
  Baseline | 18.7 (8.07)
  Change from Baseline at Day 8 | 3.7 (8.63)
  Change from Baseline at Day 15/ET | 5.7 (17.50)
  Change from Baseline at Follow-up Day 21 | 0.0 (7.59)
  Change from Baseline at Follow-up Day 28 | 0.5 (12.60)

23. Primary Outcome: Change From Baseline in Bilirubin - Part A
Description: as for outcome 19
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: micro-moles per liter (umol/L)
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
micro-moles per liter (umol/L)
  Baseline | 8.945 (4.5860)
  Change from Baseline at Day 8 | -1.052 (2.5687)
  Change from Baseline at Day 15/ET | -1.973 (2.9491)
  Change from Baseline at Follow-up Day 21 | -1.842 (3.7243)
  Change from Baseline at Follow-up Day 28 | -1.184 (2.7382)

24. Primary Outcome: Change From Baseline in Chloride - Part A
Description: as for outcome 19
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: milli-moles per liter (mmol/L)
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
milli-moles per liter (mmol/L)
  Baseline | 102.9 (3.07)
  Change from Baseline at Day 8 | 1.2 (2.55)
  Change from Baseline at Day 15/ET | 1.5 (2.96)
  Change from Baseline at Follow-up Day 21 | 1.3 (1.97)
  Change from Baseline at Follow-up Day 28 | 1.1 (2.10)

25. Primary Outcome: Change From Baseline in Carbon Dioxide - Part A
Description: as for outcome 19
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
mmol/L
  Baseline | 26.4 (2.50)
  Change from Baseline at Day 8 | -1.0 (2.35)
  Change from Baseline at Day 15/ET | -0.8 (1.63)
  Change from Baseline at Follow-up Day 21 | 0.0 (2.24)
  Change from Baseline at Follow-up Day 28 | -0.5 (1.56)

26. Primary Outcome: Change From Baseline in Creatinine - Part A
Description: as for outcome 19
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
umol/L
  Baseline | 73.848 (18.2228)
  Change from Baseline at Day 8 | -0.748 (6.7791)
  Change from Baseline at Day 15/ET | 0.136 (8.4394)
  Change from Baseline at Follow-up Day 21 | 0.952 (9.4279)
  Change from Baseline at Follow-up Day 28 | 0.816 (7.6084)

27. Primary Outcome: Change From Baseline in Potassium - Part A
Description: as for outcome 19
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
mmol/L
  Baseline | 4.25 (0.273)
  Change from Baseline at Day 8 | 0.12 (0.365)
  Change from Baseline at Day 15/ET | 0.02 (0.349)
  Change from Baseline at Follow-up Day 21 | -0.04 (0.423)
  Change from Baseline at Follow-up Day 28 | -0.10 (0.416)

28. Primary Outcome: Change From Baseline in Protein - Part A
Description: as for outcome 19
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
g/L
  Baseline | 71.8 (3.59)
  Change from Baseline at Day 8 | -0.6 (5.36)
  Change from Baseline at Day 15/ET | -0.2 (4.85)
  Change from Baseline at Follow-up Day 21 | -2.5 (4.33)
  Change from Baseline at Follow-up Day 28 | -0.1 (3.57)

29. Primary Outcome: Change From Baseline in Sodium - Part A
Description: as for outcome 19
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
mmol/L
  Baseline | 138.5 (2.18)
  Change from Baseline at Day 8 | -0.2 (2.05)
  Change from Baseline at Day 15/ET | -0.1 (2.43)
  Change from Baseline at Follow-up Day 21 | 0.5 (2.76)
  Change from Baseline at Follow-up Day 28 | 0.5 (2.90)

30. Primary Outcome: Change From Baseline in Urea Nitrogen - Part A
Description: as for outcome 19
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
mmol/L
  Baseline | 4.888 (1.4234)
  Change from Baseline at Day 8 | -0.275 (1.6435)
  Change from Baseline at Day 15/ET | -0.412 (1.4563)
  Change from Baseline at Follow-up Day 21 | -0.357 (0.9885)
  Change from Baseline at Follow-up Day 28 | -0.741 (1.3552)

31. Primary Outcome: Change From Baseline in Activated Partial Thromboplastin Time - Part A
Description: Coagulation measures included activated partial thromboplastin time, prothrombin international normalized ratio, and prothrombin time. The analysis was performed in participants included in Part A of the study. ET = Early Termination.
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Median (Full Range); unit: seconds
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
seconds
  Baseline | 28.00 [24.5 to 33.0]
  Change from Baseline at Day 8 | 1.00 [-1.0 to 171.0]
  Change from Baseline at Day 15/ET | 1.20 [-2.0 to 3.0]
  Change from Baseline at Follow-up Day 21 | 0.70 [-2.0 to 4.0]
  Change from Baseline at Follow-up Day 28 | 1.00 [-2.0 to 4.0]

32. Primary Outcome: Change From Baseline in Prothrombin International Normalized Ratio (%) - Part A
Description: Coagulation measures included activated partial thromboplastin time, prothrombin international normalized ratio, and prothrombin time. The analysis was performed in participants included in Part A of the study. ET = Early Termination. The data for prothrombin international normalized ratio are presented as SI unit, percentage (%).
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
percentage
  Baseline | 1.02 (0.055)
  Change from Baseline at Day 8 | 0.04 (0.087)
  Change from Baseline at Day 15/ET | -0.04 (0.051)
  Change from Baseline at Follow-up Day 21 | -0.01 (0.049)
  Change from Baseline at Follow-up Day 28 | -0.02 (0.038)

33. Primary Outcome: Change From Baseline in Prothrombin Time - Part A
Description: as for outcome 31
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Median (Full Range); unit: seconds
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
seconds
  Baseline | 10.50 [10.1 to 13.4]
  Change from Baseline at Day 8 | 0.10 [-0.4 to 3.1]
  Change from Baseline at Day 15/ET | -0.40 [-0.9 to 0.5]
  Change from Baseline at Follow-up Day 21 | -0.10 [-1.0 to 1.3]
  Change from Baseline at Follow-up Day 28 | 0.00 [-0.6 to 0.6]

34. Primary Outcome: Change From Baseline in pH - Part A
Description: Urinalysis measures included pH and specific gravity. The analysis was performed in participants included in Part A of the study. ET = Early Termination.
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
pH
  Baseline | 6.46 (0.803)
  Change from Baseline at Day 8 | -0.15 (1.049)
  Change from Baseline at Day 15/ET | -0.35 (0.826)
  Change from Baseline at Follow-up Day 21 | -0.31 (1.407)
  Change from Baseline at Follow-up Day 28 | -0.19 (1.300)

35. Primary Outcome: Change From Baseline in Specific Gravity - Part A
Description: as for outcome 34
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
ratio
  Baseline | 1.014 (0.0083)
  Change from Baseline at Day 8 | 0.001 (0.0075)
  Change from Baseline at Day 15/ET | 0.000 (0.0066)
  Change from Baseline at Follow-up Day 21 | 0.003 (0.0084)
  Change from Baseline at Follow-up Day 28 | -0.001 (0.0076)

36. Primary Outcome: Change From Baseline (CFB) in Supine Systolic Blood Pressure - Part A
Description: Vital signs measures included supine systolic blood pressure, supine diastolic blood pressure, standing systolic blood pressure, standing diastolic blood pressure, heart rate, respiratory rate, oral temperature, and oxygen saturation. The analysis was performed in participants included in Part A of the study. H = Hour(s). ET = Early Termination.
Time Frame: Baseline, Day 1 (0.25, 0.5, 1, 2, 12 hours postdose), Days 2, 3, 4, 5, 6 and 7 (predose, 0.25, 0.5, 1, 2, 12 hours postdose), Days 8, 9, 10, 11, 12, 13 and 14 (predose, 1 hour postdose), Day 15/ET, follow-up Day 21, follow-up Day 28
Population: The safety set included all participants who received at least one dose of the study drug. Number analyzed: Number of participants in the safety set with a non-missing value at both baseline and the visit.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
millimeter of mercury (mmHg)
  Baseline | 122.8 (15.92)
  CFB at Day 1: 0.25 H Postdose | -1.7 (10.82)
  CFB at Day 1: 0.5 H Postdose | -4.2 (9.50)
  CFB at Day 1: 1 H Postdose | -2.4 (13.88)
  CFB at Day 1: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 1: 2 H Postdose | -4.9 (13.47)
  CFB at Day 1: 12 H Postdose | -0.8 (12.12)
  CFB at Day 2: Predose | -0.8 (17.66)
  CFB at Day 2: 0.25 H Postdose | 8.2 (17.46)
  CFB at Day 2: 0.5 H Postdose | 0.8 (16.21)
  CFB at Day 2: 1 H Postdose | 2.3 (16.65)
  CFB at Day 2: 2 H Postdose | -4.7 (13.88)
  CFB at Day 2: 12 H Postdose | -0.5 (12.01)
  CFB at Day 3: Predose | -2.1 (14.33)
  CFB at Day 3: 0.25 H Postdose | 5.8 (15.21)
  CFB at Day 3: 0.5 H Postdose | 0.5 (17.08)
  CFB at Day 3: 1 H Postdose | 2.5 (13.51)
  CFB at Day 3: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 3: 2 H Postdose | -0.8 (16.49)
  CFB at Day 3: 12 H Postdose | 1.7 (12.98)
  CFB at Day 4: Predose | -0.5 (17.70)
  CFB at Day 4: 0.25 H Postdose | -0.4 (15.23)
  CFB at Day 4: 0.5 H Postdose | 1.8 (18.69)
  CFB at Day 4: 1 H Postdose | -0.4 (19.35)
  CFB at Day 4: 2 H Postdose: number analyzed (Participants) | 12
  CFB at Day 4: 2 H Postdose | -3.4 (13.58)
  CFB at Day 4: 12 H Postdose | -2.7 (18.63)
  CFB at Day 5: Predose | -0.1 (20.01)
  CFB at Day 5: 0.25 H Postdose | 3.1 (18.18)
  CFB at Day 5: 0.5 H Postdose | 0.3 (16.94)
  CFB at Day 5: 1 H Postdose | -4.8 (20.99)
  CFB at Day 5: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 5: 2 H Postdose | -2.9 (16.11)
  CFB at Day 5: 12 H Postdose | -1.5 (15.90)
  CFB at Day 6: Predose | -0.2 (15.95)
  CFB at Day 6: 0.25 H Postdose | -0.2 (17.21)
  CFB at Day 6: 0.5 H Postdose | 1.8 (14.62)
  CFB at Day 6: 1 H Postdose | 0.9 (15.86)
  CFB at Day 6: 2 H Postdose | -3.5 (16.79)
  CFB at Day 6: 12 H Postdose | -1.9 (22.35)
  CFB at Day 7: Predose | -1.2 (21.17)
  CFB at Day 7: 0.25 H Postdose | 4.0 (16.40)
  CFB at Day 7: 0.5 H Postdose | 1.5 (17.47)
  CFB at Day 7: 1 H Postdose | -3.2 (19.95)
  CFB at Day 7: 2 H Postdose | 0.3 (13.45)
  CFB at Day 7: 12 H Postdose | -4.3 (13.04)
  CFB at Day 8: Predose | 4.3 (17.77)
  CFB at Day 8: 1 H Postdose | -4.5 (13.15)
  CFB at Day 9: Predose | 9.4 (15.86)
  CFB at Day 9: 1 H Postdose | 3.3 (15.54)
  CFB at Day 10: Predose | 8.4 (14.93)
  CFB at Day 10: 1 H Postdose | 2.4 (14.19)
  CFB at Day 11: Predose: number analyzed (Participants) | 12
  CFB at Day 11: Predose | 8.8 (19.16)
  CFB at Day 11: 1 H Postdose: number analyzed (Participants) | 12
  CFB at Day 11: 1 H Postdose | -1.7 (14.26)
  CFB at Day 12: Predose | 7.4 (16.59)
  CFB at Day 12: 1 H Postdose | -0.2 (18.93)
  CFB at Day 13: Predose | 3.2 (19.62)
  CFB at Day 13: 1 H Postdose: number analyzed (Participants) | 12
  CFB at Day 13: 1 H Postdose | 1.3 (16.31)
  CFB at Day 14: Predose | -3.8 (18.20)
  CFB at Day 14: 1 H Postdose | -3.9 (15.01)
  CFB at Day 15/ET | 3.8 (17.10)
  CFB at Follow-up Day 21 | 3.9 (10.84)
  CFB at Follow-up Day 28 | 7.3 (15.19)

37. Primary Outcome: Change From Baseline (CFB) in Supine Diastolic Blood Pressure - Part A
Description: as for outcome 36
Time Frame: as for outcome 36
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
mmHg
  Baseline | 79.4 (8.84)
  CFB at Day 1: 0.25 H Postdose | -1.1 (5.50)
  CFB at Day 1: 0.5 H Postdose | -1.6 (6.27)
  CFB at Day 1: 1 H Postdose | -2.0 (7.51)
  CFB at Day 1: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 1: 2 H Postdose | -5.2 (11.69)
  CFB at Day 1: 12 H Postdose | 1.3 (7.94)
  CFB at Day 2: Predose | -3.5 (9.40)
  CFB at Day 2: 0.25 H Postdose | -0.2 (8.36)
  CFB at Day 2: 0.5 H Postdose | -2.4 (7.84)
  CFB at Day 2: 1 H Postdose | -2.5 (10.52)
  CFB at Day 2: 2 H Postdose | -5.4 (11.14)
  CFB at Day 2: 12 H Postdose | -2.4 (7.94)
  CFB at Day 3: Predose | 0.3 (6.94)
  CFB at Day 3: 0.25 H Postdose | 1.9 (10.33)
  CFB at Day 3: 0.5 H Postdose | 0.2 (9.12)
  CFB at Day 3: 1 H Postdose | -0.2 (9.13)
  CFB at Day 3: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 3: 2 H Postdose | -3.9 (10.21)
  CFB at Day 3: 12 H Postdose | 0.0 (9.64)
  CFB at Day 4: Predose | -0.8 (10.94)
  CFB at Day 4: 0.25 H Postdose | -1.1 (12.13)
  CFB at Day 4: 0.5 H Postdose | 0.1 (14.80)
  CFB at Day 4: 1 H Postdose | -3.5 (12.03)
  CFB at Day 4: 2 H Postdose: number analyzed (Participants) | 12
  CFB at Day 4: 2 H Postdose | -2.3 (10.27)
  CFB at Day 4: 12 H Postdose | -1.1 (13.51)
  CFB at Day 5: Predose | -1.3 (13.28)
  CFB at Day 5: 0.25 H Postdose | -1.5 (11.49)
  CFB at Day 5: 0.5 H Postdose | -1.3 (12.14)
  CFB at Day 5: 1 H Postdose | -6.0 (12.64)
  CFB at Day 5: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 5: 2 H Postdose | -4.3 (12.63)
  CFB at Day 5: 12 H Postdose | -1.1 (10.16)
  CFB at Day 6: Predose | -2.6 (12.05)
  CFB at Day 6: 0.25 H Postdose | -0.8 (10.38)
  CFB at Day 6: 0.5 H Postdose | 1.8 (10.30)
  CFB at Day 6: 1 H Postdose | 0.8 (11.96)
  CFB at Day 6: 2 H Postdose | -0.8 (13.04)
  CFB at Day 6: 12 H Postdose | -2.5 (14.08)
  CFB at Day 7: Predose | 2.2 (13.53)
  CFB at Day 7: 0.25 H Postdose | 2.0 (11.31)
  CFB at Day 7: 0.5 H Postdose | 0.2 (10.39)
  CFB at Day 7: 1 H Postdose | -0.2 (12.87)
  CFB at Day 7: 2 H Postdose | -1.8 (9.16)
  CFB at Day 7: 12 H Postdose | -2.5 (8.27)
  CFB at Day 8: Predose | 2.3 (11.27)
  CFB at Day 8: 1 H Postdose | -2.9 (9.28)
  CFB at Day 9: Predose | 3.2 (11.91)
  CFB at Day 9: 1 H Postdose | 0.5 (11.72)
  CFB at Day 10: Predose | 1.6 (10.02)
  CFB at Day 10: 1 H Postdose | -3.7 (9.77)
  CFB at Day 11: Predose: number analyzed (Participants) | 12
  CFB at Day 11: Predose | 5.2 (10.54)
  CFB at Day 11: 1 H Postdose: number analyzed (Participants) | 12
  CFB at Day 11: 1 H Postdose | 0.0 (9.41)
  CFB at Day 12: Predose | 0.4 (8.87)
  CFB at Day 12: 1 H Postdose | 2.1 (12.11)
  CFB at Day 13: Predose | 3.2 (9.86)
  CFB at Day 13: 1 H Postdose: number analyzed (Participants) | 12
  CFB at Day 13: 1 H Postdose | 3.7 (8.86)
  CFB at Day 14: Predose | -1.3 (10.16)
  CFB at Day 14: 1 H Postdose | -0.2 (9.08)
  CFB at Day 15/ET | -0.7 (8.73)
  CFB at Follow-up Day 21 | 3.1 (10.64)
  CFB at Follow-up Day 28 | 1.8 (11.26)

38. Primary Outcome: Change From Baseline (CFB) in Standing Systolic Blood Pressure - Part A
Description: as for outcome 36
Time Frame: as for outcome 36
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
mmHg
  Baseline | 126.8 (15.09)
  CFB at Day 1: 0.25 H Postdose | -0.1 (9.67)
  CFB at Day 1: 0.5 H Postdose | -3.8 (8.60)
  CFB at Day 1: 1 H Postdose | -6.5 (10.94)
  CFB at Day 1: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 1: 2 H Postdose | -3.9 (8.90)
  CFB at Day 1: 12 H Postdose | -4.2 (10.40)
  CFB at Day 2: Predose | -3.5 (11.74)
  CFB at Day 2: 0.25 H Postdose | -0.9 (15.14)
  CFB at Day 2: 0.5 H Postdose | -1.2 (11.29)
  CFB at Day 2: 1 H Postdose | -3.8 (13.64)
  CFB at Day 2: 2 H Postdose | -3.2 (14.52)
  CFB at Day 2: 12 H Postdose | -1.7 (13.68)
  CFB at Day 3: Predose | -0.5 (9.57)
  CFB at Day 3: 0.25 H Postdose | -0.4 (12.39)
  CFB at Day 3: 0.5 H Postdose | -1.2 (15.23)
  CFB at Day 3: 1 H Postdose | -0.6 (15.80)
  CFB at Day 3: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 3: 2 H Postdose | 3.3 (16.41)
  CFB at Day 3: 12 H Postdose | -1.0 (15.56)
  CFB at Day 4: Predose | -1.1 (15.94)
  CFB at Day 4: 0.25 H Postdose | 0.4 (13.26)
  CFB at Day 4: 0.5 H Postdose | -0.8 (13.55)
  CFB at Day 4: 1 H Postdose | -0.8 (14.81)
  CFB at Day 4: 2 H Postdose: number analyzed (Participants) | 12
  CFB at Day 4: 2 H Postdose | -5.8 (13.50)
  CFB at Day 4: 12 H Postdose | -7.1 (20.47)
  CFB at Day 5: Predose | -3.8 (16.67)
  CFB at Day 5: 0.25 H Postdose | -1.9 (16.51)
  CFB at Day 5: 0.5 H Postdose | -7.0 (15.51)
  CFB at Day 5: 1 H Postdose | -7.4 (13.74)
  CFB at Day 5: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 5: 2 H Postdose | -4.4 (10.26)
  CFB at Day 5: 12 H Postdose | -7.2 (17.29)
  CFB at Day 6: Predose | -3.7 (16.20)
  CFB at Day 6: 0.25 H Postdose | 1.2 (12.65)
  CFB at Day 6: 0.5 H Postdose | 0.3 (11.73)
  CFB at Day 6: 1 H Postdose | -3.2 (15.96)
  CFB at Day 6: 2 H Postdose | -7.1 (12.51)
  CFB at Day 6: 12 H Postdose | -5.6 (17.41)
  CFB at Day 7: Predose | -2.2 (21.07)
  CFB at Day 7: 0.25 H Postdose | -1.8 (12.25)
  CFB at Day 7: 0.5 H Postdose | -1.0 (19.46)
  CFB at Day 7: 1 H Postdose | -6.8 (12.60)
  CFB at Day 7: 2 H Postdose | -3.6 (11.35)
  CFB at Day 7: 12 H Postdose | -5.5 (14.01)
  CFB at Day 8: Predose | 1.5 (12.27)
  CFB at Day 8: 1 H Postdose | -6.6 (12.91)
  CFB at Day 9: Predose | -0.9 (12.05)
  CFB at Day 9: 1 H Postdose | -1.9 (15.18)
  CFB at Day 10: Predose | 2.8 (15.82)
  CFB at Day 10: 1 H Postdose | -4.0 (14.63)
  CFB at Day 11: Predose: number analyzed (Participants) | 12
  CFB at Day 11: Predose | 5.9 (13.63)
  CFB at Day 11: 1 H Postdose: number analyzed (Participants) | 12
  CFB at Day 11: 1 H Postdose | -4.9 (10.18)
  CFB at Day 12: Predose | 4.1 (19.31)
  CFB at Day 12: 1 H Postdose | -3.8 (19.88)
  CFB at Day 13: Predose | 0.5 (14.77)
  CFB at Day 13: 1 H Postdose: number analyzed (Participants) | 12
  CFB at Day 13: 1 H Postdose | 0.8 (13.04)
  CFB at Day 14: Predose | -0.8 (12.19)
  CFB at Day 14: 1 H Postdose | -8.9 (12.53)
  CFB at Day 15/ET | -1.4 (11.39)
  CFB at Follow-up Day 21 | 7.8 (14.23)
  CFB at Follow-up Day 28 | 3.8 (13.53)

39. Primary Outcome: Change From Baseline (CFB) in Standing Diastolic Blood Pressure - Part A
Description: as for outcome 36
Time Frame: as for outcome 36
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
mmHg
  Baseline | 83.9 (8.17)
  CFB at Day 1: 0.25 H Postdose | -0.2 (7.60)
  CFB at Day 1: 0.5 H Postdose | -1.5 (6.33)
  CFB at Day 1: 1 H Postdose | -1.8 (5.10)
  CFB at Day 1: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 1: 2 H Postdose | -1.5 (9.13)
  CFB at Day 1: 12 H Postdose | -3.5 (7.49)
  CFB at Day 2: Predose | -4.9 (5.41)
  CFB at Day 2: 0.25 H Postdose | -3.3 (9.53)
  CFB at Day 2: 0.5 H Postdose | -1.8 (7.46)
  CFB at Day 2: 1 H Postdose | -3.4 (9.90)
  CFB at Day 2: 2 H Postdose | -5.8 (9.63)
  CFB at Day 2: 12 H Postdose | -3.2 (13.06)
  CFB at Day 3: Predose | -4.2 (13.31)
  CFB at Day 3: 0.25 H Postdose | -3.6 (10.79)
  CFB at Day 3: 0.5 H Postdose | -1.9 (9.84)
  CFB at Day 3: 1 H Postdose | -0.8 (9.58)
  CFB at Day 3: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 3: 2 H Postdose | -2.2 (13.80)
  CFB at Day 3: 12 H Postdose | 0.7 (10.23)
  CFB at Day 4: Predose | -0.8 (13.05)
  CFB at Day 4: 0.25 H Postdose | -1.4 (10.91)
  CFB at Day 4: 0.5 H Postdose | -2.6 (11.00)
  CFB at Day 4: 1 H Postdose | -3.3 (9.02)
  CFB at Day 4: 2 H Postdose: number analyzed (Participants) | 12
  CFB at Day 4: 2 H Postdose | -2.9 (10.16)
  CFB at Day 4: 12 H Postdose | -2.6 (12.31)
  CFB at Day 5: Predose | -2.1 (10.54)
  CFB at Day 5: 0.25 H Postdose | -2.6 (11.99)
  CFB at Day 5: 0.5 H Postdose | -5.3 (10.71)
  CFB at Day 5: 1 H Postdose | -5.9 (13.51)
  CFB at Day 5: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 5: 2 H Postdose | -5.4 (13.26)
  CFB at Day 5: 12 H Postdose | -2.2 (12.98)
  CFB at Day 6: Predose | -2.2 (10.86)
  CFB at Day 6: 0.25 H Postdose | -0.9 (9.27)
  CFB at Day 6: 0.5 H Postdose | 1.2 (7.97)
  CFB at Day 6: 1 H Postdose | -1.8 (9.08)
  CFB at Day 6: 2 H Postdose | -2.6 (6.70)
  CFB at Day 6: 12 H Postdose | -4.5 (9.75)
  CFB at Day 7: Predose | -0.2 (14.31)
  CFB at Day 7: 0.25 H Postdose | 0.8 (9.86)
  CFB at Day 7: 0.5 H Postdose | -0.4 (12.76)
  CFB at Day 7: 1 H Postdose | -2.5 (11.33)
  CFB at Day 7: 2 H Postdose | -2.4 (7.97)
  CFB at Day 7: 12 H Postdose | -3.0 (8.23)
  CFB at Day 8: Predose | 1.3 (9.91)
  CFB at Day 8: 1 H Postdose | -4.5 (11.97)
  CFB at Day 9: Predose | -2.5 (10.83)
  CFB at Day 9: 1 H Postdose | -4.2 (10.61)
  CFB at Day 10: Predose | -2.0 (9.70)
  CFB at Day 10: 1 H Postdose | -3.7 (9.64)
  CFB at Day 11: Predose: number analyzed (Participants) | 12
  CFB at Day 11: Predose | 2.0 (9.03)
  CFB at Day 11: 1 H Postdose: number analyzed (Participants) | 12
  CFB at Day 11: 1 H Postdose | -7.1 (8.61)
  CFB at Day 12: Predose | -3.8 (10.40)
  CFB at Day 12: 1 H Postdose | -2.5 (10.62)
  CFB at Day 13: Predose | 0.5 (4.88)
  CFB at Day 13: 1 H Postdose: number analyzed (Participants) | 12
  CFB at Day 13: 1 H Postdose | 1.4 (7.08)
  CFB at Day 14: Predose | -0.7 (9.76)
  CFB at Day 14: 1 H Postdose | -3.2 (9.24)
  CFB at Day 15/ET | 0.5 (8.39)
  CFB at Follow-up Day 21 | 0.8 (10.64)
  CFB at Follow-up Day 28 | 1.7 (6.80)

40. Primary Outcome: Change From Baseline (CFB) in Heart Rate - Part A
Description: as for outcome 36
Time Frame: as for outcome 36
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: beats per minute (beats/min)
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
beats per minute (beats/min)
  Baseline | 80.0 (13.10)
  CFB at Day 1: 0.25 H Postdose | -2.7 (9.91)
  CFB at Day 1: 0.5 H Postdose | -5.9 (13.44)
  CFB at Day 1: 1 H Postdose | -4.6 (13.07)
  CFB at Day 1: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 1: 2 H Postdose | -2.6 (14.77)
  CFB at Day 1: 12 H Postdose | -2.2 (15.22)
  CFB at Day 2: Predose | -6.6 (14.66)
  CFB at Day 2: 0.25 H Postdose | -6.6 (13.64)
  CFB at Day 2: 0.5 H Postdose | -6.4 (12.96)
  CFB at Day 2: 1 H Postdose | -2.8 (16.75)
  CFB at Day 2: 2 H Postdose | -3.5 (13.97)
  CFB at Day 2: 12 H Postdose | -10.7 (14.68)
  CFB at Day 3: Predose | -4.8 (15.82)
  CFB at Day 3: 0.25 H Postdose | -6.1 (18.02)
  CFB at Day 3: 0.5 H Postdose | -6.1 (14.23)
  CFB at Day 3: 1 H Postdose | -1.2 (13.83)
  CFB at Day 3: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 3: 2 H Postdose | -1.4 (16.19)
  CFB at Day 3: 12 H Postdose | -8.2 (15.60)
  CFB at Day 4: Predose | -6.8 (15.33)
  CFB at Day 4: 0.25 H Postdose | -8.5 (15.58)
  CFB at Day 4: 0.5 H Postdose | -5.3 (14.09)
  CFB at Day 4: 1 H Postdose | -5.0 (15.46)
  CFB at Day 4: 2 H Postdose: number analyzed (Participants) | 12
  CFB at Day 4: 2 H Postdose | 0.7 (12.21)
  CFB at Day 4: 12 H Postdose | -5.2 (12.39)
  CFB at Day 5: Predose | -5.2 (12.39)
  CFB at Day 5: 0.25 H Postdose | -6.7 (16.93)
  CFB at Day 5: 0.5 H Postdose | -4.4 (16.11)
  CFB at Day 5: 1 H Postdose | -3.2 (13.57)
  CFB at Day 5: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 5: 2 H Postdose | -1.0 (13.21)
  CFB at Day 5: 12 H Postdose | -2.6 (14.71)
  CFB at Day 6: Predose | -2.2 (13.98)
  CFB at Day 6: 0.25 H Postdose | -4.8 (13.49)
  CFB at Day 6: 0.5 H Postdose | -4.8 (14.90)
  CFB at Day 6: 1 H Postdose | -0.5 (15.98)
  CFB at Day 6: 2 H Postdose | -3.5 (13.48)
  CFB at Day 6: 12 H Postdose | -5.8 (20.85)
  CFB at Day 7: Predose | -3.0 (20.13)
  CFB at Day 7: 0.25 H Postdose | -4.6 (16.86)
  CFB at Day 7: 0.5 H Postdose | -6.2 (15.53)
  CFB at Day 7: 1 H Postdose | -1.0 (16.64)
  CFB at Day 7: 2 H Postdose | -0.1 (16.12)
  CFB at Day 7: 12 H Postdose | -7.0 (18.16)
  CFB at Day 8: Predose | -2.1 (15.74)
  CFB at Day 8: 1 H Postdose | -1.0 (16.07)
  CFB at Day 9: Predose | -0.1 (15.18)
  CFB at Day 9: 1 H Postdose | 0.2 (18.44)
  CFB at Day 10: Predose | -1.8 (15.39)
  CFB at Day 10: 1 H Postdose | 0.7 (13.91)
  CFB at Day 11: Predose: number analyzed (Participants) | 12
  CFB at Day 11: Predose | 3.3 (12.80)
  CFB at Day 11: 1 H Postdose: number analyzed (Participants) | 12
  CFB at Day 11: 1 H Postdose | -5.2 (13.56)
  CFB at Day 12: Predose | 1.9 (10.30)
  CFB at Day 12: 1 H Postdose | -1.2 (16.61)
  CFB at Day 13: Predose | 0.2 (16.69)
  CFB at Day 13: 1 H Postdose: number analyzed (Participants) | 12
  CFB at Day 13: 1 H Postdose | 2.9 (13.76)
  CFB at Day 14: Predose | -3.7 (15.16)
  CFB at Day 14: 1 H Postdose | -2.2 (17.24)
  CFB at Day 15/ET | -3.5 (16.06)
  CFB at Follow-up Day 21 | -6.5 (17.66)
  CFB at Follow-up Day 28 | -6.8 (13.53)

41. Primary Outcome: Change From Baseline (CFB) in Respiratory Rate - Part A
Description: as for outcome 36
Time Frame: as for outcome 36
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: breaths per minute (breaths/min)
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
breaths per minute (breaths/min)
  Baseline | 16.9 (1.75)
  CFB at Day 1: 0.25 H Postdose | 0.5 (1.45)
  CFB at Day 1: 0.5 H Postdose | 0.5 (1.45)
  CFB at Day 1: 1 H Postdose | 0.3 (1.80)
  CFB at Day 1: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 1: 2 H Postdose | 0.4 (1.57)
  CFB at Day 1: 12 H Postdose | -0.1 (1.26)
  CFB at Day 2: Predose | 0.5 (1.56)
  CFB at Day 2: 0.25 H Postdose | 0.3 (2.10)
  CFB at Day 2: 0.5 H Postdose | -0.1 (1.66)
  CFB at Day 2: 1 H Postdose | -0.2 (1.72)
  CFB at Day 2: 2 H Postdose | -0.5 (1.66)
  CFB at Day 2: 12 H Postdose | -0.5 (1.71)
  CFB at Day 3: Predose | -0.4 (1.61)
  CFB at Day 3: 0.25 H Postdose | 0.4 (1.76)
  CFB at Day 3: 0.5 H Postdose | -0.3 (1.65)
  CFB at Day 3: 1 H Postdose | -0.2 (1.17)
  CFB at Day 3: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 3: 2 H Postdose | -0.7 (1.35)
  CFB at Day 3: 12 H Postdose | -0.1 (1.66)
  CFB at Day 4: Predose | 0.1 (1.55)
  CFB at Day 4: 0.25 H Postdose | 0.3 (1.55)
  CFB at Day 4: 0.5 H Postdose | 0.3 (1.60)
  CFB at Day 4: 1 H Postdose | 0.5 (1.20)
  CFB at Day 4: 2 H Postdose: number analyzed (Participants) | 12
  CFB at Day 4: 2 H Postdose | 0.3 (1.67)
  CFB at Day 4: 12 H Postdose | 0.4 (1.94)
  CFB at Day 5: Predose | 0.2 (1.57)
  CFB at Day 5: 0.25 H Postdose | 0.4 (1.39)
  CFB at Day 5: 0.5 H Postdose | 0.4 (1.50)
  CFB at Day 5: 1 H Postdose | 0.2 (1.64)
  CFB at Day 5: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 5: 2 H Postdose | -0.5 (1.75)
  CFB at Day 5: 12 H Postdose | -0.5 (2.99)
  CFB at Day 6: Predose | 0.2 (1.83)
  CFB at Day 6: 0.25 H Postdose | 0.2 (1.83)
  CFB at Day 6: 0.5 H Postdose | 0.1 (1.89)
  CFB at Day 6: 1 H Postdose | 0.1 (1.55)
  CFB at Day 6: 2 H Postdose | 0.1 (2.10)
  CFB at Day 6: 12 H Postdose | -0.1 (1.12)
  CFB at Day 7: Predose | 0.1 (1.55)
  CFB at Day 7: 0.25 H Postdose | 0.8 (1.99)
  CFB at Day 7: 0.5 H Postdose | 0.2 (0.83)
  CFB at Day 7: 1 H Postdose | 0.5 (1.85)
  CFB at Day 7: 2 H Postdose | -0.1 (2.02)
  CFB at Day 7: 12 H Postdose | -0.3 (2.53)
  CFB at Day 8: Predose | 1.2 (2.28)
  CFB at Day 8: 1 H Postdose | -0.3 (1.84)
  CFB at Day 9: Predose | 0.5 (2.18)
  CFB at Day 9: 1 H Postdose | 0.5 (2.67)
  CFB at Day 10: Predose | 0.6 (2.50)
  CFB at Day 10: 1 H Postdose | 0.0 (1.96)
  CFB at Day 11: Predose: number analyzed (Participants) | 12
  CFB at Day 11: Predose | 0.8 (1.95)
  CFB at Day 11: 1 H Postdose: number analyzed (Participants) | 12
  CFB at Day 11: 1 H Postdose | -0.2 (1.80)
  CFB at Day 12: Predose | 0.5 (1.85)
  CFB at Day 12: 1 H Postdose | 0.5 (2.54)
  CFB at Day 13: Predose | 0.3 (2.39)
  CFB at Day 13: 1 H Postdose: number analyzed (Participants) | 12
  CFB at Day 13: 1 H Postdose | 0.5 (1.00)
  CFB at Day 14: Predose | 0.3 (1.55)
  CFB at Day 14: 1 H Postdose | 0.0 (2.12)
  CFB at Day 15/ET | 0.1 (2.10)
  CFB at Follow-up Day 21 | 0.8 (1.92)
  CFB at Follow-up Day 28 | 0.3 (1.60)

42. Primary Outcome: Change From Baseline (CFB) in Oral Temperature - Part A
Description: as for outcome 36
Time Frame: as for outcome 36
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: degrees Celsius (degrees C)
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
degrees Celsius (degrees C)
  Baseline | 36.71 (0.278)
  CFB at Day 1: 0.25 H Postdose | -0.17 (0.457)
  CFB at Day 1: 0.5 H Postdose | 0.12 (0.302)
  CFB at Day 1: 1 H Postdose | 0.11 (0.468)
  CFB at Day 1: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 1: 2 H Postdose | 0.03 (0.438)
  CFB at Day 1: 12 H Postdose | -0.09 (0.433)
  CFB at Day 2: Predose | -0.05 (0.410)
  CFB at Day 2: 0.25 H Postdose | 0.04 (0.532)
  CFB at Day 2: 0.5 H Postdose | 0.00 (0.493)
  CFB at Day 2: 1 H Postdose | 0.20 (0.555)
  CFB at Day 2: 2 H Postdose | 0.01 (0.497)
  CFB at Day 2: 12 H Postdose | -0.05 (0.399)
  CFB at Day 3: Predose | 0.02 (0.580)
  CFB at Day 3: 0.25 H Postdose | -0.08 (0.563)
  CFB at Day 3: 0.5 H Postdose | -0.17 (0.497)
  CFB at Day 3: 1 H Postdose | -0.02 (0.597)
  CFB at Day 3: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 3: 2 H Postdose | -0.11 (0.459)
  CFB at Day 3: 12 H Postdose | -0.22 (0.389)
  CFB at Day 4: Predose | -0.05 (0.525)
  CFB at Day 4: 0.25 H Postdose | 0.00 (0.473)
  CFB at Day 4: 0.5 H Postdose | 0.26 (0.459)
  CFB at Day 4: 1 H Postdose | -0.05 (0.619)
  CFB at Day 4: 2 H Postdose: number analyzed (Participants) | 12
  CFB at Day 4: 2 H Postdose | -0.04 (0.373)
  CFB at Day 4: 12 H Postdose | -0.11 (0.373)
  CFB at Day 5: Predose | -0.06 (0.498)
  CFB at Day 5: 0.25 H Postdose | 0.01 (0.350)
  CFB at Day 5: 0.5 H Postdose | -0.05 (0.418)
  CFB at Day 5: 1 H Postdose | -0.08 (0.458)
  CFB at Day 5: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 5: 2 H Postdose | -0.18 (0.523)
  CFB at Day 5: 12 H Postdose | -0.09 (0.499)
  CFB at Day 6: Predose | 0.09 (0.560)
  CFB at Day 6: 0.25 H Postdose | 0.13 (0.512)
  CFB at Day 6: 0.5 H Postdose | -0.05 (0.405)
  CFB at Day 6: 1 H Postdose | 0.06 (0.601)
  CFB at Day 6: 2 H Postdose | -0.12 (0.526)
  CFB at Day 6: 12 H Postdose | -0.04 (0.566)
  CFB at Day 7: Predose | -0.11 (0.722)
  CFB at Day 7: 0.25 H Postdose | -0.11 (0.566)
  CFB at Day 7: 0.5 H Postdose | -0.08 (0.639)
  CFB at Day 7: 1 H Postdose | -0.14 (0.588)
  CFB at Day 7: 2 H Postdose | -0.02 (0.453)
  CFB at Day 7: 12 H Postdose: number analyzed (Participants) | 12
  CFB at Day 7: 12 H Postdose | -0.10 (0.534)
  CFB at Day 8: Predose | -0.02 (0.589)
  CFB at Day 8: 1 H Postdose | 0.02 (0.351)
  CFB at Day 9: Predose | -0.28 (0.675)
  CFB at Day 9: 1 H Postdose | -0.17 (0.609)
  CFB at Day 10: Predose | -0.20 (0.471)
  CFB at Day 10: 1 H Postdose | -0.23 (0.624)
  CFB at Day 11: Predose: number analyzed (Participants) | 12
  CFB at Day 11: Predose | 0.03 (0.483)
  CFB at Day 11: 1 H Postdose: number analyzed (Participants) | 12
  CFB at Day 11: 1 H Postdose | -0.28 (0.506)
  CFB at Day 12: Predose | -0.18 (0.504)
  CFB at Day 12: 1 H Postdose | -0.10 (0.512)
  CFB at Day 13: Predose | -0.12 (0.448)
  CFB at Day 13: 1 H Postdose: number analyzed (Participants) | 12
  CFB at Day 13: 1 H Postdose | -0.23 (0.342)
  CFB at Day 14: Predose | 0.01 (0.475)
  CFB at Day 14: 1 H Postdose | 0.05 (0.570)
  CFB at Day 15/ET | -0.05 (0.326)
  CFB at Follow-up Day 21 | -0.10 (0.372)
  CFB at Follow-up Day 28 | -0.12 (0.326)

43. Primary Outcome: Change From Baseline (CFB) in Oxygen Saturation - Part A
Description: Vital signs measures included supine systolic blood pressure, supine diastolic blood pressure, standing systolic blood pressure, standing diastolic blood pressure, heart rate, respiratory rate, oral temperature, and oxygen saturation. The analysis was performed in participants included in Part A of the study. H = Hour(s).
Time Frame: Baseline, Day 1 (0.25, 0.5, 1, 2, 12 hours postdose), Days 2, 3, 4, 5, 6 and 7 (predose, 0.25, 0.5, 1, 2, 12 hours postdose), Day 8 (predose, 1 hour postdose)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 12
percentage of oxygen saturation
  Baseline | 98.6 (1.08)
  CFB at Day 1: 0.25 H Postdose | 0.0 (1.65)
  CFB at Day 1: 0.5 H Postdose | -0.4 (2.02)
  CFB at Day 1: 1 H Postdose | 0.3 (1.22)
  CFB at Day 1: 2 H Postdose: number analyzed (Participants) | 10
  CFB at Day 1: 2 H Postdose | -0.3 (2.16)
  CFB at Day 1: 12 H Postdose | 0.3 (1.07)
  CFB at Day 2: Predose | -0.4 (1.62)
  CFB at Day 2: 0.25 H Postdose | -0.1 (1.83)
  CFB at Day 2: 0.5 H Postdose | -0.3 (1.44)
  CFB at Day 2: 1 H Postdose | 0.1 (1.62)
  CFB at Day 2: 2 H Postdose | -0.2 (1.34)
  CFB at Day 2: 12 H Postdose | -0.6 (1.62)
  CFB at Day 3: Predose | 0.3 (1.60)
  CFB at Day 3: 0.25 H Postdose | -0.9 (1.68)
  CFB at Day 3: 0.5 H Postdose | -1.3 (2.23)
  CFB at Day 3: 1 H Postdose | -0.3 (1.87)
  CFB at Day 3: 2 H Postdose: number analyzed (Participants) | 10
  CFB at Day 3: 2 H Postdose | 0.1 (1.37)
  CFB at Day 3: 12 H Postdose | -0.9 (1.68)
  CFB at Day 4: Predose | -1.1 (2.23)
  CFB at Day 4: 0.25 H Postdose | -0.2 (1.85)
  CFB at Day 4: 0.5 H Postdose | -0.6 (2.19)
  CFB at Day 4: 1 H Postdose | -0.5 (1.68)
  CFB at Day 4: 2 H Postdose: number analyzed (Participants) | 11
  CFB at Day 4: 2 H Postdose | -0.4 (1.50)
  CFB at Day 4: 12 H Postdose | -0.5 (2.07)
  CFB at Day 5: Predose | -0.4 (1.78)
  CFB at Day 5: 0.25 H Postdose | -0.6 (2.11)
  CFB at Day 5: 0.5 H Postdose | -0.2 (1.53)
  CFB at Day 5: 1 H Postdose | -0.5 (1.88)
  CFB at Day 5: 2 H Postdose: number analyzed (Participants) | 10
  CFB at Day 5: 2 H Postdose | -0.7 (2.21)
  CFB at Day 5: 12 H Postdose | -0.2 (1.34)
  CFB at Day 6: Predose | -0.4 (1.00)
  CFB at Day 6: 0.25 H Postdose | -0.5 (1.51)
  CFB at Day 6: 0.5 H Postdose | -0.5 (1.98)
  CFB at Day 6: 1 H Postdose | -0.3 (0.97)
  CFB at Day 6: 2 H Postdose | -0.3 (1.22)
  CFB at Day 6: 12 H Postdose | 0.3 (1.42)
  CFB at Day 7: Predose: number analyzed (Participants) | 11
  CFB at Day 7: Predose | -0.5 (1.44)
  CFB at Day 7: 0.25 H Postdose: number analyzed (Participants) | 11
  CFB at Day 7: 0.25 H Postdose | -0.4 (2.06)
  CFB at Day 7: 0.5 H Postdose | -0.5 (1.51)
  CFB at Day 7: 1 H Postdose | -1.1 (1.93)
  CFB at Day 7: 2 H Postdose | -0.6 (1.31)
  CFB at Day 7: 12 H Postdose: number analyzed (Participants) | 11
  CFB at Day 7: 12 H Postdose | -0.5 (1.63)
  CFB at Day 8: Predose | 0.2 (1.53)
  CFB at Day 8: 1 H Postdose | -0.3 (1.82)

44. Primary Outcome: Change From Baseline in QT Interval - Part A
Description: Electrocardiogram (ECG) measures included QT interval, QTc based on Fridericia formula (QTcF interval), ECG mean heart rate, RR interval, PR interval, and QRS duration. The analysis was performed in participants included in Part A of the study.
Time Frame: Baseline, Days 1, 2, 7, 14 and follow-up Day 21
Population: as for outcome 36
Measure: Median (Full Range); unit: milliseconds (msec)
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
milliseconds (msec)
  Baseline | 401.0 [383 to 452]
  Change from Baseline at Day 1 | -8.0 [-51 to 29]
  Change from Baseline at Day 2 | -12.0 [-67 to 16]
  Change from Baseline at Day 7 | -22.0 [-52 to 10]
  Change from Baseline at Day 14 | -16.0 [-113 to 12]
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 10
  Change from Baseline at Follow-up Day 21 | -17.5 [-46 to 8]

45. Primary Outcome: Change From Baseline in QTcF Interval - Part A
Description: ECG measures included QT interval, QTcF interval, ECG mean heart rate, RR interval, PR interval, and QRS duration. The analysis was performed in participants included in Part A of the study.
Time Frame: Baseline, Days 1, 2, 7, 14 and follow-up Day 21
Population: as for outcome 36
Measure: Median (Full Range); unit: msec
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
msec
  Baseline | 423.0 [393 to 479]
  Change from Baseline at Day 1 | 2.0 [-26 to 17]
  Change from Baseline at Day 2 | -5.0 [-42 to 29]
  Change from Baseline at Day 7 | -4.0 [-44 to 18]
  Change from Baseline at Day 14 | -8.0 [-92 to 15]
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 10
  Change from Baseline at Follow-up Day 21 | -7.0 [-26 to 3]

46. Primary Outcome: Change From Baseline in ECG Mean Heart Rate - Part A
Description: as for outcome 45
Time Frame: Baseline, Days 1, 2, 7, 14 and follow-up Day 21
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
beats/min
  Baseline | 65.6 (7.74)
  Change from Baseline at Day 1 | 5.8 (7.83)
  Change from Baseline at Day 2 | 5.6 (7.05)
  Change from Baseline at Day 7 | 8.8 (9.72)
  Change from Baseline at Day 14 | 6.0 (10.79)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 10
  Change from Baseline at Follow-up Day 21 | 7.0 (6.06)

47. Primary Outcome: Change From Baseline in RR Interval - Part A
Description: as for outcome 45
Time Frame: Baseline, Days 1, 2, 7, 14 and follow-up Day 21
Population: as for outcome 36
Measure: Median (Full Range); unit: msec
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
msec
  Baseline | 952.0 [723 to 1071]
  Change from Baseline at Day 1 | -65.0 [-294 to 78]
  Change from Baseline at Day 2 | -45.0 [-228 to 61]
  Change from Baseline at Day 7 | -88.0 [-330 to 88]
  Change from Baseline at Day 14 | -107.0 [-363 to 147]
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 10
  Change from Baseline at Follow-up Day 21 | -97.0 [-242 to 39]

48. Primary Outcome: Change From Baseline in PR Interval - Part A
Description: as for outcome 45
Time Frame: Baseline, Days 1, 2, 7, 14 and follow-up Day 21
Population: as for outcome 36
Measure: Median (Full Range); unit: msec
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
msec
  Baseline | 158.0 [150 to 338]
  Change from Baseline at Day 1 | 1.0 [-84 to 18]
  Change from Baseline at Day 2 | -8.0 [-134 to 26]
  Change from Baseline at Day 7 | 2.0 [-58 to 20]
  Change from Baseline at Day 14 | 5.0 [-14 to 48]
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 10
  Change from Baseline at Follow-up Day 21 | -3.5 [-23 to 18]

49. Primary Outcome: Change From Baseline in QRS Interval - Part A
Description: as for outcome 45
Time Frame: Baseline, Days 1, 2, 7, 14 and follow-up Day 21
Population: as for outcome 36
Measure: Median (Full Range); unit: msec
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
msec
  Baseline | 94.0 [81 to 114]
  Change from Baseline at Day 1 | 0.0 [-16 to 11]
  Change from Baseline at Day 2 | -2.0 [-22 to 11]
  Change from Baseline at Day 7 | -1.0 [-25 to 10]
  Change from Baseline at Day 14 | 4.0 [-20 to 16]
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 10
  Change from Baseline at Follow-up Day 21 | -0.5 [-14 to 27]

50. Primary Outcome: Percentage of Participants With a Response of 'Yes' to Any Columbia Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation Item - Part A
Description: The C-SSRS scale consisted of a baseline evaluation (at screening) that assessed the lifetime experience of participants with suicidal ideation (SI) and behavior and a postbaseline evaluation that focused on suicidality since the last study visit. The C-SSRS included "yes" or "no"' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe). The C-SSRS SI items involved wish to be dead, non-specific active suicidal thoughts, active SI with any methods, active SI with some intent and active SI with specific plan. The analysis was performed in participants included in Part A of the study.
Time Frame: Day 1 up to Day 28
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
percentage of participants | 0

51. Primary Outcome: Change From Baseline in Stanford Sleepiness Scale (SSS) Score at Day 15 - Part A
Description: The SSS was participant-rated scale designed to quickly assess how alert a participant was feeling. Degrees of sleepiness and alertness were rated on a scale of one to seven, where the lowest score of 'one' indicated the participant was 'feeling active, vital, alert, or wide awake' and the highest score of 'seven' indicated the participant was 'no longer fighting sleep, sleep onset soon; having dream-like thoughts'. A negative change from baseline indicated less sleepiness. A positive change from baseline indicated more sleepiness. The analysis was performed in participants included in Part A of the study.
Time Frame: Baseline, Day 15
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
score on a scale
  Baseline | 2.3 (1.60)
  Change from Baseline at Day 15 | -0.6 (1.50)

52. Primary Outcome: Change From Baseline in the 17-item Hamilton Rating Scale for Depression (HAM-D) Total Score at Day 15 - Part B
Description: The HAM-D total score comprised a sum of 17 individual item scores. Items scored in a range of 0 to 2 included: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score could range from 0 to 52. Higher scores indicated a greater degree of depression. A negative change from baseline indicated less depression. A positive change from baseline indicated more depression. The analysis was performed in participants included in Part B of the study.
Time Frame: Baseline, Day 15
Population: The efficacy set included all participants who were randomized and received at least 1 dose of the double-blind study drug and had a baseline and at least 1 post-baseline efficacy evaluation.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
score on a scale | -10.3 (1.33) | -17.4 (1.31)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE-217; Test type: Superiority; p < 0.0001, Mixed Effect Model for Repeated Measures; The Mixed Effect Model for Repeated Measures (MMRM) included the change from baseline in HAM-D total score at each visit as the dependent variables; Least Squares Mean Difference = -7.0, 95% CI 2-sided [-10.2 to -3.9], Standard Error of Mean 1.60

53. Secondary Outcome: Change From Baseline in the HAM-D Total Score at Day 15 and All Other Time Points - Part A
Description: The HAM-D total score comprised a sum of 17 individual item scores. Items scored in a range of 0 to 2 included: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score could range from 0 to 52. Higher scores indicate a greater degree of depression. A negative change from baseline indicated less depression. A positive change from baseline indicated more depression. The analysis was performed in participants included in Part A of the study.
Time Frame: Baseline, Days 2, 3, 4, 5, 6, 7, 8, 15, 21 and 28
Population: The efficacy set included all participants who received at least one dose of the study drug and had a baseline and at least one postbaseline efficacy evaluation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
score on a scale
  Baseline | 27.2 (3.06)
  Change from Baseline at Day 2 | -5.9 (4.44)
  Change from Baseline at Day 3 | -9.1 (4.82)
  Change from Baseline at Day 4 | -12.4 (5.74)
  Change from Baseline at Day 5 | -14.4 (5.68)
  Change from Baseline at Day 6 | -16.0 (5.48)
  Change from Baseline at Day 7 | -16.2 (6.01)
  Change from Baseline at Day 8 | -18.2 (5.94)
  Change from Baseline at Day 15 | -19.9 (5.78)
  Change from Baseline at Day 21 | -20.5 (7.11)
  Change from Baseline at Day 28 | -19.7 (8.09)

54. Secondary Outcome: Percentage of Participants With TEAEs - Part B
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A TEAE was defined as an adverse event with onset after the start of study drug, or any worsening of a pre-existing medical condition/adverse event with onset after the start of study drug and until 7 days after the last dose. The analysis was performed in participants included in Part B of the study.
Time Frame: Day 1 up to Day 21
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
percentage of participants | 45.5 | 53.3

55. Secondary Outcome: Percentage of Participants With AEs During Post-TEAE Period
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. TEAE was defined as an adverse event with onset after the start of study drug, or any worsening of a pre-existing medical condition/adverse event with onset after the start of study drug and until 7 days after the last dose. Post-TEAE period was defined as 7 days after final dose through last follow-up (Day 42). The analysis was performed in participants included in Part B of the study.
Time Frame: Day 21 up to Day 42
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
percentage of participants | 22.7 | 8.9

56. Secondary Outcome: Percentage of Participants With TEAEs, Graded by Severity - Part B
Description: Severity was assessed according to the following scale: mild (awareness of sign or symptom, but easily tolerated); moderate (discomfort sufficient to cause interference with normal activities); severe (incapacitating, with inability to perform normal activities). The analysis was performed in participants included in Part B of the study.
Time Frame: Day 1 up to Day 21
Population: The safety set included all participants who received at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
percentage of participants
  Moderate or Severe | 5 | 6
  Severe | 0 | 0

57. Secondary Outcome: Change From Baseline in Basophils - Part B
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, hematocrit, hemoglobin, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets, erythrocytes, reticulocytes, reticulocytes to erythrocytes ratio and leukocytes. The analysis was performed in participants included in Part B of the study. ET = Early Termination.
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: The safety set included all participants who received at least one dose of the study drug. Number analyzed: Number of participants in safety set with a non-missing value at both baseline and the visit within each treatment group.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
10^9 cells/L
  Baseline | 0.038 (0.0478) | 0.041 (0.0489)
  Change from Baseline at Day 8: number analyzed (Participants) | 41 | 42
  Change from Baseline at Day 8 | 0.012 (0.0495) | -0.004 (0.0520)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | 0.005 (0.0486) | 0.001 (0.0359)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | 0.000 (0.0484) | -0.013 (0.0396)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | 0.008 (0.0497) | -0.018 (0.0436)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 40
  Change from Baseline at Follow-up Day 35 | 0.008 (0.0561) | 0.007 (0.0352)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | 0.011 (0.0483) | -0.006 (0.0494)

58. Secondary Outcome: Change From Baseline in Basophils to Leukocytes Ratio (%) - Part B
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, hematocrit, hemoglobin, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets, erythrocytes, reticulocytes, reticulocytes to erythrocytes ratio and leukocytes. The analysis was performed in participants included in Part B of the study. ET = Early Termination. The blood cell differential (ratio) data are presented as SI unit, percentage (%).
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: The safety set included all participants who received at least one dose of the study drug. Number analyzed: Number of participants in the safety set with a non-missing value at both baseline and the visit within each treatment group.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
percentage
  Baseline | 0.63 (0.302) | 0.63 (0.274)
  Change from Baseline at Day 8: number analyzed (Participants) | 41 | 42
  Change from Baseline at Day 8 | 0.11 (0.241) | 0.04 (0.229)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | 0.05 (0.174) | 0.11 (0.231)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | 0.06 (0.227) | 0.02 (0.240)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | 0.05 (0.258) | -0.01 (0.318)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 40
  Change from Baseline at Follow-up Day 35 | 0.04 (0.265) | 0.10 (0.180)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | 0.10 (0.240) | 0.07 (0.255)

59. Secondary Outcome: Change From Baseline in Eosinophils - Part B
Description: as for outcome 57
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
10^9 cells/L
  Baseline | 0.147 (0.0818) | 0.126 (0.0801)
  Change from Baseline at Day 8: number analyzed (Participants) | 41 | 42
  Change from Baseline at Day 8 | 0.004 (0.0578) | 0.025 (0.0795)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | 0.027 (0.0804) | 0.037 (0.0890)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | 0.020 (0.0789) | 0.027 (0.0696)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | 0.022 (0.0940) | 0.015 (0.0724)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 40
  Change from Baseline at Follow-up Day 35 | 0.006 (0.0799) | 0.012 (0.0760)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | 0.017 (0.0772) | 0.017 (0.0735)

60. Secondary Outcome: Change From Baseline in Eosinophils to Leukocytes Ratio (%) - Part B
Description: as for outcome 58
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
percentage
  Baseline | 1.95 (1.018) | 1.96 (1.267)
  Change from Baseline at Day 8: number analyzed (Participants) | 41 | 42
  Change from Baseline at Day 8 | 0.15 (0.780) | 0.44 (1.102)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | 0.53 (1.042) | 0.60 (1.166)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | 0.48 (1.080) | 0.53 (0.916)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | 0.48 (1.221) | 0.39 (1.092)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 40
  Change from Baseline at Follow-up Day 35 | 0.42 (0.996) | 0.37 (1.015)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | 0.55 (1.089) | 0.46 (1.192)

61. Secondary Outcome: Change From Baseline in Hematocrit - Part B
Description: as for outcome 57
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: fraction of one
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
fraction of one
  Baseline | 0.424 (0.0372) | 0.436 (0.0389)
  Change from Baseline at Day 8: number analyzed (Participants) | 41 | 42
  Change from Baseline at Day 8 | -0.004 (0.0240) | -0.004 (0.0281)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | -0.006 (0.0210) | -0.010 (0.0230)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -0.015 (0.0233) | -0.020 (0.0249)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -0.015 (0.0235) | -0.015 (0.0220)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 40
  Change from Baseline at Follow-up Day 35 | -0.011 (0.0253) | -0.015 (0.0244)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | -0.015 (0.0223) | -0.019 (0.0245)

62. Secondary Outcome: Change From Baseline in Hemoglobin - Part B
Description: as for outcome 57
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
g/L
  Baseline | 136.1 (13.79) | 141.0 (14.98)
  Change from Baseline at Day 8: number analyzed (Participants) | 41 | 42
  Change from Baseline at Day 8 | -1.3 (7.72) | -2.3 (9.09)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | -1.8 (6.88) | -3.8 (7.80)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -5.2 (7.41) | -6.6 (7.91)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -4.9 (7.44) | -4.9 (7.29)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 40
  Change from Baseline at Follow-up Day 35 | -3.8 (8.16) | -5.1 (8.18)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | -4.7 (6.44) | -5.6 (8.18)

63. Secondary Outcome: Change From Baseline in Lymphocytes - Part B
Description: as for outcome 57
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
10^9 cells/L
  Baseline | 2.294 (0.6093) | 2.162 (0.6275)
  Change from Baseline at Day 8: number analyzed (Participants) | 41 | 42
  Change from Baseline at Day 8 | -0.053 (0.4033) | -0.054 (0.4501)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | 0.066 (0.5139) | 0.025 (0.4944)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -0.106 (0.5656) | -0.104 (0.5341)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -0.073 (0.5071) | -0.247 (0.5428)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 40
  Change from Baseline at Follow-up Day 35 | -0.153 (0.4178) | -0.209 (0.5137)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | -0.168 (0.4661) | -0.133 (0.4544)

64. Secondary Outcome: Change From Baseline in Lymphocytes to Leukocytes Ratio (%) - Part B
Description: as for outcome 58
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
percentage
  Baseline | 33.06 (7.144) | 33.87 (10.189)
  Change from Baseline at Day 8: number analyzed (Participants) | 41 | 42
  Change from Baseline at Day 8 | -0.43 (6.613) | 1.86 (7.057)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | 1.25 (7.203) | 1.96 (8.304)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | 0.04 (7.177) | -0.13 (9.353)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | 0.61 (9.038) | -0.61 (9.527)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 40
  Change from Baseline at Follow-up Day 35 | -0.75 (7.861) | -0.02 (8.937)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | 0.91 (6.960) | 0.30 (8.641)

65. Secondary Outcome: Change From Baseline in Monocytes - Part B
Description: as for outcome 57
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
10^9 cells/L
  Baseline | 0.442 (0.1206) | 0.438 (0.1339)
  Change from Baseline at Day 8: number analyzed (Participants) | 41 | 42
  Change from Baseline at Day 8 | 0.003 (0.1209) | 0.035 (0.1631)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | 0.017 (0.1253) | 0.028 (0.1185)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | 0.007 (0.1063) | 0.025 (0.1333)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | 0.045 (0.1415) | -0.010 (0.1523)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 40
  Change from Baseline at Follow-up Day 35 | 0.024 (0.1364) | 0.002 (0.1381)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | 0.011 (0.1050) | 0.004 (0.1313)

66. Secondary Outcome: Change From Baseline in Monocytes to Leukocytes Ratio (%) - Part B
Description: as for outcome 58
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
percentage
  Baseline | 6.33 (1.760) | 6.78 (1.970)
  Change from Baseline at Day 8: number analyzed (Participants) | 41 | 42
  Change from Baseline at Day 8 | 0.20 (1.430) | 0.98 (1.661)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | 0.40 (1.942) | 0.79 (1.617)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | 0.57 (1.473) | 0.90 (2.030)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | 0.97 (1.869) | 0.77 (2.562)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 40
  Change from Baseline at Follow-up Day 35 | 0.66 (1.546) | 0.78 (2.374)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | 0.94 (1.270) | 0.74 (2.076)

67. Secondary Outcome: Change From Baseline in Neutrophils - Part B
Description: as for outcome 57
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
10^9 cells/L
  Baseline | 4.174 (1.4046) | 3.852 (1.5129)
  Change from Baseline at Day 8: number analyzed (Participants) | 41 | 42
  Change from Baseline at Day 8 | -0.100 (1.1146) | -0.399 (1.7192)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | -0.389 (1.2882) | -0.406 (1.2479)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -0.354 (1.0854) | -0.280 (1.3687)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -0.363 (1.2994) | -0.454 (1.3814)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 40
  Change from Baseline at Follow-up Day 35 | -0.209 (1.3250) | -0.494 (1.0343)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | -0.584 (1.2204) | -0.323 (1.4669)

68. Secondary Outcome: Change From Baseline in Neutrophils to Leukocytes Ratio (%) - Part B
Description: as for outcome 58
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
percentage
  Baseline | 58.03 (7.850) | 56.76 (10.809)
  Change from Baseline at Day 8: number analyzed (Participants) | 41 | 42
  Change from Baseline at Day 8 | -0.03 (7.549) | -3.32 (8.015)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | -2.23 (8.600) | -3.46 (9.345)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -1.15 (8.173) | -1.32 (10.154)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -2.11 (10.514) | -0.63 (11.160)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 40
  Change from Baseline at Follow-up Day 35 | -0.38 (9.087) | -1.22 (9.600)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | -2.50 (7.678) | -1.58 (9.818)

69. Secondary Outcome: Change From Baseline in Platelets - Part B
Description: as for outcome 57
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 44
10^9 cells/L
  Baseline | 287.0 (74.33) | 272.2 (60.08)
  Change from Baseline at Day 8: number analyzed (Participants) | 40 | 41
  Change from Baseline at Day 8 | -8.5 (42.93) | -0.9 (36.43)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 40
  Change from Baseline at Day 15/ET | 6.8 (39.39) | 3.7 (36.16)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 41
  Change from Baseline at Follow-up Day 21 | 4.7 (32.94) | 7.4 (29.01)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 41
  Change from Baseline at Follow-up Day 28 | 3.5 (40.30) | 5.0 (31.48)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 39
  Change from Baseline at Follow-up Day 35 | -4.9 (43.23) | -1.7 (31.25)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 41
  Change from Baseline at Follow-up Day 42 | -1.8 (48.71) | -2.7 (33.61)

70. Secondary Outcome: Change From Baseline in Erythrocytes - Part B
Description: as for outcome 57
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
10^12 cells/L
  Baseline | 4.811 (0.4827) | 4.902 (0.4956)
  Change from Baseline at Day 8: number analyzed (Participants) | 41 | 42
  Change from Baseline at Day 8 | -0.041 (0.2802) | -0.074 (0.2889)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | -0.069 (0.2436) | -0.128 (0.2714)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -0.182 (0.2841) | -0.225 (0.2794)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -0.176 (0.2599) | -0.172 (0.2684)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 40
  Change from Baseline at Follow-up Day 35 | -0.134 (0.3050) | -0.189 (0.2675)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | -0.161 (0.2365) | -0.202 (0.3181)

71. Secondary Outcome: Change From Baseline in Reticulocytes - Part B
Description: as for outcome 57
Time Frame: Baseline, Day 8, Day 15/ET
Population: The safety set included all participants who received at least one dose of the study drug. Overall number of participants analyzed: Number of participants analyzed in this outcome measure. Number analyzed: Number of participants in the safety set with a non-missing value at both baseline and the visit within each treatment group.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 3 | 2
10^9 cells/L
  Baseline | 32.313 (19.0547) | 78.735 (58.5272)
  Change from Baseline at Day 8: number analyzed (Participants) | 2 | 0
  Change from Baseline at Day 8 | -19.035 (12.9613) |
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 1 | 0
  Change from Baseline at Day 15/ET | 9.240 (NA) — Standard deviation was not calculated since only one participant was analyzed. |

72. Secondary Outcome: Change From Baseline in Reticulocytes to Erythrocytes Ratio (%) - Part B
Description: as for outcome 58
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 42 | 43
percentage
  Baseline | 1.32 (0.360) | 1.40 (0.517)
  Change from Baseline at Day 8: number analyzed (Participants) | 38 | 40
  Change from Baseline at Day 8 | -0.02 (0.290) | -0.07 (0.363)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 40 | 39
  Change from Baseline at Day 15/ET | -0.03 (0.310) | 0.00 (0.372)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 36 | 40
  Change from Baseline at Follow-up Day 21 | 0.14 (0.352) | 0.05 (0.359)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 37 | 40
  Change from Baseline at Follow-up Day 28 | 0.17 (0.289) | 0.03 (0.296)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 38 | 39
  Change from Baseline at Follow-up Day 35 | 0.15 (0.254) | 0.07 (0.320)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 37 | 40
  Change from Baseline at Follow-up Day 42 | 0.12 (0.227) | 0.03 (0.312)

73. Secondary Outcome: Change From Baseline in Leukocytes - Part B
Description: as for outcome 57
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
10^9 cells/L
  Baseline | 7.08 (1.778) | 6.63 (1.688)
  Change from Baseline at Day 8: number analyzed (Participants) | 41 | 42
  Change from Baseline at Day 8 | -0.11 (1.324) | -0.40 (1.913)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | -0.27 (1.435) | -0.34 (1.241)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -0.41 (1.258) | -0.35 (1.410)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -0.34 (1.266) | -0.70 (1.348)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 40
  Change from Baseline at Follow-up Day 35 | -0.32 (1.355) | -0.70 (0.993)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | -0.69 (1.421) | -0.45 (1.443)

74. Secondary Outcome: Change From Baseline in Albumin - Part B
Description: Clinical chemistry measures included albumin, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, bilirubin, calcium, chloride, carbon dioxide, creatinine, glucose, potassium, magnesium, phosphate, protein, sodium, thyrotropin, and urea nitrogen. The analysis was performed in participants included in Part B of the study. ET = Early Termination.
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
g/L
  Baseline | 44.6 (2.69) | 44.6 (3.30)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 8 | -1.1 (2.66) | -0.8 (3.24)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 42
  Change from Baseline at Day 15/ET | -0.8 (2.73) | -0.9 (3.23)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -1.1 (2.72) | -1.4 (3.40)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -0.2 (3.01) | -0.9 (3.07)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  Change from Baseline at Follow-up Day 35 | -0.5 (2.90) | -1.0 (3.40)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | -0.5 (2.30) | -0.7 (3.43)

75. Secondary Outcome: Change From Baseline in Alkaline Phosphatase - Part B
Description: as for outcome 74
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
U/L
  Baseline | 80.9 (19.18) | 85.5 (27.97)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 8 | -0.1 (8.95) | 1.3 (14.37)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 42
  Change from Baseline at Day 15/ET | 1.6 (10.39) | 3.1 (17.84)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -0.9 (7.66) | -2.9 (13.64)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -0.8 (8.50) | -2.5 (11.01)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  Change from Baseline at Follow-up Day 35 | 1.0 (8.28) | -4.3 (8.87)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | -0.4 (12.97) | -4.4 (9.26)

76. Secondary Outcome: Change From Baseline in Alanine Aminotransferase - Part B
Description: as for outcome 74
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
U/L
  Baseline | 22.9 (11.09) | 22.2 (9.43)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 8 | 4.1 (13.09) | 11.0 (28.79)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | 7.3 (22.23) | 9.1 (32.27)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | 3.4 (22.86) | 0.1 (6.50)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | 1.6 (9.57) | -0.8 (6.21)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  Change from Baseline at Follow-up Day 35 | 0.5 (8.55) | 0.5 (10.11)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | -0.2 (10.12) | -1.0 (6.30)

77. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase - Part B
Description: as for outcome 74
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
U/L
  Baseline | 23.0 (5.19) | 23.5 (6.49)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 8 | -0.5 (6.31) | 10.0 (43.42)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | 2.2 (12.54) | 5.0 (27.21)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | 1.4 (11.60) | -0.1 (6.79)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -0.5 (4.89) | -0.3 (7.62)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  Change from Baseline at Follow-up Day 35 | -1.2 (5.43) | -0.5 (7.36)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | 0.1 (7.03) | -0.1 (6.40)

78. Secondary Outcome: Change From Baseline in Bilirubin - Part B
Description: as for outcome 74
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
umol/L
  Baseline | 8.157 (3.5160) | 9.422 (7.5457)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 8 | -1.095 (2.7830) | -1.670 (4.7335)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 42
  Change from Baseline at Day 15/ET | -0.652 (3.3092) | -1.673 (3.1661)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -0.453 (3.7470) | -0.978 (3.0372)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -1.049 (3.0737) | 0.162 (3.7768)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  Change from Baseline at Follow-up Day 35 | -0.945 (3.6470) | -1.170 (4.3101)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | -0.708 (3.9947) | -0.526 (4.4450)

79. Secondary Outcome: Change From Baseline in Calcium - Part B
Description: as for outcome 74
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
mmol/L
  Baseline | 2.359 (0.0909) | 2.364 (0.1517)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 8 | -0.021 (0.0911) | -0.033 (0.1220)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 42
  Change from Baseline at Day 15/ET | -0.019 (0.1083) | -0.041 (0.1171)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -0.038 (0.0900) | -0.065 (0.1120)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -0.035 (0.1138) | -0.044 (0.0961)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  Change from Baseline at Follow-up Day 35 | -0.038 (0.1024) | -0.048 (0.1201)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | -0.041 (0.0954) | -0.041 (0.1290)

80. Secondary Outcome: Change From Baseline in Chloride - Part B
Description: as for outcome 74
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
mmol/L
  Baseline | 104.7 (1.87) | 104.4 (2.53)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 8 | -0.2 (2.49) | -0.2 (2.86)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 42
  Change from Baseline at Day 15/ET | -0.4 (2.10) | -0.1 (2.83)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | 0.8 (2.59) | 0.5 (2.37)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | 0.6 (2.47) | 0.3 (3.27)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  Change from Baseline at Follow-up Day 35 | 0.0 (2.50) | 1.1 (2.49)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | 0.4 (2.39) | 0.8 (2.75)

81. Secondary Outcome: Change From Baseline in Carbon Dioxide - Part B
Description: as for outcome 74
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
mmol/L
  Baseline | 29.3 (2.32) | 28.8 (2.25)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 8 | -1.1 (2.87) | 0.0 (2.61)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 42
  Change from Baseline at Day 15/ET | -0.3 (2.41) | 0.7 (2.32)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -1.1 (2.31) | 0.2 (2.50)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -1.0 (2.84) | -0.5 (2.69)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  Change from Baseline at Follow-up Day 35 | -1.0 (2.56) | -0.1 (2.68)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | -0.8 (2.86) | -0.8 (2.70)

82. Secondary Outcome: Change From Baseline in Creatinine - Part B
Description: as for outcome 74
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
umol/L
  Baseline | 76.363 (16.0294) | 77.894 (14.1946)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 8 | 0.036 (7.6537) | -1.710 (8.0850)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 42
  Change from Baseline at Day 15/ET | 1.028 (9.1198) | 0.566 (7.9601)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | 0.632 (8.8186) | 1.495 (9.8651)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | 4.462 (7.4979) | 2.614 (6.6486)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  Change from Baseline at Follow-up Day 35 | 2.300 (9.0428) | 1.263 (14.2508)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | 1.949 (8.5582) | 0.852 (9.5738)

83. Secondary Outcome: Change From Baseline in Glucose - Part B
Description: as for outcome 74
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
mmol/L
  Baseline | 5.438 (1.8453) | 5.114 (0.9726)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 8 | 0.103 (1.4778) | 0.045 (1.4529)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 42
  Change from Baseline at Day 15/ET | 0.203 (1.5462) | 0.390 (1.5054)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 37 | 42
  Change from Baseline at Follow-up Day 21 | -0.031 (1.2125) | -0.308 (1.3738)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -0.053 (1.1142) | 0.166 (1.3791)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  Change from Baseline at Follow-up Day 35 | -0.094 (1.5798) | 0.355 (1.6032)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | 0.114 (1.3631) | 0.059 (1.1655)

84. Secondary Outcome: Change From Baseline in Potassium - Part B
Description: as for outcome 74
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
mmol/L
  Baseline | 4.33 (0.362) | 4.36 (0.442)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 8 | 0.05 (0.432) | 0.09 (0.517)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 42
  Change from Baseline at Day 15/ET | 0.05 (0.402) | 0.03 (0.408)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 37 | 42
  Change from Baseline at Follow-up Day 21 | 0.01 (0.371) | -0.01 (0.467)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | 0.05 (0.342) | 0.00 (0.581)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  Change from Baseline at Follow-up Day 35 | 0.07 (0.351) | -0.04 (0.468)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | 0.04 (0.420) | -0.06 (0.491)

85. Secondary Outcome: Change From Baseline in Magnesium - Part B
Description: as for outcome 74
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 42 | 45
mmol/L
  Baseline | 0.891 (0.0772) | 0.879 (0.0977)
  Change from Baseline at Day 8: number analyzed (Participants) | 40 | 44
  Change from Baseline at Day 8 | -0.020 (0.0911) | -0.011 (0.0950)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 40 | 42
  Change from Baseline at Day 15/ET | -0.025 (0.0980) | -0.014 (0.1095)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 36 | 42
  Change from Baseline at Follow-up Day 21 | -0.023 (0.0864) | -0.025 (0.0998)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 37 | 42
  Change from Baseline at Follow-up Day 28 | -0.009 (0.0996) | -0.030 (0.0804)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 38 | 41
  Change from Baseline at Follow-up Day 35 | -0.033 (0.0981) | -0.033 (0.1046)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 37 | 45
  Change from Baseline at Follow-up Day 42 | -0.012 (0.1070) | -0.025 (0.0929)

86. Secondary Outcome: Change From Baseline in Phosphate - Part B
Description: as for outcome 74
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 42 | 45
mmol/L
  Baseline | 1.245 (0.1623) | 1.212 (0.1359)
  Change from Baseline at Day 8: number analyzed (Participants) | 40 | 44
  Change from Baseline at Day 8 | 0.053 (0.2050) | 0.048 (0.2078)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 40 | 41
  Change from Baseline at Day 15/ET | 0.019 (0.1969) | 0.010 (0.1798)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 35 | 42
  Change from Baseline at Follow-up Day 21 | -0.015 (0.1609) | -0.102 (0.1652)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 37 | 42
  Change from Baseline at Follow-up Day 28 | -0.022 (0.1657) | -0.084 (0.2291)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 38 | 41
  Change from Baseline at Follow-up Day 35 | -0.108 (0.1761) | -0.120 (0.2033)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 37 | 42
  Change from Baseline at Follow-up Day 42 | -0.102 (0.1600) | -0.089 (0.1941)

87. Secondary Outcome: Change From Baseline in Protein - Part B
Description: as for outcome 74
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
g/L
  Baseline | 75.0 (5.02) | 76.0 (5.90)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 8 | -2.1 (4.47) | -1.3 (5.47)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 42
  Change from Baseline at Day 15/ET | -1.3 (4.45) | -1.6 (5.90)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -2.1 (4.05) | -2.5 (5.77)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -0.9 (5.05) | -1.9 (5.58)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  Change from Baseline at Follow-up Day 35 | -1.2 (4.61) | -2.3 (5.72)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | -1.4 (4.01) | -2.1 (5.73)

88. Secondary Outcome: Change From Baseline in Sodium - Part B
Description: as for outcome 74
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
mmol/L
  Baseline | 140.8 (1.78) | 140.5 (1.82)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 8 | -0.7 (1.74) | 0.1 (2.08)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 42
  Change from Baseline at Day 15/ET | -0.6 (1.94) | 0.0 (2.60)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | 0.3 (2.00) | 0.0 (2.33)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -0.1 (2.14) | -0.1 (2.68)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  Change from Baseline at Follow-up Day 35 | -0.8 (2.20) | 0.3 (2.26)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | -0.6 (2.10) | -0.1 (2.28)

89. Secondary Outcome: Change From Baseline in Thyrotropin - Part B
Description: as for outcome 74
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: milli-international units per liter
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
milli-international units per liter
  Baseline | 1.328 (0.7996) | 1.398 (0.9451)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 8 | 0.464 (0.8096) | 0.445 (0.7181)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 41 | 41
  Change from Baseline at Day 15/ET | 0.668 (1.5106) | 0.315 (0.6782)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -0.011 (0.7579) | -0.014 (0.7316)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | 0.218 (0.8047) | 0.099 (0.6297)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  Change from Baseline at Follow-up Day 35 | 0.156 (0.7314) | 0.103 (0.5723)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | 0.156 (1.0520) | 0.124 (0.5530)

90. Secondary Outcome: Change From Baseline in Urea Nitrogen - Part B
Description: as for outcome 74
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
mmol/L
  Baseline | 4.186 (1.4151) | 4.644 (2.0582)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 8 | 0.322 (1.0179) | 0.334 (1.6435)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 42
  Change from Baseline at Day 15/ET | 0.330 (1.2817) | 0.189 (1.6860)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -0.096 (1.1059) | 0.196 (1.0191)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | 0.057 (1.2372) | 0.186 (1.0919)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  Change from Baseline at Follow-up Day 35 | 0.138 (1.0796) | 0.078 (1.4422)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 41
  Change from Baseline at Follow-up Day 42 | 0.057 (1.2051) | -0.275 (1.1708)

91. Secondary Outcome: Change From Baseline in Activated Partial Thromboplastin Time - Part B
Description: Coagulation measures included activated partial thromboplastin time, prothrombin international normalized ratio, and prothrombin time. The analysis was performed in participants included in Part B of the study. ET = Early Termination.
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Median (Full Range); unit: sec
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
sec
  Baseline | 27.60 [24.0 to 32.4] | 27.80 [23.6 to 33.0]
  Change from Baseline at Day 8: number analyzed (Participants) | 40 | 41
  Change from Baseline at Day 8 | 0.20 [-5.1 to 24.2] | -0.20 [-2.8 to 4.5]
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 40 | 41
  Change from Baseline at Day 15/ET | 0.10 [-3.5 to 3.6] | 0.40 [-3.0 to 6.4]
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 37 | 40
  Change from Baseline at Follow-up Day 21 | 0.40 [-4.2 to 3.0] | 0.05 [-3.5 to 3.3]
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 40
  Change from Baseline at Follow-up Day 28 | 0.40 [-3.1 to 2.6] | 0.30 [-2.1 to 3.8]
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 38 | 40
  Change from Baseline at Follow-up Day 35 | 0.10 [-2.9 to 4.1] | -0.25 [-4.1 to 3.5]
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 41
  Change from Baseline at Follow-up Day 42 | 0.30 [-3.1 to 4.5] | 0.20 [-3.5 to 6.2]

92. Secondary Outcome: Change From Baseline in Prothrombin International Normalized Ratio (%) - Part B
Description: Coagulation measures included activated partial thromboplastin time, prothrombin international normalized ratio, and prothrombin time. The analysis was performed in participants included in Part B of the study. ET = Early Termination. The data for prothrombin international normalized ratio are presented as SI unit, percentage (%).
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
percentage
  Baseline | 1.006 (0.0394) | 1.032 (0.0527)
  Change from Baseline at Day 8: number analyzed (Participants) | 40 | 41
  Change from Baseline at Day 8 | 0.011 (0.0466) | -0.016 (0.0436)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 40 | 41
  Change from Baseline at Day 15/ET | -0.003 (0.0426) | -0.010 (0.0628)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 37 | 40
  Change from Baseline at Follow-up Day 21 | 0.002 (0.0380) | -0.003 (0.0372)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 40
  Change from Baseline at Follow-up Day 28 | -0.007 (0.0337) | 0.002 (0.0440)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 38 | 40
  Change from Baseline at Follow-up Day 35 | -0.002 (0.0439) | -0.005 (0.0384)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 41
  Change from Baseline at Follow-up Day 42 | 0.002 (0.0390) | 0.003 (0.0420)

93. Secondary Outcome: Change From Baseline in Prothrombin Time - Part B
Description: as for outcome 91
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Median (Full Range); unit: sec
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
sec
  Baseline | 10.40 [9.7 to 11.4] | 10.60 [9.9 to 12.2]
  Change from Baseline at Day 8: number analyzed (Participants) | 40 | 41
  Change from Baseline at Day 8 | 0.00 [-0.7 to 2.0] | -0.20 [-1.0 to 0.7]
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 40 | 41
  Change from Baseline at Day 15/ET | 0.00 [-1.1 to 1.0] | -0.20 [-1.0 to 2.6]
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 37 | 40
  Change from Baseline at Follow-up Day 21 | 0.10 [-1.0 to 0.8] | -0.10 [-0.8 to 0.7]
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 40
  Change from Baseline at Follow-up Day 28 | -0.10 [-0.8 to 0.8] | 0.10 [-1.0 to 1.6]
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 36 | 38
  Change from Baseline at Follow-up Day 35 | 0.00 [-1.0 to 1.4] | 0.05 [-0.8 to 0.6]
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 38 | 40
  Change from Baseline at Follow-up Day 42 | 0.10 [-0.7 to 0.8] | 0.00 [-0.8 to 1.2]

94. Secondary Outcome: Change From Baseline in pH - Part B
Description: Urinalysis measures included pH and specific gravity. The analysis was performed in participants included in Part B of the study. ET = Early Termination.
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
pH
  Baseline | 6.22 (0.879) | 6.23 (0.857)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 43
  Change from Baseline at Day 8 | -0.32 (0.923) | -0.16 (1.169)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | -0.37 (0.877) | -0.23 (0.909)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -0.32 (0.940) | -0.15 (0.852)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | -0.27 (0.945) | -0.31 (1.065)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 39 | 41
  Change from Baseline at Follow-up Day 35 | -0.01 (1.275) | -0.17 (0.933)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | -0.12 (1.109) | -0.42 (0.962)

95. Secondary Outcome: Change From Baseline in Specific Gravity - Part B
Description: as for outcome 94
Time Frame: Baseline, Day 8, Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
ratio
  Baseline | 1.016 (0.0086) | 1.018 (0.0092)
  Change from Baseline at Day 8: number analyzed (Participants) | 42 | 43
  Change from Baseline at Day 8 | 0.002 (0.0092) | 0.000 (0.0090)
  Change from Baseline at Day 15/ET: number analyzed (Participants) | 42 | 41
  Change from Baseline at Day 15/ET | 0.003 (0.0092) | -0.001 (0.0106)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | 0.003 (0.0101) | 0.000 (0.0094)
  Change from Baseline at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 28 | 0.004 (0.0093) | 0.002 (0.0087)
  Change from Baseline at Follow-up Day 35: number analyzed (Participants) | 39 | 41
  Change from Baseline at Follow-up Day 35 | 0.001 (0.0096) | 0.001 (0.0099)
  Change from Baseline at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  Change from Baseline at Follow-up Day 42 | 0.004 (0.0086) | 0.002 (0.0112)

96. Secondary Outcome: Change From Baseline (CFB) in Supine Systolic Blood Pressure - Part B
Description: Vital signs measures included supine systolic blood pressure, supine diastolic blood pressure, standing systolic blood pressure, standing diastolic blood pressure, heart rate, respiratory rate, oral temperature, and oxygen saturation. The analysis was performed in participants included in Part B of the study. H = Hour(s). ET = Early Termination.
Time Frame: Baseline, Day 1 (0.25, 0.5, 1, 2, 12 hours postdose), Days 2, 3, 4, 5, 6 and 7 (predose, 0.25, 0.5, 1, 2, 12 hours postdose), Days 8, 9, 10, 11, 12, 13 and 14 (predose, 1 hour postdose), Day 15/ET, follow-up Days 21, 28, 35 and 42
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
mmHg
  Baseline | 120.5 (15.41) | 120.6 (13.95)
  CFB at Day 1: 0.25 H Postdose | 1.7 (9.33) | 0.6 (9.57)
  CFB at Day 1: 0.5 H Postdose | 1.3 (8.38) | 0.7 (10.38)
  CFB at Day 1: 1 H Postdose | 1.1 (8.63) | -0.3 (11.09)
  CFB at Day 1: 2 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 1: 2 H Postdose | 2.3 (11.51) | -0.5 (11.92)
  CFB at Day 1: 12 H Postdose | 0.0 (12.72) | -1.5 (10.58)
  CFB at Day 2: Predose | -0.3 (10.62) | -0.9 (10.72)
  CFB at Day 2: 0.25 H Postdose | 2.7 (12.88) | 0.9 (12.39)
  CFB at Day 2: 0.5 H Postdose | 1.9 (9.49) | 0.2 (13.18)
  CFB at Day 2: 1 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 2: 1 H Postdose | 2.2 (10.83) | -0.5 (11.19)
  CFB at Day 2: 2 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 2: 2 H Postdose | 1.7 (11.72) | -0.2 (12.39)
  CFB at Day 2: 12 H Postdose | -1.2 (11.11) | -1.4 (12.55)
  CFB at Day 3: Predose | 1.3 (10.50) | -0.1 (12.61)
  CFB at Day 3: 0.25 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 3: 0.25 H Postdose | 2.4 (10.49) | 0.4 (12.37)
  CFB at Day 3: 0.5 H Postdose | 3.4 (13.80) | -0.9 (13.55)
  CFB at Day 3: 1 H Postdose | 2.2 (10.18) | -0.3 (12.76)
  CFB at Day 3: 2 H Postdose | 1.5 (12.35) | -0.2 (14.21)
  CFB at Day 3: 12 H Postdose | -2.7 (13.22) | -3.9 (12.84)
  CFB at Day 4: Predose | 1.1 (13.77) | 0.6 (12.38)
  CFB at Day 4: 0.25 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 4: 0.25 H Postdose | 1.3 (11.83) | 2.8 (11.28)
  CFB at Day 4: 0.5 H Postdose | 2.2 (12.29) | 0.7 (10.42)
  CFB at Day 4: 1 H Postdose | -0.5 (11.88) | 0.4 (11.41)
  CFB at Day 4: 2 H Postdose | -1.4 (13.06) | 0.3 (12.84)
  CFB at Day 4: 12 H Postdose: number analyzed (Participants) | 43 | 44
  CFB at Day 4: 12 H Postdose | -2.8 (14.65) | -0.1 (14.51)
  CFB at Day 5: Predose | -1.9 (12.82) | 1.0 (13.67)
  CFB at Day 5: 0.25 H Postdose | -0.8 (11.60) | 2.6 (11.60)
  CFB at Day 5: 0.5 H Postdose | 0.3 (14.05) | 1.2 (9.26)
  CFB at Day 5: 1 H Postdose | -0.4 (10.26) | 2.3 (11.04)
  CFB at Day 5: 2 H Postdose | 0.8 (10.42) | -2.4 (10.78)
  CFB at Day 5: 12 H Postdose | -1.7 (13.79) | -1.8 (12.13)
  CFB at Day 6: Predose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: Predose | 0.5 (13.69) | 5.3 (13.08)
  CFB at Day 6: 0.25 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.25 H Postdose | 0.9 (12.24) | 6.3 (10.66)
  CFB at Day 6: 0.5 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.5 H Postdose | -0.4 (13.01) | 4.3 (12.23)
  CFB at Day 6: 1 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 1 H Postdose | 0.5 (12.91) | 4.7 (12.07)
  CFB at Day 6: 2 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 2 H Postdose | 2.6 (16.10) | 3.9 (14.18)
  CFB at Day 6: 12 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 12 H Postdose | -1.6 (11.10) | -0.2 (12.90)
  CFB at Day 7: Predose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: Predose | -1.0 (12.54) | 3.2 (11.76)
  CFB at Day 7: 0.25 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 0.25 H Postdose | 0.5 (14.43) | 1.8 (10.44)
  CFB at Day 7: 0.5 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 7: 0.5 H Postdose | 0.4 (14.04) | 2.4 (11.22)
  CFB at Day 7: 1 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 1 H Postdose | -0.7 (13.83) | 3.0 (11.35)
  CFB at Day 7: 2 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 2 H Postdose | 0.2 (15.73) | 0.8 (12.29)
  CFB at Day 7: 12 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 12 H Postdose | -3.4 (11.68) | 0.5 (12.11)
  CFB at Day 8: Predose: number analyzed (Participants) | 42 | 44
  CFB at Day 8: Predose | -0.8 (13.53) | 2.3 (12.96)
  CFB at Day 8: 1 H Postdose: number analyzed (Participants) | 41 | 44
  CFB at Day 8: 1 H Postdose | 1.6 (12.35) | 1.6 (14.27)
  CFB at Day 9: Predose: number analyzed (Participants) | 42 | 43
  CFB at Day 9: Predose | 0.5 (14.43) | 1.7 (11.76)
  CFB at Day 9: 1 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 9: 1 H Postdose | 2.8 (16.01) | -0.1 (14.04)
  CFB at Day 10: Predose: number analyzed (Participants) | 42 | 42
  CFB at Day 10: Predose | 0.0 (14.32) | -0.2 (12.08)
  CFB at Day 10: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 10: 1 H Postdose | 0.0 (16.48) | 0.2 (11.39)
  CFB at Day 11: Predose: number analyzed (Participants) | 41 | 41
  CFB at Day 11: Predose | -2.5 (16.30) | 4.4 (13.67)
  CFB at Day 11: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 11: 1 H Postdose | -3.6 (16.84) | 3.1 (13.00)
  CFB at Day 12: Predose: number analyzed (Participants) | 42 | 41
  CFB at Day 12: Predose | -2.2 (11.70) | 1.7 (12.05)
  CFB at Day 12: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 12: 1 H Postdose | 0.4 (11.64) | 2.0 (12.33)
  CFB at Day 13: Predose: number analyzed (Participants) | 39 | 40
  CFB at Day 13: Predose | -0.2 (13.23) | 1.4 (11.04)
  CFB at Day 13: 1 H Postdose: number analyzed (Participants) | 38 | 40
  CFB at Day 13: 1 H Postdose | 2.3 (13.27) | -0.2 (10.27)
  CFB at Day 14: Predose: number analyzed (Participants) | 41 | 41
  CFB at Day 14: Predose | -2.7 (14.09) | 2.4 (12.12)
  CFB at Day 14: 1 H Postdose: number analyzed (Participants) | 41 | 41
  CFB at Day 14: 1 H Postdose | 0.1 (14.54) | 2.9 (12.28)
  CFB at Day 15/ET: number analyzed (Participants) | 42 | 42
  CFB at Day 15/ET | 0.0 (14.14) | 5.8 (12.10)
  CFB at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  CFB at Follow-up Day 21 | 2.4 (13.92) | 6.2 (14.18)
  CFB at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  CFB at Follow-up Day 28 | 1.0 (13.83) | 5.5 (11.63)
  CFB at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  CFB at Follow-up Day 35 | 2.9 (15.58) | 7.8 (13.89)
  CFB at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  CFB at Follow-up Day 42 | -0.9 (15.02) | 8.3 (13.06)

97. Secondary Outcome: Change From Baseline (CFB) in Supine Diastolic Blood Pressure - Part B
Description: as for outcome 96
Time Frame: as for outcome 96
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
mmHg
  Baseline | 76.1 (10.10) | 75.2 (7.91)
  CFB at Day 1: 0.25 H Postdose | 0.8 (5.04) | 1.0 (7.26)
  CFB at Day 1: 0.5 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 1: 0.5 H Postdose | -0.1 (6.38) | 0.6 (7.09)
  CFB at Day 1: 1 H Postdose | 0.6 (6.40) | 0.3 (8.43)
  CFB at Day 1: 2 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 1: 2 H Postdose | 0.8 (7.32) | -0.2 (8.16)
  CFB at Day 1: 12 H Postdose | 1.7 (9.22) | 0.2 (7.98)
  CFB at Day 2: Predose | -0.5 (8.77) | 0.3 (7.21)
  CFB at Day 2: 0.25 H Postdose | 1.8 (8.23) | 0.8 (9.53)
  CFB at Day 2: 0.5 H Postdose | 1.6 (7.86) | 0.2 (9.30)
  CFB at Day 2: 1 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 2: 1 H Postdose | 2.2 (8.74) | -0.3 (7.97)
  CFB at Day 2: 2 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 2: 2 H Postdose | 0.8 (7.88) | 1.3 (10.10)
  CFB at Day 2: 12 H Postdose | -0.1 (7.15) | -0.5 (10.11)
  CFB at Day 3: Predose | 1.7 (7.35) | 0.1 (9.03)
  CFB at Day 3: 0.25 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 3: 0.25 H Postdose | 3.4 (8.57) | 0.6 (8.99)
  CFB at Day 3: 0.5 H Postdose | 3.0 (7.96) | -0.4 (9.78)
  CFB at Day 3: 1 H Postdose | 1.3 (8.29) | 0.0 (10.69)
  CFB at Day 3: 2 H Postdose | 1.3 (7.97) | -0.7 (10.86)
  CFB at Day 3: 12 H Postdose | -0.5 (7.14) | -1.7 (10.42)
  CFB at Day 4: Predose | 1.9 (9.49) | 1.5 (9.23)
  CFB at Day 4: 0.25 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 4: 0.25 H Postdose | 1.8 (9.53) | 0.3 (10.77)
  CFB at Day 4: 0.5 H Postdose | 0.9 (10.07) | 0.6 (10.50)
  CFB at Day 4: 1 H Postdose | 1.3 (9.83) | 0.4 (9.16)
  CFB at Day 4: 2 H Postdose | 0.3 (9.61) | 0.9 (10.25)
  CFB at Day 4: 12 H Postdose: number analyzed (Participants) | 43 | 44
  CFB at Day 4: 12 H Postdose | -0.1 (9.06) | -1.3 (9.86)
  CFB at Day 5: Predose | -1.5 (9.88) | 0.0 (8.94)
  CFB at Day 5: 0.25 H Postdose | 0.8 (9.99) | 0.1 (8.78)
  CFB at Day 5: 0.5 H Postdose | 1.3 (9.75) | 0.7 (9.12)
  CFB at Day 5: 1 H Postdose | 0.3 (9.49) | 0.3 (9.45)
  CFB at Day 5: 2 H Postdose | 0.8 (10.59) | -1.3 (9.92)
  CFB at Day 5: 12 H Postdose | 0.0 (9.72) | -1.3 (8.16)
  CFB at Day 6: Predose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: Predose | 1.4 (10.96) | 2.1 (9.04)
  CFB at Day 6: 0.25 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.25 H Postdose | 0.6 (10.12) | 2.7 (7.23)
  CFB at Day 6: 0.5 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.5 H Postdose | 1.3 (11.29) | 2.0 (8.85)
  CFB at Day 6: 1 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 1 H Postdose | 1.5 (9.74) | 0.9 (10.62)
  CFB at Day 6: 2 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 2 H Postdose | 2.9 (11.43) | 2.7 (11.00)
  CFB at Day 6: 12 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 12 H Postdose | -1.0 (8.30) | 0.4 (10.66)
  CFB at Day 7: Predose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: Predose | 0.0 (8.25) | 0.5 (8.78)
  CFB at Day 7: 0.25 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 0.25 H Postdose | 1.4 (10.33) | 1.5 (9.49)
  CFB at Day 7: 0.5 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 7: 0.5 H Postdose | 0.2 (10.10) | 2.3 (9.66)
  CFB at Day 7: 1 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 1 H Postdose | 0.1 (9.03) | 2.0 (9.14)
  CFB at Day 7: 2 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 2 H Postdose | 1.3 (11.20) | 2.1 (9.90)
  CFB at Day 7: 12 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 12 H Postdose | -0.4 (8.09) | 2.0 (10.00)
  CFB at Day 8: Predose: number analyzed (Participants) | 42 | 44
  CFB at Day 8: Predose | -0.1 (9.22) | 0.6 (7.76)
  CFB at Day 8: 1 H Postdose: number analyzed (Participants) | 41 | 44
  CFB at Day 8: 1 H Postdose | 0.9 (9.85) | 1.9 (9.92)
  CFB at Day 9: Predose: number analyzed (Participants) | 42 | 43
  CFB at Day 9: Predose | -0.1 (9.03) | 1.0 (8.18)
  CFB at Day 9: 1 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 9: 1 H Postdose | 0.4 (9.87) | -0.5 (10.18)
  CFB at Day 10: Predose: number analyzed (Participants) | 42 | 42
  CFB at Day 10: Predose | -0.5 (10.94) | 0.7 (10.23)
  CFB at Day 10: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 10: 1 H Postdose | 0.8 (9.97) | -0.5 (9.14)
  CFB at Day 11: Predose: number analyzed (Participants) | 41 | 41
  CFB at Day 11: Predose | -0.5 (11.53) | 0.6 (8.57)
  CFB at Day 11: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 11: 1 H Postdose | -2.1 (10.72) | 2.2 (9.15)
  CFB at Day 12: Predose: number analyzed (Participants) | 42 | 41
  CFB at Day 12: Predose | -1.0 (8.94) | 1.1 (7.98)
  CFB at Day 12: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 12: 1 H Postdose | -0.5 (9.17) | 0.0 (9.06)
  CFB at Day 13: Predose: number analyzed (Participants) | 39 | 40
  CFB at Day 13: Predose | 0.7 (11.64) | 0.5 (9.33)
  CFB at Day 13: 1 H Postdose: number analyzed (Participants) | 38 | 40
  CFB at Day 13: 1 H Postdose | 2.7 (10.42) | -0.1 (8.04)
  CFB at Day 14: Predose: number analyzed (Participants) | 41 | 41
  CFB at Day 14: Predose | -3.3 (9.52) | 1.6 (9.68)
  CFB at Day 14: 1 H Postdose: number analyzed (Participants) | 41 | 41
  CFB at Day 14: 1 H Postdose | 1.3 (9.96) | 2.1 (8.38)
  CFB at Day 15/ET: number analyzed (Participants) | 42 | 42
  CFB at Day 15/ET | 2.4 (10.00) | 4.1 (8.94)
  CFB at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  CFB at Follow-up Day 21 | 2.8 (9.47) | 3.9 (9.13)
  CFB at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  CFB at Follow-up Day 28 | 2.9 (9.73) | 3.4 (8.42)
  CFB at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  CFB at Follow-up Day 35 | -0.4 (11.31) | 4.3 (9.86)
  CFB at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  CFB at Follow-up Day 42 | 0.5 (10.98) | 4.6 (10.46)

98. Secondary Outcome: Change From Baseline (CFB) in Standing Systolic Blood Pressure - Part B
Description: as for outcome 96
Time Frame: as for outcome 96
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
mmHg
  Baseline | 125.9 (14.19) | 125.1 (14.00)
  CFB at Day 1: 0.25 H Postdose | 0.3 (8.48) | 0.8 (8.20)
  CFB at Day 1: 0.5 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 1: 0.5 H Postdose | -0.7 (8.88) | -1.7 (12.05)
  CFB at Day 1: 1 H Postdose | -0.7 (9.44) | -0.3 (12.46)
  CFB at Day 1: 2 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 1: 2 H Postdose | 0.2 (11.68) | -2.6 (10.56)
  CFB at Day 1: 12 H Postdose | -3.8 (13.79) | -4.5 (11.27)
  CFB at Day 2: Predose | -1.3 (9.20) | -0.3 (14.50)
  CFB at Day 2: 0.25 H Postdose | 1.1 (10.10) | -3.9 (15.98)
  CFB at Day 2: 0.5 H Postdose | -0.2 (10.16) | 0.4 (11.25)
  CFB at Day 2: 1 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 2: 1 H Postdose | -0.7 (11.01) | -1.8 (10.26)
  CFB at Day 2: 2 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 2: 2 H Postdose | -1.5 (11.38) | -2.7 (12.51)
  CFB at Day 2: 12 H Postdose | -5.5 (11.62) | -2.4 (12.67)
  CFB at Day 3: Predose | -3.0 (10.48) | 0.1 (13.03)
  CFB at Day 3: 0.25 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 3: 0.25 H Postdose | -0.1 (11.97) | -0.2 (12.78)
  CFB at Day 3: 0.5 H Postdose | -1.0 (12.26) | -2.1 (10.83)
  CFB at Day 3: 1 H Postdose | -0.7 (12.22) | -1.7 (13.34)
  CFB at Day 3: 2 H Postdose | -1.9 (11.45) | -1.4 (14.55)
  CFB at Day 3: 12 H Postdose | -4.3 (8.94) | -3.4 (11.42)
  CFB at Day 4: Predose | -1.2 (16.11) | -0.2 (10.91)
  CFB at Day 4: 0.25 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 4: 0.25 H Postdose | -1.3 (13.21) | 1.6 (11.83)
  CFB at Day 4: 0.5 H Postdose | -1.9 (10.60) | -0.4 (9.38)
  CFB at Day 4: 1 H Postdose | -3.1 (13.79) | 1.2 (10.70)
  CFB at Day 4: 2 H Postdose | -2.5 (13.34) | -1.8 (13.77)
  CFB at Day 4: 12 H Postdose: number analyzed (Participants) | 43 | 44
  CFB at Day 4: 12 H Postdose | -5.5 (13.01) | -4.5 (11.79)
  CFB at Day 5: Predose | -1.3 (12.57) | 1.3 (13.70)
  CFB at Day 5: 0.25 H Postdose | -0.5 (11.86) | 1.4 (13.22)
  CFB at Day 5: 0.5 H Postdose | -1.0 (11.04) | 1.3 (11.90)
  CFB at Day 5: 1 H Postdose | -2.4 (10.89) | 1.8 (11.63)
  CFB at Day 5: 2 H Postdose | -1.6 (13.12) | -2.2 (12.56)
  CFB at Day 5: 12 H Postdose | -5.5 (14.11) | -3.5 (13.36)
  CFB at Day 6: Predose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: Predose | -4.2 (14.69) | 3.2 (13.50)
  CFB at Day 6: 0.25 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.25 H Postdose | -1.6 (11.52) | 2.8 (12.65)
  CFB at Day 6: 0.5 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.5 H Postdose | -3.6 (12.23) | 1.7 (14.73)
  CFB at Day 6: 1 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 1 H Postdose | -1.9 (12.98) | 2.3 (14.61)
  CFB at Day 6: 2 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 2 H Postdose | -2.9 (12.89) | 2.2 (13.98)
  CFB at Day 6: 12 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 12 H Postdose | -5.7 (11.59) | -1.6 (13.21)
  CFB at Day 7: Predose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: Predose | -2.8 (14.48) | 4.3 (15.71)
  CFB at Day 7: 0.25 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 0.25 H Postdose | -2.6 (15.62) | 1.2 (13.56)
  CFB at Day 7: 0.5 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 7: 0.5 H Postdose | -2.6 (15.42) | 1.0 (11.22)
  CFB at Day 7: 1 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 1 H Postdose | -1.5 (15.18) | 1.5 (12.20)
  CFB at Day 7: 2 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 2 H Postdose | -2.9 (16.37) | -1.9 (10.48)
  CFB at Day 7: 12 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 12 H Postdose | -6.9 (12.84) | -3.2 (11.19)
  CFB at Day 8: Predose: number analyzed (Participants) | 42 | 44
  CFB at Day 8: Predose | -2.2 (13.37) | 1.9 (10.57)
  CFB at Day 8: 1 H Postdose: number analyzed (Participants) | 41 | 44
  CFB at Day 8: 1 H Postdose | -0.9 (10.82) | 0.6 (11.49)
  CFB at Day 9: Predose: number analyzed (Participants) | 42 | 43
  CFB at Day 9: Predose | -3.9 (13.94) | 1.5 (13.77)
  CFB at Day 9: 1 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 9: 1 H Postdose | -2.6 (14.50) | 0.8 (11.08)
  CFB at Day 10: Predose: number analyzed (Participants) | 42 | 42
  CFB at Day 10: Predose | -2.1 (16.07) | -0.7 (11.64)
  CFB at Day 10: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 10: 1 H Postdose | -1.2 (16.73) | -0.6 (16.41)
  CFB at Day 11: Predose: number analyzed (Participants) | 41 | 41
  CFB at Day 11: Predose | -4.8 (16.81) | 2.0 (17.24)
  CFB at Day 11: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 11: 1 H Postdose | -6.1 (16.18) | -0.1 (12.09)
  CFB at Day 12: Predose: number analyzed (Participants) | 42 | 41
  CFB at Day 12: Predose | -2.3 (13.70) | 2.4 (12.20)
  CFB at Day 12: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 12: 1 H Postdose | -2.5 (13.80) | 3.1 (14.10)
  CFB at Day 13: Predose: number analyzed (Participants) | 39 | 40
  CFB at Day 13: Predose | -4.1 (12.65) | 0.6 (11.69)
  CFB at Day 13: 1 H Postdose: number analyzed (Participants) | 38 | 40
  CFB at Day 13: 1 H Postdose | -1.6 (10.92) | 1.8 (11.83)
  CFB at Day 14: Predose: number analyzed (Participants) | 41 | 41
  CFB at Day 14: Predose | -4.4 (12.31) | 2.3 (11.60)
  CFB at Day 14: 1 H Postdose: number analyzed (Participants) | 41 | 41
  CFB at Day 14: 1 H Postdose | -1.2 (13.75) | 3.1 (13.90)
  CFB at Day 15/ET: number analyzed (Participants) | 42 | 42
  CFB at Day 15/ET | -2.8 (13.56) | -0.3 (11.32)
  CFB at Follow-up Day 21: number analyzed (Participants) | 38 | 45
  CFB at Follow-up Day 21 | -1.7 (14.21) | 1.7 (12.63)
  CFB at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  CFB at Follow-up Day 28 | -3.2 (12.13) | -1.9 (11.32)
  CFB at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  CFB at Follow-up Day 35 | -1.0 (13.00) | 2.6 (12.04)
  CFB at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  CFB at Follow-up Day 42 | -2.5 (14.02) | 0.8 (9.94)

99. Secondary Outcome: Change From Baseline (CFB) in Standing Diastolic Blood Pressure - Part B
Description: as for outcome 96
Time Frame: as for outcome 96
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
mmHg
  Baseline | 81.9 (9.32) | 80.1 (8.26)
  CFB at Day 1: 0.25 H Postdose | 1.0 (7.45) | 2.6 (6.06)
  CFB at Day 1: 0.5 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 1: 0.5 H Postdose | 0.7 (7.24) | 1.5 (7.30)
  CFB at Day 1: 1 H Postdose | -0.7 (7.75) | 0.8 (9.09)
  CFB at Day 1: 2 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 1: 2 H Postdose | 1.5 (7.41) | 0.4 (8.13)
  CFB at Day 1: 12 H Postdose | -0.1 (9.77) | 0.0 (7.96)
  CFB at Day 2: Predose | -1.5 (8.02) | 0.9 (8.07)
  CFB at Day 2: 0.25 H Postdose | 1.7 (6.86) | -1.2 (11.02)
  CFB at Day 2: 0.5 H Postdose | -0.2 (7.06) | 0.1 (8.21)
  CFB at Day 2: 1 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 2: 1 H Postdose | 0.8 (6.27) | -1.8 (8.47)
  CFB at Day 2: 2 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 2: 2 H Postdose | 0.0 (7.65) | 0.6 (8.05)
  CFB at Day 2: 12 H Postdose | -0.1 (7.87) | 1.1 (9.87)
  CFB at Day 3: Predose | -1.5 (7.83) | -0.4 (8.08)
  CFB at Day 3: 0.25 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 3: 0.25 H Postdose | 1.0 (8.05) | 0.4 (8.02)
  CFB at Day 3: 0.5 H Postdose | 1.3 (8.28) | -0.4 (8.11)
  CFB at Day 3: 1 H Postdose | 0.3 (8.17) | -0.7 (9.97)
  CFB at Day 3: 2 H Postdose | -0.4 (8.57) | -0.1 (10.06)
  CFB at Day 3: 12 H Postdose | -0.5 (6.72) | -0.4 (8.59)
  CFB at Day 4: Predose | -0.7 (9.70) | 2.4 (9.41)
  CFB at Day 4: 0.25 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 4: 0.25 H Postdose | 0.1 (9.23) | 2.2 (9.94)
  CFB at Day 4: 0.5 H Postdose | 0.3 (8.49) | 0.2 (9.36)
  CFB at Day 4: 1 H Postdose | 0.2 (8.06) | 0.3 (10.05)
  CFB at Day 4: 2 H Postdose | 0.6 (9.46) | -0.8 (10.84)
  CFB at Day 4: 12 H Postdose: number analyzed (Participants) | 43 | 44
  CFB at Day 4: 12 H Postdose | 0.0 (8.35) | -0.6 (9.38)
  CFB at Day 5: Predose | -1.1 (8.74) | -0.2 (8.65)
  CFB at Day 5: 0.25 H Postdose | 0.2 (8.12) | 0.6 (9.08)
  CFB at Day 5: 0.5 H Postdose | -1.1 (10.02) | 0.8 (9.19)
  CFB at Day 5: 1 H Postdose | -0.7 (8.56) | 1.3 (10.24)
  CFB at Day 5: 2 H Postdose | -1.3 (9.05) | -0.5 (9.62)
  CFB at Day 5: 12 H Postdose | -2.1 (8.54) | -0.3 (11.77)
  CFB at Day 6: Predose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: Predose | -0.9 (9.09) | 1.8 (11.79)
  CFB at Day 6: 0.25 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.25 H Postdose | -0.6 (10.69) | 3.0 (8.78)
  CFB at Day 6: 0.5 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.5 H Postdose | 0.0 (10.09) | 1.3 (12.70)
  CFB at Day 6: 1 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 1 H Postdose | 1.2 (9.07) | 2.3 (11.84)
  CFB at Day 6: 2 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 2 H Postdose | 1.0 (9.85) | 1.7 (9.93)
  CFB at Day 6: 12 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 12 H Postdose | -0.7 (7.21) | 1.6 (12.66)
  CFB at Day 7: Predose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: Predose | -0.6 (9.33) | -0.5 (8.27)
  CFB at Day 7: 0.25 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 0.25 H Postdose | 2.3 (8.89) | 0.2 (9.03)
  CFB at Day 7: 0.5 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 7: 0.5 H Postdose | 0.1 (11.03) | 0.7 (11.28)
  CFB at Day 7: 1 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 1 H Postdose | 0.8 (10.89) | 0.8 (10.27)
  CFB at Day 7: 2 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 2 H Postdose | -0.2 (9.69) | 0.6 (8.90)
  CFB at Day 7: 12 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 12 H Postdose | -2.7 (7.17) | 0.4 (9.28)
  CFB at Day 8: Predose: number analyzed (Participants) | 42 | 44
  CFB at Day 8: Predose | -0.3 (9.52) | 0.7 (9.77)
  CFB at Day 8: 1 H Postdose: number analyzed (Participants) | 41 | 44
  CFB at Day 8: 1 H Postdose | -0.4 (7.18) | 2.3 (8.57)
  CFB at Day 9: Predose: number analyzed (Participants) | 42 | 43
  CFB at Day 9: Predose | -1.5 (9.64) | 0.5 (7.27)
  CFB at Day 9: 1 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 9: 1 H Postdose | 0.6 (9.66) | 1.7 (8.83)
  CFB at Day 10: Predose: number analyzed (Participants) | 42 | 42
  CFB at Day 10: Predose | 0.2 (8.57) | 2.0 (10.21)
  CFB at Day 10: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 10: 1 H Postdose | 0.0 (10.47) | 1.7 (12.59)
  CFB at Day 11: Predose: number analyzed (Participants) | 41 | 41
  CFB at Day 11: Predose | -2.3 (12.73) | 1.6 (13.81)
  CFB at Day 11: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 11: 1 H Postdose | -4.3 (12.66) | 0.0 (10.73)
  CFB at Day 12: Predose: number analyzed (Participants) | 42 | 41
  CFB at Day 12: Predose | 2.1 (9.35) | 1.2 (10.41)
  CFB at Day 12: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 12: 1 H Postdose | -1.4 (11.63) | 2.0 (12.93)
  CFB at Day 13: Predose: number analyzed (Participants) | 39 | 40
  CFB at Day 13: Predose | 0.0 (9.92) | 2.1 (8.87)
  CFB at Day 13: 1 H Postdose: number analyzed (Participants) | 38 | 40
  CFB at Day 13: 1 H Postdose | 0.7 (7.60) | -0.8 (9.39)
  CFB at Day 14: Predose: number analyzed (Participants) | 41 | 41
  CFB at Day 14: Predose | -2.8 (9.26) | 2.5 (9.59)
  CFB at Day 14: 1 H Postdose: number analyzed (Participants) | 41 | 41
  CFB at Day 14: 1 H Postdose | 1.2 (10.72) | 1.8 (8.36)
  CFB at Day 15/ET: number analyzed (Participants) | 42 | 42
  CFB at Day 15/ET | 0.8 (9.09) | 1.5 (8.41)
  CFB at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  CFB at Follow-up Day 21 | 1.7 (8.65) | 2.3 (8.58)
  CFB at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  CFB at Follow-up Day 28 | -0.3 (7.05) | 1.9 (9.00)
  CFB at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  CFB at Follow-up Day 35 | -0.4 (8.34) | 3.5 (9.60)
  CFB at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  CFB at Follow-up Day 42 | 0.3 (9.61) | 2.5 (7.69)

100. Secondary Outcome: Change From Baseline (CFB) in Heart Rate - Part B
Description: as for outcome 96
Time Frame: as for outcome 96
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
beats/min
  Baseline | 74.3 (12.80) | 76.8 (12.33)
  CFB at Day 1: 0.25 H Postdose | -1.9 (9.96) | -2.8 (8.50)
  CFB at Day 1: 0.5 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 1: 0.5 H Postdose | -2.1 (10.77) | -2.5 (9.26)
  CFB at Day 1: 1 H Postdose | -1.8 (11.14) | -4.6 (9.13)
  CFB at Day 1: 2 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 1: 2 H Postdose | -0.8 (12.63) | -1.1 (9.30)
  CFB at Day 1: 12 H Postdose | -1.0 (11.53) | -4.3 (12.18)
  CFB at Day 2: Predose | 2.5 (11.80) | -1.8 (11.47)
  CFB at Day 2: 0.25 H Postdose | -0.2 (10.75) | -1.8 (11.79)
  CFB at Day 2: 0.5 H Postdose | -1.0 (10.98) | -2.4 (10.50)
  CFB at Day 2: 1 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 2: 1 H Postdose | -0.2 (11.79) | -3.0 (11.15)
  CFB at Day 2: 2 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 2: 2 H Postdose | -1.7 (8.50) | -1.3 (11.50)
  CFB at Day 2: 12 H Postdose | -2.3 (11.09) | -4.0 (11.51)
  CFB at Day 3: Predose | 2.5 (12.40) | -0.7 (13.35)
  CFB at Day 3: 0.25 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 3: 0.25 H Postdose | 0.0 (9.56) | -1.4 (10.93)
  CFB at Day 3: 0.5 H Postdose | -0.5 (10.82) | -1.8 (11.57)
  CFB at Day 3: 1 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 3: 1 H Postdose | 0.8 (10.24) | -1.2 (11.03)
  CFB at Day 3: 2 H Postdose | 0.4 (12.45) | -0.5 (11.19)
  CFB at Day 3: 12 H Postdose | -3.0 (10.46) | -4.2 (11.62)
  CFB at Day 4: Predose | 4.9 (10.28) | 2.0 (10.30)
  CFB at Day 4: 0.25 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 4: 0.25 H Postdose | 2.8 (9.06) | 3.5 (15.13)
  CFB at Day 4: 0.5 H Postdose | 1.9 (10.43) | -1.4 (10.73)
  CFB at Day 4: 1 H Postdose | 1.4 (9.75) | -0.8 (10.63)
  CFB at Day 4: 2 H Postdose | 1.1 (11.94) | 1.6 (12.66)
  CFB at Day 4: 12 H Postdose: number analyzed (Participants) | 43 | 44
  CFB at Day 4: 12 H Postdose | -0.6 (11.36) | -3.6 (11.76)
  CFB at Day 5: Predose | 4.3 (11.14) | 1.9 (9.70)
  CFB at Day 5: 0.25 H Postdose | 2.4 (11.59) | 0.3 (12.44)
  CFB at Day 5: 0.5 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 5: 0.5 H Postdose | 3.7 (11.81) | 0.0 (9.57)
  CFB at Day 5: 1 H Postdose | 0.6 (10.52) | 2.0 (12.34)
  CFB at Day 5: 2 H Postdose | 1.5 (11.68) | 2.5 (10.62)
  CFB at Day 5: 12 H Postdose | -0.2 (14.80) | -1.4 (12.45)
  CFB at Day 6: Predose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: Predose | 4.7 (10.64) | 3.9 (8.00)
  CFB at Day 6: 0.25 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.25 H Postdose | 3.1 (11.30) | 0.7 (9.81)
  CFB at Day 6: 0.5 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.5 H Postdose | 2.5 (11.80) | 0.4 (10.44)
  CFB at Day 6: 1 H Postdose: number analyzed (Participants) | 42 | 45
  CFB at Day 6: 1 H Postdose | 3.2 (12.71) | 0.4 (8.54)
  CFB at Day 6: 2 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 2 H Postdose | 2.6 (9.70) | 0.5 (11.53)
  CFB at Day 6: 12 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 12 H Postdose | 1.4 (12.65) | -2.3 (12.57)
  CFB at Day 7: Predose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: Predose | 3.7 (10.26) | 3.0 (11.63)
  CFB at Day 7: 0.25 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 0.25 H Postdose | 3.9 (12.00) | 1.5 (11.16)
  CFB at Day 7: 0.5 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 7: 0.5 H Postdose | 3.7 (12.25) | -0.4 (11.19)
  CFB at Day 7: 1 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 1 H Postdose | 5.5 (13.30) | 1.4 (11.25)
  CFB at Day 7: 2 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 2 H Postdose | 0.9 (10.64) | 2.2 (13.04)
  CFB at Day 7: 12 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 12 H Postdose | -0.4 (11.53) | -1.3 (13.75)
  CFB at Day 8: Predose: number analyzed (Participants) | 42 | 44
  CFB at Day 8: Predose | 10.1 (14.90) | 6.9 (14.46)
  CFB at Day 8: 1 H Postdose: number analyzed (Participants) | 41 | 44
  CFB at Day 8: 1 H Postdose | 8.5 (12.78) | 6.9 (12.02)
  CFB at Day 9: Predose: number analyzed (Participants) | 42 | 43
  CFB at Day 9: Predose | 7.7 (10.64) | 7.5 (12.00)
  CFB at Day 9: 1 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 9: 1 H Postdose | 5.9 (10.94) | 4.4 (12.05)
  CFB at Day 10: Predose: number analyzed (Participants) | 42 | 42
  CFB at Day 10: Predose | 6.4 (11.40) | 8.9 (13.59)
  CFB at Day 10: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 10: 1 H Postdose | 4.0 (12.11) | 6.1 (13.09)
  CFB at Day 11: Predose: number analyzed (Participants) | 41 | 41
  CFB at Day 11: Predose | 6.2 (15.10) | 4.6 (11.26)
  CFB at Day 11: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 11: 1 H Postdose | 4.3 (14.76) | 4.5 (11.22)
  CFB at Day 12: Predose: number analyzed (Participants) | 42 | 41
  CFB at Day 12: Predose | 4.4 (11.99) | 3.8 (13.85)
  CFB at Day 12: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 12: 1 H Postdose | 4.8 (13.56) | 2.1 (13.19)
  CFB at Day 13: Predose: number analyzed (Participants) | 39 | 40
  CFB at Day 13: Predose | 3.1 (12.72) | 4.1 (11.22)
  CFB at Day 13: 1 H Postdose: number analyzed (Participants) | 38 | 40
  CFB at Day 13: 1 H Postdose | 2.9 (10.46) | 5.0 (11.53)
  CFB at Day 14: Predose: number analyzed (Participants) | 41 | 41
  CFB at Day 14: Predose | 6.4 (12.18) | 4.6 (10.91)
  CFB at Day 14: 1 H Postdose: number analyzed (Participants) | 41 | 41
  CFB at Day 14: 1 H Postdose | 3.6 (10.21) | 2.8 (9.96)
  CFB at Day 15/ET: number analyzed (Participants) | 42 | 42
  CFB at Day 15/ET | -1.6 (12.73) | -0.1 (10.78)
  CFB at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  CFB at Follow-up Day 21 | 0.1 (10.32) | -5.9 (10.54)
  CFB at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  CFB at Follow-up Day 28 | -0.5 (13.06) | -5.3 (15.54)
  CFB at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  CFB at Follow-up Day 35 | -3.8 (11.13) | -3.9 (13.47)
  CFB at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  CFB at Follow-up Day 42 | -3.7 (11.93) | -6.0 (12.73)

101. Secondary Outcome: Change From Baseline (CFB) in Respiratory Rate - Part B
Description: as for outcome 96
Time Frame: as for outcome 96
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
breaths/min
  Baseline | 16.7 (1.72) | 16.8 (1.41)
  CFB at Day 1: 0.25 H Postdose | 0.2 (1.24) | -0.1 (1.05)
  CFB at Day 1: 0.5 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 1: 0.5 H Postdose | 0.4 (1.08) | 0.0 (0.71)
  CFB at Day 1: 1 H Postdose | 0.3 (1.76) | 0.1 (1.00)
  CFB at Day 1: 2 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 1: 2 H Postdose | 0.4 (1.66) | -0.1 (0.98)
  CFB at Day 1: 12 H Postdose | -0.3 (1.99) | 0.2 (1.65)
  CFB at Day 2: Predose | -0.1 (2.36) | 0.0 (1.48)
  CFB at Day 2: 0.25 H Postdose | 0.0 (1.86) | 0.0 (1.41)
  CFB at Day 2: 0.5 H Postdose | 0.4 (1.94) | 0.1 (1.59)
  CFB at Day 2: 1 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 2: 1 H Postdose | 0.1 (1.89) | -0.2 (1.40)
  CFB at Day 2: 2 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 2: 2 H Postdose | 0.3 (1.88) | 0.0 (1.45)
  CFB at Day 2: 12 H Postdose | -0.2 (2.14) | 0.0 (1.83)
  CFB at Day 3: Predose | 0.0 (1.88) | 0.1 (2.07)
  CFB at Day 3: 0.25 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 3: 0.25 H Postdose | 0.0 (1.87) | 0.0 (1.52)
  CFB at Day 3: 0.5 H Postdose | 0.0 (2.00) | 0.0 (1.45)
  CFB at Day 3: 1 H Postdose | 0.2 (2.14) | 0.2 (1.51)
  CFB at Day 3: 2 H Postdose | 0.4 (1.94) | 0.3 (1.63)
  CFB at Day 3: 12 H Postdose | 0.0 (2.33) | 0.2 (1.82)
  CFB at Day 4: Predose | 0.3 (1.92) | -0.1 (1.75)
  CFB at Day 4: 0.25 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 4: 0.25 H Postdose | 0.4 (1.94) | -0.1 (2.03)
  CFB at Day 4: 0.5 H Postdose | 0.2 (2.12) | 0.2 (1.90)
  CFB at Day 4: 1 H Postdose | 0.3 (1.71) | 0.4 (2.01)
  CFB at Day 4: 2 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 4: 2 H Postdose | 0.2 (1.80) | 0.1 (1.90)
  CFB at Day 4: 12 H Postdose: number analyzed (Participants) | 43 | 44
  CFB at Day 4: 12 H Postdose | 0.2 (2.46) | 0.2 (2.43)
  CFB at Day 5: Predose | 0.3 (2.23) | 0.0 (1.82)
  CFB at Day 5: 0.25 H Postdose | 0.0 (2.10) | 0.1 (1.87)
  CFB at Day 5: 0.5 H Postdose | 0.1 (2.10) | 0.0 (1.82)
  CFB at Day 5: 1 H Postdose | 0.2 (2.16) | 0.2 (1.66)
  CFB at Day 5: 2 H Postdose | 0.2 (2.13) | 0.1 (1.90)
  CFB at Day 5: 12 H Postdose | 0.1 (2.24) | 0.4 (2.01)
  CFB at Day 6: Predose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: Predose | 0.5 (2.02) | 0.6 (2.56)
  CFB at Day 6: 0.25 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.25 H Postdose | 0.6 (2.11) | 0.2 (1.85)
  CFB at Day 6: 0.5 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.5 H Postdose | 0.3 (1.95) | 0.2 (1.81)
  CFB at Day 6: 1 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 1 H Postdose | 0.3 (1.71) | 0.2 (2.00)
  CFB at Day 6: 2 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 2 H Postdose | 0.5 (2.18) | 0.4 (1.84)
  CFB at Day 6: 12 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 12 H Postdose | 0.1 (1.92) | 1.4 (8.64)
  CFB at Day 7: Predose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: Predose | 0.8 (2.70) | 0.7 (1.91)
  CFB at Day 7: 0.25 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 0.25 H Postdose | 1.0 (2.71) | 0.0 (2.01)
  CFB at Day 7: 0.5 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 7: 0.5 H Postdose | 1.1 (2.28) | 0.3 (1.48)
  CFB at Day 7: 1 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 1 H Postdose | 0.8 (2.48) | 0.4 (1.99)
  CFB at Day 7: 2 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 2 H Postdose | 0.5 (2.26) | 0.5 (1.91)
  CFB at Day 7: 12 H Postdose: number analyzed (Participants) | 41 | 44
  CFB at Day 7: 12 H Postdose | -0.2 (1.96) | 0.1 (1.73)
  CFB at Day 8: Predose: number analyzed (Participants) | 42 | 44
  CFB at Day 8: Predose | 0.5 (2.05) | 0.4 (1.88)
  CFB at Day 8: 1 H Postdose: number analyzed (Participants) | 41 | 44
  CFB at Day 8: 1 H Postdose | 1.0 (2.26) | 0.4 (1.65)
  CFB at Day 9: Predose: number analyzed (Participants) | 42 | 43
  CFB at Day 9: Predose | 0.7 (2.22) | 0.3 (1.81)
  CFB at Day 9: 1 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 9: 1 H Postdose | 0.4 (1.91) | 0.1 (1.82)
  CFB at Day 10: Predose: number analyzed (Participants) | 42 | 42
  CFB at Day 10: Predose | 0.5 (1.60) | 0.5 (2.05)
  CFB at Day 10: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 10: 1 H Postdose | 0.5 (2.21) | 0.6 (1.67)
  CFB at Day 11: Predose: number analyzed (Participants) | 41 | 41
  CFB at Day 11: Predose | 0.3 (1.97) | 0.5 (1.99)
  CFB at Day 11: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 11: 1 H Postdose | 0.3 (2.18) | 0.3 (2.04)
  CFB at Day 12: Predose: number analyzed (Participants) | 42 | 41
  CFB at Day 12: Predose | 0.7 (2.27) | 0.5 (1.93)
  CFB at Day 12: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 12: 1 H Postdose | 0.6 (2.05) | 0.4 (1.83)
  CFB at Day 13: Predose: number analyzed (Participants) | 39 | 40
  CFB at Day 13: Predose | 1.0 (1.94) | 0.4 (1.96)
  CFB at Day 13: 1 H Postdose: number analyzed (Participants) | 38 | 40
  CFB at Day 13: 1 H Postdose | 1.0 (2.18) | 0.3 (1.79)
  CFB at Day 14: Predose: number analyzed (Participants) | 41 | 41
  CFB at Day 14: Predose | 0.8 (2.08) | 0.1 (2.89)
  CFB at Day 14: 1 H Postdose: number analyzed (Participants) | 41 | 41
  CFB at Day 14: 1 H Postdose | 0.9 (1.98) | 0.4 (1.61)
  CFB at Day 15/ET: number analyzed (Participants) | 41 | 42
  CFB at Day 15/ET | 1.2 (8.39) | -0.4 (1.59)
  CFB at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  CFB at Follow-up Day 21 | 0.1 (2.21) | 0.2 (1.70)
  CFB at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  CFB at Follow-up Day 28 | 0.0 (2.15) | 0.0 (1.88)
  CFB at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  CFB at Follow-up Day 35 | 0.0 (2.40) | 0.1 (1.64)
  CFB at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  CFB at Follow-up Day 42 | -0.2 (2.48) | 0.1 (1.50)

102. Secondary Outcome: Change From Baseline (CFB) in Oral Temperature - Part B
Description: as for outcome 96
Time Frame: as for outcome 96
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
degrees C
  Baseline | 36.72 (0.298) | 36.72 (0.324)
  CFB at Day 1: 0.25 H Postdose | 0.03 (0.309) | 0.03 (0.374)
  CFB at Day 1: 0.5 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 1: 0.5 H Postdose | 0.03 (0.315) | 0.05 (0.367)
  CFB at Day 1: 1 H Postdose | 0.05 (0.311) | -0.02 (0.414)
  CFB at Day 1: 2 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 1: 2 H Postdose | 0.03 (0.360) | -0.05 (0.384)
  CFB at Day 1: 12 H Postdose | -0.09 (0.328) | -0.10 (0.382)
  CFB at Day 2: Predose | -0.04 (0.250) | -0.01 (0.283)
  CFB at Day 2: 0.25 H Postdose | -0.03 (0.330) | -0.04 (0.421)
  CFB at Day 2: 0.5 H Postdose | 0.01 (0.284) | -0.06 (0.539)
  CFB at Day 2: 1 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 2: 1 H Postdose | -0.05 (0.242) | -0.02 (0.371)
  CFB at Day 2: 2 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 2: 2 H Postdose | -0.06 (0.257) | -0.05 (0.327)
  CFB at Day 2: 12 H Postdose | -0.13 (0.307) | -0.06 (0.397)
  CFB at Day 3: Predose | -0.03 (0.403) | -0.02 (0.321)
  CFB at Day 3: 0.25 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 3: 0.25 H Postdose | -0.06 (0.417) | -0.05 (0.332)
  CFB at Day 3: 0.5 H Postdose | 0.08 (0.408) | -0.03 (0.361)
  CFB at Day 3: 1 H Postdose | 0.03 (0.430) | -0.04 (0.330)
  CFB at Day 3: 2 H Postdose | -0.03 (0.353) | 0.00 (0.380)
  CFB at Day 3: 12 H Postdose | -0.13 (0.269) | -0.08 (0.339)
  CFB at Day 4: Predose | -0.14 (0.421) | -0.03 (0.348)
  CFB at Day 4: 0.25 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 4: 0.25 H Postdose | -0.07 (0.335) | -0.04 (0.343)
  CFB at Day 4: 0.5 H Postdose | -0.03 (0.414) | -0.04 (0.333)
  CFB at Day 4: 1 H Postdose | -0.11 (0.310) | 0.01 (0.392)
  CFB at Day 4: 2 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 4: 2 H Postdose | -0.02 (0.458) | -0.04 (0.367)
  CFB at Day 4: 12 H Postdose: number analyzed (Participants) | 43 | 44
  CFB at Day 4: 12 H Postdose | -0.07 (0.370) | 0.01 (0.586)
  CFB at Day 5: Predose | 0.01 (0.414) | -0.01 (0.343)
  CFB at Day 5: 0.25 H Postdose | 0.01 (0.376) | -0.03 (0.349)
  CFB at Day 5: 0.5 H Postdose | 0.07 (0.359) | -0.08 (0.359)
  CFB at Day 5: 1 H Postdose | -0.01 (0.345) | -0.01 (0.354)
  CFB at Day 5: 2 H Postdose | -0.04 (0.301) | -0.08 (0.349)
  CFB at Day 5: 12 H Postdose | -0.09 (0.322) | -0.12 (0.277)
  CFB at Day 6: Predose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: Predose | 0.06 (0.381) | 0.07 (0.428)
  CFB at Day 6: 0.25 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.25 H Postdose | 0.01 (0.381) | 0.04 (0.523)
  CFB at Day 6: 0.5 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.5 H Postdose | 0.04 (0.401) | 0.00 (0.376)
  CFB at Day 6: 1 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 1 H Postdose | 0.04 (0.373) | -0.05 (0.392)
  CFB at Day 6: 2 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 2 H Postdose | 0.05 (0.405) | 0.01 (0.452)
  CFB at Day 6: 12 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 12 H Postdose | -0.10 (0.341) | -0.10 (0.366)
  CFB at Day 7: Predose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: Predose | 0.02 (0.386) | 0.02 (0.430)
  CFB at Day 7: 0.25 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 0.25 H Postdose | -0.04 (0.341) | -0.02 (0.358)
  CFB at Day 7: 0.5 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 7: 0.5 H Postdose | 0.05 (0.402) | 0.00 (0.390)
  CFB at Day 7: 1 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 1 H Postdose | 0.05 (0.388) | 0.06 (0.444)
  CFB at Day 7: 2 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 2 H Postdose | 0.01 (0.489) | 0.01 (0.387)
  CFB at Day 7: 12 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 7: 12 H Postdose | -0.06 (0.350) | -0.10 (0.353)
  CFB at Day 8: Predose: number analyzed (Participants) | 42 | 44
  CFB at Day 8: Predose | 0.05 (0.350) | 0.02 (0.388)
  CFB at Day 8: 1 H Postdose: number analyzed (Participants) | 41 | 44
  CFB at Day 8: 1 H Postdose | 0.11 (0.372) | 0.02 (0.355)
  CFB at Day 9: Predose: number analyzed (Participants) | 42 | 43
  CFB at Day 9: Predose | 0.04 (0.421) | 0.04 (0.414)
  CFB at Day 9: 1 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 9: 1 H Postdose | 0.09 (0.404) | 0.05 (0.389)
  CFB at Day 10: Predose: number analyzed (Participants) | 42 | 42
  CFB at Day 10: Predose | -0.01 (0.409) | -0.04 (0.402)
  CFB at Day 10: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 10: 1 H Postdose | 0.06 (0.454) | 0.01 (0.412)
  CFB at Day 11: Predose: number analyzed (Participants) | 41 | 41
  CFB at Day 11: Predose | -0.02 (0.536) | -0.06 (0.382)
  CFB at Day 11: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 11: 1 H Postdose | -0.05 (0.374) | -0.10 (0.387)
  CFB at Day 12: Predose: number analyzed (Participants) | 42 | 41
  CFB at Day 12: Predose | 0.01 (0.422) | -0.06 (0.358)
  CFB at Day 12: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 12: 1 H Postdose | 0.01 (0.364) | -0.12 (0.359)
  CFB at Day 13: Predose: number analyzed (Participants) | 39 | 40
  CFB at Day 13: Predose | -0.01 (0.348) | 0.04 (0.353)
  CFB at Day 13: 1 H Postdose: number analyzed (Participants) | 38 | 40
  CFB at Day 13: 1 H Postdose | 0.03 (0.449) | 0.02 (0.418)
  CFB at Day 14: Predose: number analyzed (Participants) | 41 | 41
  CFB at Day 14: Predose | 0.06 (0.416) | -0.01 (0.315)
  CFB at Day 14: 1 H Postdose: number analyzed (Participants) | 41 | 41
  CFB at Day 14: 1 H Postdose | 0.06 (0.378) | 0.00 (0.419)
  CFB at Day 15/ET: number analyzed (Participants) | 42 | 42
  CFB at Day 15/ET | -0.09 (0.320) | -0.03 (0.391)
  CFB at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  CFB at Follow-up Day 21 | -0.12 (0.281) | -0.03 (0.314)
  CFB at Follow-up Day 28: number analyzed (Participants) | 39 | 42
  CFB at Follow-up Day 28 | -0.04 (0.321) | -0.07 (0.352)
  CFB at Follow-up Day 35: number analyzed (Participants) | 40 | 41
  CFB at Follow-up Day 35 | -0.05 (0.324) | -0.05 (0.359)
  CFB at Follow-up Day 42: number analyzed (Participants) | 39 | 42
  CFB at Follow-up Day 42 | 0.03 (0.338) | -0.08 (0.389)

103. Secondary Outcome: Change From Baseline (CFB) in Oxygen Saturation - Part B
Description: as for outcome 96
Time Frame: as for outcome 43
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
percentage of oxygen saturation
  Baseline | 97.95 (1.509) | 98.02 (1.485)
  CFB at Day 1: 0.25 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 1: 0.25 H Postdose | -0.11 (1.768) | -0.02 (1.502)
  CFB at Day 1: 0.5 H Postdose: number analyzed (Participants) | 43 | 44
  CFB at Day 1: 0.5 H Postdose | 0.12 (1.384) | 0.00 (1.510)
  CFB at Day 1: 1 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 1: 1 H Postdose | 0.02 (1.470) | -0.39 (1.401)
  CFB at Day 1: 2 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 1: 2 H Postdose | 0.11 (1.513) | -0.32 (1.459)
  CFB at Day 1: 12 H Postdose | 0.09 (1.789) | -0.24 (1.827)
  CFB at Day 2: Predose | -0.23 (1.939) | -0.29 (1.576)
  CFB at Day 2: 0.25 H Postdose | -0.23 (1.915) | -0.22 (1.475)
  CFB at Day 2: 0.5 H Postdose | -0.20 (2.041) | -0.44 (1.726)
  CFB at Day 2: 1 H Postdose | -0.09 (1.902) | -0.38 (1.762)
  CFB at Day 2: 2 H Postdose | -0.11 (1.907) | -0.36 (1.654)
  CFB at Day 2: 12 H Postdose | -0.34 (5.278) | -0.47 (2.599)
  CFB at Day 3: Predose | -0.32 (1.827) | -0.29 (1.766)
  CFB at Day 3: 0.25 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 3: 0.25 H Postdose | -0.09 (1.789) | -0.32 (1.695)
  CFB at Day 3: 0.5 H Postdose | -0.11 (1.742) | -0.42 (1.712)
  CFB at Day 3: 1 H Postdose | -0.27 (1.860) | -0.44 (1.902)
  CFB at Day 3: 2 H Postdose | -0.32 (2.340) | -0.78 (1.894)
  CFB at Day 3: 12 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 3: 12 H Postdose | 0.14 (1.959) | -0.24 (1.824)
  CFB at Day 4: Predose | -0.20 (1.579) | -0.27 (1.643)
  CFB at Day 4: 0.25 H Postdose | 0.09 (1.709) | -0.24 (1.667)
  CFB at Day 4: 0.5 H Postdose | -0.20 (1.720) | -0.33 (1.581)
  CFB at Day 4: 1 H Postdose | -0.41 (1.933) | -0.29 (1.646)
  CFB at Day 4: 2 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 4: 2 H Postdose | -0.70 (2.018) | -1.16 (2.667)
  CFB at Day 4: 12 H Postdose | 0.00 (2.000) | -1.31 (4.986)
  CFB at Day 5: Predose | -0.16 (1.539) | -0.36 (2.165)
  CFB at Day 5: 0.25 H Postdose | 0.20 (1.407) | -0.58 (2.179)
  CFB at Day 5: 0.5 H Postdose | -0.09 (1.736) | -0.49 (2.564)
  CFB at Day 5: 1 H Postdose: number analyzed (Participants) | 44 | 44
  CFB at Day 5: 1 H Postdose | -0.07 (2.161) | -0.61 (2.895)
  CFB at Day 5: 2 H Postdose | -0.05 (1.765) | -0.62 (2.338)
  CFB at Day 5: 12 H Postdose | 0.11 (1.979) | 0.09 (1.856)
  CFB at Day 6: Predose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: Predose | -0.02 (1.933) | -0.13 (1.424)
  CFB at Day 6: 0.25 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.25 H Postdose | 0.09 (1.525) | -0.02 (1.631)
  CFB at Day 6: 0.5 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.5 H Postdose | 0.12 (1.749) | 0.16 (1.147)
  CFB at Day 6: 1 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 1 H Postdose | 0.09 (1.849) | -0.22 (1.820)
  CFB at Day 6: 2 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 2 H Postdose | -0.07 (1.920) | 0.16 (1.492)
  CFB at Day 6: 12 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 12 H Postdose | 0.37 (1.852) | 0.02 (1.672)
  CFB at Day 7: Predose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: Predose | -0.31 (1.932) | -0.16 (1.656)
  CFB at Day 7: 0.25 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 0.25 H Postdose | 0.05 (2.129) | 0.07 (1.516)
  CFB at Day 7: 0.5 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 0.5 H Postdose | -0.21 (2.007) | -0.16 (1.928)
  CFB at Day 7: 1 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 1 H Postdose | -0.05 (1.987) | -0.45 (1.663)
  CFB at Day 7: 2 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 2 H Postdose | 0.17 (1.987) | -0.55 (2.757)
  CFB at Day 7: 12 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 12 H Postdose | 0.31 (2.089) | -0.11 (1.833)
  CFB at Day 8: Predose: number analyzed (Participants) | 38 | 42
  CFB at Day 8: Predose | 0.21 (1.510) | -0.26 (1.499)
  CFB at Day 8: 1 H Postdose: number analyzed (Participants) | 36 | 36
  CFB at Day 8: 1 H Postdose | 0.08 (2.005) | -0.67 (1.789)

104. Secondary Outcome: Change From Baseline in QT Interval - Part B
Description: ECG measures included QT interval, QTcF interval, ECG mean heart rate, RR interval, PR interval, and QRS duration. The analysis was performed in participants included in Part B of the study.
Time Frame: Baseline, Days 1, 2, 7, 14 and follow-up Day 21
Population: as for outcome 58
Measure: Median (Full Range); unit: msec
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
msec
  Baseline | 403.5 [332 to 498] | 398.0 [343 to 461]
  Change from Baseline at Day 1: number analyzed (Participants) | 44 | 44
  Change from Baseline at Day 1 | -9.0 [-85 to 40] | -7.0 [-52 to 71]
  Change from Baseline at Day 2: number analyzed (Participants) | 44 | 44
  Change from Baseline at Day 2 | -12.0 [-81 to 30] | -15.0 [-62 to 55]
  Change from Baseline at Day 7: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 7 | -22.0 [-81 to 19] | -25.5 [-95 to 58]
  Change from Baseline at Day 14: number analyzed (Participants) | 41 | 40
  Change from Baseline at Day 14 | -23.0 [-86 to 26] | -25.5 [-109 to 55]
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -12.5 [-59 to 52] | -7.5 [-412 to 66]

105. Secondary Outcome: Change From Baseline in QTcF Interval - Part B
Description: as for outcome 104
Time Frame: Baseline, Days 1, 2, 7, 14 and follow-up Day 21
Population: as for outcome 58
Measure: Median (Full Range); unit: msec
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
msec
  Baseline | 406.0 [347 to 450] | 410.0 [365 to 464]
  Change from Baseline at Day 1: number analyzed (Participants) | 44 | 44
  Change from Baseline at Day 1 | 0.0 [-46 to 30] | -2.0 [-24 to 73]
  Change from Baseline at Day 2: number analyzed (Participants) | 44 | 44
  Change from Baseline at Day 2 | -2.5 [-41 to 24] | -4.0 [-42 to 38]
  Change from Baseline at Day 7: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 7 | -5.0 [-35 to 35] | -7.5 [-64 to 37]
  Change from Baseline at Day 14: number analyzed (Participants) | 41 | 40
  Change from Baseline at Day 14 | -8.0 [-37 to 35] | -3.0 [-61 to 51]
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -2.0 [-36 to 33] | 0.5 [-435 to 33]

106. Secondary Outcome: Change From Baseline in ECG Mean Heart Rate - Part B
Description: as for outcome 104
Time Frame: Baseline, Days 1, 2, 7, 14 and follow-up Day 21
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
beats/min
  Baseline | 65.0 (11.17) | 64.8 (10.06)
  Change from Baseline at Day 1: number analyzed (Participants) | 44 | 44
  Change from Baseline at Day 1 | 3.2 (8.74) | 4.5 (10.25)
  Change from Baseline at Day 2: number analyzed (Participants) | 44 | 44
  Change from Baseline at Day 2 | 6.0 (9.58) | 4.7 (10.91)
  Change from Baseline at Day 7: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 7 | 8.3 (9.67) | 7.2 (10.37)
  Change from Baseline at Day 14: number analyzed (Participants) | 41 | 40
  Change from Baseline at Day 14 | 7.1 (9.22) | 11.0 (11.23)
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | 5.1 (9.22) | -0.5 (15.10)

107. Secondary Outcome: Change From Baseline in RR Interval - Part B
Description: as for outcome 104
Time Frame: Baseline, Days 1, 2, 7, 14 and follow-up Day 21
Population: as for outcome 58
Measure: Median (Full Range); unit: msec
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
msec
  Baseline | 952.0 [606 to 1429] | 938.0 [674 to 1250]
  Change from Baseline at Day 1: number analyzed (Participants) | 44 | 44
  Change from Baseline at Day 1 | -50.0 [-341 to 224] | -52.5 [-376 to 241]
  Change from Baseline at Day 2: number analyzed (Participants) | 44 | 44
  Change from Baseline at Day 2 | -46.0 [-327 to 108] | -51.0 [-387 to 225]
  Change from Baseline at Day 7: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 7 | -115.5 [-378 to 113] | -92.0 [-417 to 179]
  Change from Baseline at Day 14: number analyzed (Participants) | 41 | 40
  Change from Baseline at Day 14 | -111.0 [-478 to 163] | -142.0 [-397 to 139]
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -68.5 [-395 to 205] | -32.0 [-845 to 241]

108. Secondary Outcome: Change From Baseline in PR Interval - Part B
Description: as for outcome 104
Time Frame: Baseline, Days 1, 2, 7, 14 and follow-up Day 21
Population: as for outcome 58
Measure: Median (Full Range); unit: msec
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
msec
  Baseline | 149.5 [120 to 224] | 162.0 [131 to 203]
  Change from Baseline at Day 1: number analyzed (Participants) | 44 | 44
  Change from Baseline at Day 1 | 1.0 [-42 to 33] | 2.0 [-31 to 92]
  Change from Baseline at Day 2: number analyzed (Participants) | 44 | 44
  Change from Baseline at Day 2 | 1.5 [-30 to 31] | 4.0 [-24 to 79]
  Change from Baseline at Day 7: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 7 | 3.5 [-151 to 46] | 1.5 [-60 to 78]
  Change from Baseline at Day 14: number analyzed (Participants) | 41 | 40
  Change from Baseline at Day 14 | 4.0 [-151 to 50] | 3.0 [-26 to 70]
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | 0.0 [-27 to 23] | 0.5 [-163 to 85]

109. Secondary Outcome: Change From Baseline in QRS Duration - Part B
Description: as for outcome 104
Time Frame: Baseline, Days 1, 2, 7, 14 and follow-up Day 21
Population: as for outcome 58
Measure: Median (Full Range); unit: msec
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
msec
  Baseline | 88.0 [74 to 122] | 89.0 [66 to 121]
  Change from Baseline at Day 1: number analyzed (Participants) | 44 | 44
  Change from Baseline at Day 1 | 0.5 [-21 to 15] | 0.5 [-16 to 20]
  Change from Baseline at Day 2: number analyzed (Participants) | 44 | 44
  Change from Baseline at Day 2 | 1.0 [-13 to 14] | 1.0 [-19 to 16]
  Change from Baseline at Day 7: number analyzed (Participants) | 42 | 44
  Change from Baseline at Day 7 | -0.5 [-29 to 13] | -1.5 [-17 to 27]
  Change from Baseline at Day 14: number analyzed (Participants) | 41 | 40
  Change from Baseline at Day 14 | 0.0 [-23 to 11] | 0.0 [-19 to 21]
  Change from Baseline at Follow-up Day 21: number analyzed (Participants) | 38 | 42
  Change from Baseline at Follow-up Day 21 | -0.5 [-18 to 21] | 0.0 [-94 to 22]

110. Secondary Outcome: Percentage of Participants With a Response of "Yes" to Any C-SSRS Suicidal Ideation (SI) Item - Part B
Description: The C-SSRS scale consisted of a baseline evaluation (at screening) that assessed the lifetime experience of participants with suicidal ideation and behavior and a postbaseline evaluation that focused on suicidality since the last study visit. The C-SSRS included "yes" or "no"' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe). The C-SSRS SI items involved wish to be dead, non-specific active suicidal thoughts, active SI with any methods, active SI with some intent and active SI with specific plan. The analysis was performed in participants included in Part B of the study. SCLR = screening: lifetime recall.
Time Frame: Screening, Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 15, 21, 28, 35 and 42
Population: The safety set included all participants who received at least one dose of the study drug. Number analyzed: Number of participants in the safety set with a non-missing value at the visit within each treatment group.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
percentage of participants
  SCLR: Wish to be Dead | 11 | 8
  SCLR: Non-specific Active Suicidal Thoughts | 3 | 0
  SCLR: Active SI with Any Methods | 1 | 0
  SCLR: Active SI with Some Intent | 1 | 0
  Day 1: Wish to be Dead | 9.1 | 2.2
  Day 2: Wish to be Dead | 2.3 | 2.2
  Day 3: Wish to be Dead | 2.3 | 2.2
  Day 4: Wish to be Dead | 2.3 | 2.2
  Day 5: Wish to be Dead: number analyzed (Participants) | 43 | 45
  Day 5: Wish to be Dead | 2.3 | 2.2
  Day 6: Wish to be Dead | 2.3 | 2.2
  Day 7: Wish to be Dead: number analyzed (Participants) | 43 | 45
  Day 7: Wish to be Dead | 2.3 | 0
  Day 8: Wish to be Dead: number analyzed (Participants) | 42 | 44
  Day 8: Wish to be Dead | 2.4 | 0
  Day 9: Wish to be Dead: number analyzed (Participants) | 42 | 43
  Day 9: Wish to be Dead | 2.4 | 0
  Day 11: Wish to be Dead: number analyzed (Participants) | 42 | 43
  Day 11: Wish to be Dead | 2.4 | 0
  Day 12: Wish to be Dead: number analyzed (Participants) | 42 | 41
  Day 12: Wish to be Dead | 2.4 | 0
  Day 13: Wish to be Dead: number analyzed (Participants) | 40 | 40
  Day 13: Wish to be Dead | 2.5 | 0
  Day 15: Wish to be Dead: number analyzed (Participants) | 42 | 42
  Day 15: Wish to be Dead | 2.4 | 0
  Day 21: Wish to be Dead: number analyzed (Participants) | 38 | 42
  Day 21: Wish to be Dead | 2.6 | 0
  Day 28: Wish to be Dead: number analyzed (Participants) | 39 | 42
  Day 28: Wish to be Dead | 2.6 | 0
  Day 35: Wish to be Dead: number analyzed (Participants) | 40 | 41
  Day 35: Wish to be Dead | 2.5 | 0
  Day 42: Wish to be Dead: number analyzed (Participants) | 39 | 42
  Day 42: Wish to be Dead | 2.6 | 0

111. Secondary Outcome: Percentage of Participants With HAM-D Response - Part A
Description: HAM-D response was defined as having a 50% or greater reduction from baseline in HAM-D total score. The HAM-D total score comprised a sum of 17 individual item scores. Items scored in a range of 0 to 2 included: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score could range from 0 to 52. Higher scores indicate a greater degree of depression. A negative change from baseline indicated less depression. A positive change from baseline indicated more depression. The analysis was performed in participants included in Part A of the study. Data is reported for participants who had HAM-D response.
Time Frame: Days 2, 3, 4, 5, 6, 7, 8, 15, 21 and 28
Population: as for outcome 52
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
percentage of participants
  Day 2 | 15.4
  Day 3 | 15.4
  Day 4 | 30.8
  Day 5 | 53.8
  Day 6 | 61.5
  Day 7 | 61.5
  Day 8 | 84.6
  Day 15 | 84.6
  Day 21 | 76.9
  Day 28 | 76.9

112. Secondary Outcome: Percentage of Participants With HAM-D Remission - Part A
Description: HAM-D remission was defined as having a HAM-D total score of ≤7. The HAM-D total score comprised a sum of the 17 individual item scores. Items scored in a range of 0 to 2 included: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score could range from 0 to 52. Higher scores indicated a greater degree of depression. A negative change from baseline indicated less depression. A positive change from baseline indicated more depression. The analysis was performed in participants included in Part A of the study.
Time Frame: Days 2, 3, 4, 5, 6, 7, 8, 15, 21 and 28
Population: as for outcome 52
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
percentage of participants
  Day 2 | 0
  Day 3 | 0
  Day 4 | 15.4
  Day 5 | 15.4
  Day 6 | 38.5
  Day 7 | 38.5
  Day 8 | 46.2
  Day 15 | 61.5
  Day 21 | 69.2
  Day 28 | 69.2

113. Secondary Outcome: Change From Baseline in the Montgomery and Åsberg Depression Rating Scale (MADRS) Total Score at Day 15 and All Other Time Points - Part A
Description: The MADRS was a ten-item diagnostic questionnaire which psychiatrists used to measure the severity of depressive episodes in participants with mood disorders. It was designed as an adjunct to the HAM-D, to be more sensitive than the Hamilton Scale to the changes brought on by antidepressants and other forms of treatment. Each item yielded a score of 0 to 6. The MADRS total score was calculated as the sum of the 10 individual item scores, which ranged from 0 to 60. Higher MADRS scores indicated more severe depression. A negative change from baseline indicated less severe depression. A positive change from baseline indicated more severe depression. The analysis was performed in participants included in Part A of the study.
Time Frame: Baseline, Days 2, 3, 4, 5, 6, 7, 8, 15, 21 and 28
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
score on a scale
  Baseline | 36.9 (5.22)
  Change from Baseline at Day 2 | -6.4 (5.72)
  Change from Baseline at Day 3 | -9.6 (7.05)
  Change from Baseline at Day 4 | -14.2 (8.85)
  Change from Baseline at Day 5 | -16.2 (9.38)
  Change from Baseline at Day 6 | -18.9 (9.84)
  Change from Baseline at Day 7 | -19.3 (9.28)
  Change from Baseline at Day 8 | -22.8 (9.71)
  Change from Baseline at Day 15 | -26.4 (9.30)
  Change from Baseline at Day 21 | -26.1 (11.15)
  Change from Baseline at Day 28 | -25.0 (12.77)

114. Secondary Outcome: Change From Baseline in HAM-D Subscale Scores at Day 15 and All Other Time Points - Part A
Description: HAM-D subscales were: Core, symptoms: depressed mood (DM), feelings of guilt (FG), suicide, work and activities (WA), and retardation (RE); Anxiety, symptoms: anxiety (psychic and somatic), somatic symptoms (SS) (gastrointestinal and general), hypochondriasis, and loss of weight; Bech-6, symptoms: DM, FG, WA, RE, anxiety psychic (AP), and SS general; and Maier, symptoms: DM, FG, WA, RE, agitation, and AP. Each item was scored in a range of 0 to 2 or 0 to 4. Higher scores indicated a greater degree of depression. Subscale scores were calculated as sum of individual rating scores related to each subscale, divided by total possible score within subscale, multiplied by 100, and rounded to a whole number. Therefore, subscale scores would be within range of 0-100 and might be larger than total score. A negative change from baseline indicated less depression. A positive change from baseline indicated more depression. The analysis was performed in participants included in Part A of study.
Time Frame: Baseline, Days 2, 3, 4, 5, 6, 7, 8, 15, 21 and 28
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
score on a scale
  Core: Baseline | 45.0 (5.77)
  Core: Change from Baseline at Day 2 | -5.4 (8.03)
  Core: Change from Baseline at Day 3 | -12.3 (11.48)
  Core: Change from Baseline at Day 4 | -18.5 (13.90)
  Core: Change from Baseline at Day 5 | -21.9 (14.22)
  Core: Change from Baseline at Day 6 | -25.4 (11.27)
  Core: Change from Baseline at Day 7 | -25.4 (15.06)
  Core: Change from Baseline at Day 8 | -28.8 (14.88)
  Core: Change from Baseline at Day 15 | -34.6 (12.98)
  Core: Change from Baseline at Day 21 | -35.0 (15.68)
  Core: Change from Baseline at Day 28 | -33.5 (16.88)
  Anxiety: Baseline | 50.1 (10.52)
  Anxiety: Change from Baseline at Day 2 | -10.4 (8.89)
  Anxiety: Change from Baseline at Day 3 | -15.4 (9.79)
  Anxiety: Change from Baseline at Day 4 | -21.8 (12.16)
  Anxiety: Change from Baseline at Day 5 | -24.9 (14.23)
  Anxiety: Change from Baseline at Day 6 | -29.1 (13.70)
  Anxiety: Change from Baseline at Day 7 | -29.2 (13.44)
  Anxiety: Change from Baseline at Day 8 | -32.5 (15.86)
  Anxiety: Change from Baseline at Day 15 | -34.2 (14.73)
  Anxiety: Change from Baseline at Day 21 | -34.2 (14.62)
  Anxiety: Change from Baseline at Day 28 | -34.2 (15.79)
  Bech-6: Baseline | 61.6 (7.38)
  Bech-6: Change from Baseline at Day 2 | -8.2 (11.02)
  Bech-6: Change from Baseline at Day 3 | -16.6 (14.52)
  Bech-6: Change from Baseline at Day 4 | -25.5 (17.43)
  Bech-6: Change from Baseline at Day 5 | -29.4 (16.94)
  Bech-6: Change from Baseline at Day 6 | -34.0 (16.80)
  Bech-6: Change from Baseline at Day 7 | -34.4 (17.82)
  Bech-6: Change from Baseline at Day 8 | -38.9 (18.23)
  Bech-6: Change from Baseline at Day 15 | -45.4 (16.04)
  Bech-6: Change from Baseline at Day 21 | -44.5 (20.11)
  Bech-6: Change from Baseline at Day 28 | -42.2 (22.12)
  Meier: Baseline | 54.2 (8.57)
  Meier: Change from Baseline at Day 2 | -7.1 (8.80)
  Meier: Change from Baseline at Day 3 | -16.1 (10.87)
  Meier: Change from Baseline at Day 4 | -23.6 (11.99)
  Meier: Change from Baseline at Day 5 | -27.2 (12.55)
  Meier: Change from Baseline at Day 6 | -31.6 (12.13)
  Meier: Change from Baseline at Day 7 | -31.7 (14.49)
  Meier: Change from Baseline at Day 8 | -35.7 (14.57)
  Meier: Change from Baseline at Day 15 | -40.4 (13.78)
  Meier: Change from Baseline at Day 21 | -40.5 (17.23)
  Meier: Change from Baseline at Day 28 | -38.2 (18.78)

115. Secondary Outcome: Change From Baseline (CFB) in HAM-D Individual Item Scores at Day 15 and All Other Time Points - Part A
Description: The HAM-D comprised individual ratings of the following symptoms scored in a range of 0 to 2: insomnia (early, middle, late), somatic symptoms [gastrointestinal (GI) and general], genital symptoms, loss of weight, and insight. The following symptoms were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. Higher scores indicated a greater degree of depression. A negative change from baseline indicated less depression. A positive change from baseline indicated more depression. The analysis was performed in participants included in Part A of the study.
Time Frame: Baseline, Days 2, 3, 4, 5, 6, 7, 8, 15, 21 and 28
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
score on a scale
  Depressed Mood: Baseline | 3.2 (0.55)
  Depressed Mood: CFB at Day 2 | -0.2 (0.60)
  Depressed Mood: CFB at Day 3 | -0.8 (0.83)
  Depressed Mood: CFB at Day 4 | -1.3 (1.18)
  Depressed Mood: CFB at Day 5 | -1.4 (1.33)
  Depressed Mood: CFB at Day 6 | -1.6 (1.19)
  Depressed Mood: CFB at Day 7 | -1.6 (1.19)
  Depressed Mood: CFB at Day 8 | -1.8 (1.14)
  Depressed Mood: CFB at Day 15 | -2.2 (1.07)
  Depressed Mood: CFB at Day 21 | -2.2 (1.24)
  Depressed Mood: CFB at Day 28 | -2.0 (1.29)
  Work and Activities: Baseline | 3.1 (0.28)
  Work and Activities: CFB at Day 2 | -0.3 (0.48)
  Work and Activities: CFB at Day 3 | -0.7 (0.85)
  Work and Activities: CFB at Day 4 | -0.9 (0.86)
  Work and Activities: CFB at Day 5 | -1.4 (0.87)
  Work and Activities: CFB at Day 6 | -1.4 (0.96)
  Work and Activities: CFB at Day 7 | -1.5 (1.13)
  Work and Activities: CFB at Day 8 | -1.8 (1.21)
  Work and Activities: CFB at Day 15 | -2.5 (0.78)
  Work and Activities: CFB at Day 21 | -2.3 (1.11)
  Work and Activities: CFB at Day 28 | -2.2 (1.30)
  Insomnia Early: Baseline | 1.8 (0.55)
  Insomnia Early: CFB at Day 2 | -0.9 (0.86)
  Insomnia Early: CFB at Day 3 | -1.2 (0.90)
  Insomnia Early: CFB at Day 4 | -1.5 (0.88)
  Insomnia Early: CFB at Day 5 | -1.5 (0.78)
  Insomnia Early: CFB at Day 6 | -1.6 (0.77)
  Insomnia Early: CFB at Day 7 | -1.5 (0.78)
  Insomnia Early: CFB at Day 8 | -1.8 (0.55)
  Insomnia Early: CFB at Day 15 | -1.8 (0.55)
  Insomnia Early: CFB at Day 21 | -1.8 (0.60)
  Insomnia Early: CFB at Day 28 | -1.5 (0.88)
  Insomnia Middle: Baseline | 2.0 (0.00)
  Insomnia Middle: CFB at Day 2 | -0.9 (0.95)
  Insomnia Middle: CFB at Day 3 | -1.1 (0.76)
  Insomnia Middle: CFB at Day 4 | -1.2 (0.80)
  Insomnia Middle: CFB at Day 5 | -1.4 (0.65)
  Insomnia Middle: CFB at Day 6 | -1.4 (0.65)
  Insomnia Middle: CFB at Day 7 | -1.5 (0.78)
  Insomnia Middle: CFB at Day 8 | -1.6 (0.65)
  Insomnia Middle: CFB at Day 15 | -1.7 (0.48)
  Insomnia Middle: CFB at Day 21 | -1.5 (0.66)
  Insomnia Middle: CFB at Day 28 | -1.5 (0.66)
  Insomnia Late: Baseline | 1.8 (0.38)
  Insomnia Late: CFB at Day 2 | -0.8 (0.93)
  Insomnia Late: CFB at Day 3 | -0.8 (0.80)
  Insomnia Late: CFB at Day 4 | -1.0 (0.82)
  Insomnia Late: CFB at Day 5 | -1.3 (0.85)
  Insomnia Late: CFB at Day 6 | -1.2 (0.93)
  Insomnia Late: CFB at Day 7 | -1.3 (0.85)
  Insomnia Late: CFB at Day 8 | -1.3 (0.85)
  Insomnia Late: CFB at Day 15 | -1.5 (0.78)
  Insomnia Late: CFB at Day 21 | -1.5 (0.78)
  Insomnia Late: CFB at Day 28 | -1.4 (0.96)
  Genital Symptoms: Baseline | 2.0 (0.00)
  Genital Symptoms: CFB at Day 2 | -0.1 (0.28)
  Genital Symptoms: CFB at Day 3 | -0.1 (0.28)
  Genital Symptoms: CFB at Day 4 | -0.2 (0.60)
  Genital Symptoms: CFB at Day 5 | -0.3 (0.63)
  Genital Symptoms: CFB at Day 6 | -0.5 (0.66)
  Genital Symptoms: CFB at Day 7 | -0.5 (0.78)
  Genital Symptoms: CFB at Day 8 | -0.6 (0.77)
  Genital Symptoms: CFB at Day 15 | -0.8 (0.73)
  Genital Symptoms: CFB at Day 21 | -1.3 (0.85)
  Genital Symptoms: CFB at Day 28 | -1.3 (0.85)
  Somatic Symptoms GI: Baseline | 1.3 (0.75)
  Somatic Symptoms GI: CFB at Day 2 | -0.3 (0.63)
  Somatic Symptoms GI: CFB at Day 3 | -0.7 (0.63)
  Somatic Symptoms GI: CFB at Day 4 | -0.8 (0.60)
  Somatic Symptoms GI: CFB at Day 5 | -0.8 (0.73)
  Somatic Symptoms GI: CFB at Day 6 | -0.9 (0.64)
  Somatic Symptoms GI: CFB at Day 7 | -0.8 (0.69)
  Somatic Symptoms GI: CFB at Day 8 | -0.9 (0.76)
  Somatic Symptoms GI: CFB at Day 15 | -1.0 (0.82)
  Somatic Symptoms GI: CFB at Day 21 | -1.1 (0.76)
  Somatic Symptoms GI: CFB at Day 28 | -1.0 (0.82)
  Loss of Weight: Baseline | 0.5 (0.78)
  Loss of Weight: CFB at Day 2 | -0.5 (0.78)
  Loss of Weight: CFB at Day 3 | -0.4 (0.77)
  Loss of Weight: CFB at Day 4 | -0.4 (0.87)
  Loss of Weight: CFB at Day 5 | -0.4 (0.87)
  Loss of Weight: CFB at Day 6 | -0.5 (0.78)
  Loss of Weight: CFB at Day 7 | -0.5 (0.78)
  Loss of Weight: CFB at Day 8 | -0.4 (0.77)
  Loss of Weight: CFB at Day 15 | -0.3 (0.85)
  Loss of Weight: CFB at Day 21 | -0.5 (0.78)
  Loss of Weight: CFB at Day 28 | -0.5 (0.78)
  Somatic Symptoms General: Baseline | 1.9 (0.28)
  Somatic Symptoms General: CFB at Day 2 | -0.3 (0.63)
  Somatic Symptoms General: CFB at Day 3 | -0.4 (0.77)
  Somatic Symptoms General: CFB at Day 4 | -0.7 (0.85)
  Somatic Symptoms General: CFB at Day 5 | -0.8 (0.83)
  Somatic Symptoms General: CFB at Day 6 | -0.7 (0.95)
  Somatic Symptoms General: CFB at Day 7 | -0.8 (0.80)
  Somatic Symptoms General: CFB at Day 8 | -1.0 (0.82)
  Somatic Symptoms General: CFB at Day 15 | -1.2 (0.73)
  Somatic Symptoms General: CFB at Day 21 | -1.2 (0.80)
  Somatic Symptoms General: CFB at Day 28 | -1.2 (0.90)
  Feelings of Guilt: Baseline | 1.7 (0.63)
  Feelings of Guilt: CFB at Day 2 | -0.1 (0.49)
  Feelings of Guilt: CFB at Day 3 | -0.3 (1.03)
  Feelings of Guilt: CFB at Day 4 | -0.8 (0.83)
  Feelings of Guilt: CFB at Day 5 | -0.8 (0.99)
  Feelings of Guilt: CFB at Day 6 | -1.1 (0.86)
  Feelings of Guilt: CFB at Day 7 | -1.0 (0.91)
  Feelings of Guilt: CFB at Day 8 | -1.2 (0.80)
  Feelings of Guilt: CFB at Day 15 | -1.3 (0.75)
  Feelings of Guilt: CFB at Day 21 | -1.4 (0.77)
  Feelings of Guilt: CFB at Day 28 | -1.4 (0.77)
  Suicide: Baseline | 0.1 (0.28)
  Suicide: CFB at Day 2 | -0.1 (0.28)
  Suicide: CFB at Day 3 | -0.1 (0.28)
  Suicide: CFB at Day 4 | -0.1 (0.28)
  Suicide: CFB at Day 5 | -0.1 (0.28)
  Suicide: CFB at Day 6 | -0.1 (0.28)
  Suicide: CFB at Day 7 | -0.1 (0.28)
  Suicide: CFB at Day 8 | -0.1 (0.28)
  Suicide: CFB at Day 15 | -0.1 (0.28)
  Suicide: CFB at Day 21 | -0.1 (0.28)
  Suicide: CFB at Day 28 | -0.1 (0.28)
  Anxiety Psychic: Baseline | 2.7 (0.63)
  Anxiety Psychic: CFB at Day 2 | -0.5 (0.52)
  Anxiety Psychic: CFB at Day 3 | -0.8 (0.55)
  Anxiety Psychic: CFB at Day 4 | -1.3 (0.85)
  Anxiety Psychic: CFB at Day 5 | -1.4 (0.87)
  Anxiety Psychic: CFB at Day 6 | -1.8 (1.09)
  Anxiety Psychic: CFB at Day 7 | -1.7 (1.03)
  Anxiety Psychic: CFB at Day 8 | -1.8 (0.99)
  Anxiety Psychic: CFB at Day 15 | -1.9 (0.95)
  Anxiety Psychic: CFB at Day 21 | -1.7 (0.95)
  Anxiety Psychic: CFB at Day 28 | -1.5 (0.97)
  Anxiety Somatic: Baseline | 1.5 (0.66)
  Anxiety Somatic: CFB at Day 2 | -0.2 (0.55)
  Anxiety Somatic: CFB at Day 3 | -0.2 (0.73)
  Anxiety Somatic: CFB at Day 4 | -0.5 (0.78)
  Anxiety Somatic: CFB at Day 5 | -0.8 (0.60)
  Anxiety Somatic: CFB at Day 6 | -0.8 (0.60)
  Anxiety Somatic: CFB at Day 7 | -0.8 (0.69)
  Anxiety Somatic: CFB at Day 8 | -0.8 (0.80)
  Anxiety Somatic: CFB at Day 15 | -1.1 (0.64)
  Anxiety Somatic: CFB at Day 21 | -1.1 (0.86)
  Anxiety Somatic: CFB at Day 28 | -1.2 (0.69)
  Hypochondriasis: Baseline | 1.1 (0.76)
  Hypochondriasis: CFB at Day 2 | -0.2 (0.90)
  Hypochondriasis: CFB at Day 3 | -0.2 (0.60)
  Hypochondriasis: CFB at Day 4 | -0.3 (0.48)
  Hypochondriasis: CFB at Day 5 | -0.4 (0.51)
  Hypochondriasis: CFB at Day 6 | -0.6 (0.51)
  Hypochondriasis: CFB at Day 7 | -0.5 (0.52)
  Hypochondriasis: CFB at Day 8 | -0.8 (0.55)
  Hypochondriasis: CFB at Day 15 | -0.6 (0.51)
  Hypochondriasis: CFB at Day 21 | -0.7 (0.75)
  Hypochondriasis: CFB at Day 28 | -0.8 (0.80)
  Insight: Baseline | 0.2 (0.38)
  Insight: CFB at Day 2 | -0.1 (0.28)
  Insight: CFB at Day 3 | -0.1 (0.28)
  Insight: CFB at Day 4 | -0.2 (0.38)
  Insight: CFB at Day 5 | -0.2 (0.38)
  Insight: CFB at Day 6 | -0.2 (0.38)
  Insight: CFB at Day 7 | -0.2 (0.38)
  Insight: CFB at Day 8 | -0.2 (0.38)
  Insight: CFB at Day 15 | -0.2 (0.38)
  Insight: CFB at Day 21 | -0.2 (0.38)
  Insight: CFB at Day 28 | -0.2 (0.38)
  Agitation: Baseline | 1.4 (0.87)
  Agitation: CFB at Day 2 | -0.2 (0.44)
  Agitation: CFB at Day 3 | -0.6 (0.87)
  Agitation: CFB at Day 4 | -0.8 (0.83)
  Agitation: CFB at Day 5 | -0.8 (0.90)
  Agitation: CFB at Day 6 | -0.8 (0.69)
  Agitation: CFB at Day 7 | -0.9 (0.64)
  Agitation: CFB at Day 8 | -1.0 (0.71)
  Agitation: CFB at Day 15 | -0.9 (0.76)
  Agitation: CFB at Day 21 | -1.1 (0.76)
  Agitation: CFB at Day 28 | -1.0 (0.91)
  Retardation: Baseline | 1.0 (0.71)
  Retardation: CFB at Day 2 | -0.4 (0.65)
  Retardation: CFB at Day 3 | -0.6 (0.65)
  Retardation: CFB at Day 4 | -0.6 (0.65)
  Retardation: CFB at Day 5 | -0.7 (0.63)
  Retardation: CFB at Day 6 | -0.9 (0.76)
  Retardation: CFB at Day 7 | -0.8 (0.69)
  Retardation: CFB at Day 8 | -0.8 (0.69)
  Retardation: CFB at Day 15 | -0.9 (0.64)
  Retardation: CFB at Day 21 | -1.0 (0.71)
  Retardation: CFB at Day 28 | -1.0 (0.71)

116. Secondary Outcome: Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score at All Time Points - Part A
Description: The 14-item HAM-A was used to rate the severity of symptoms of anxiety. Each of the 14 items was defined by a series of symptoms, and measured both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Scoring for HAM-A was calculated by assigning scores of 0 (not present) to 4 (very severe), with a total score range of 0 to 56, where 0-13=Normal, 14-17 Mild Anxiety, 18-24 Moderate Anxiety, >=25 Severe Anxiety, per the Psych Congress Network. The HAM-A total score was calculated as the sum of the 14 individual item scores. A negative change from baseline indicated less anxiety. A positive change from baseline indicated more anxiety. The analysis was performed in participants included in Part A of the study.
Time Frame: Baseline, Days 2, 3, 8, 15, 21 and 28
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
score on a scale
  Baseline | 23.2 (5.65)
  Change from Baseline at Day 2 | -2.8 (3.44)
  Change from Baseline at Day 3 | -5.6 (3.59)
  Change from Baseline at Day 8 | -13.3 (6.25)
  Change from Baseline at Day 15 | -15.5 (6.19)
  Change from Baseline at Day 21 | -15.6 (7.05)
  Change from Baseline at Day 28 | -15.5 (7.22)

117. Secondary Outcome: Percentage of Participants With Clinical Global Impression - Improvement (CGI-I) Response - Part A
Description: The CGI-I item employed a 7-point Likert scale to measure the overall improvement in the participant's condition post-treatment. The investigator rated the participant's total improvement whether or not it was due entirely to drug treatment. Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. The CGI-I was only rated at post-treatment assessments. By definition, all CGI-I assessments were evaluated against baseline conditions. CGI-I response was defined as having a CGI-I global improvement score of 1 (very much improved) or 2 (much improved). The analysis was performed in participants included in Part A of the study. Data is reported for participants who had CGI-I response.
Time Frame: Days 2, 3, 8, 15, 21 and 28
Population: as for outcome 52
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SAGE-217
Number analyzed (Participants) | 13
percentage of participants
  Day 2 | 7.7
  Day 3 | 15.4
  Day 8 | 84.6
  Day 15 | 92.3
  Day 21 | 84.6
  Day 28 | 76.9

118. Secondary Outcome: Change From Baseline (CFB) in the SSS Score - Part B
Description: The SSS was participant-rated scale designed to quickly assess how alert a participant was feeling. Degrees of sleepiness and alertness were rated on a scale of one to seven, where the lowest score of 'one' indicated the participant was 'feeling active, vital, alert, or wide awake' and the highest score of 'seven' indicated the participant was 'no longer fighting sleep, sleep onset soon; having dream-like thoughts'. A negative change from baseline indicated less sleepiness. A positive change from baseline indicated more sleepiness. The analysis was performed in participants included in Part B of the study. H = Hour(s).
Time Frame: Baseline, Day 1 (0.25, 0.5, 1, 2 hours postdose), Days 2, 3, 4, 5, 6 and 7 (predose, 0.25, 0.5, 1, 2 hours postdose), Days 8, 9, 10, 11, 12, 13 and 14 (predose, 1 hour postdose), Day 15
Population: The safety set included all participants who received at least 1 dose of the double-blind study drug. Number analyzed: Number of participants in the safety set with a non-missing value at both baseline and the visit within each treatment group.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part B: Placebo: Eligible participants received matching placebo once daily for 14 days.
- Part B: SAGE-217: Eligible participants received SAGE-217, 30 mg, oral solution, once daily for 14 days.
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
score on a scale
  Baseline | 2.7 (1.47) | 2.6 (1.31)
  CFB at Day 1: 0.25 H Postdose | 0.0 (0.94) | 0.0 (0.82)
  CFB at Day 1: 0.5 H Postdose | -0.1 (0.73) | 0.0 (1.20)
  CFB at Day 1: 1 H Postdose | -0.1 (0.84) | 0.2 (1.54)
  CFB at Day 1: 2 H Postdose | -0.1 (1.26) | 0.6 (1.70)
  CFB at Day 2: Predose | -0.6 (1.19) | -0.1 (1.39)
  CFB at Day 2: 0.25 H Postdose | -0.5 (1.28) | 0.1 (1.59)
  CFB at Day 2: 0.5 H Postdose | -0.5 (1.13) | 0.2 (1.62)
  CFB at Day 2: 1 H Postdose | -0.3 (1.06) | 0.5 (1.75)
  CFB at Day 2: 2 H Postdose | 0.1 (1.29) | 0.4 (1.73)
  CFB at Day 3: Predose | -0.6 (1.14) | -0.4 (1.11)
  CFB at Day 3: 0.25 H Postdose | -0.7 (1.20) | -0.2 (1.45)
  CFB at Day 3: 0.5 H Postdose | -0.5 (1.05) | -0.1 (1.50)
  CFB at Day 3: 1 H Postdose | -0.3 (1.06) | 0.1 (1.55)
  CFB at Day 3: 2 H Postdose | 0.0 (1.21) | 0.5 (1.53)
  CFB at Day 4: Predose | -0.7 (1.22) | -0.3 (1.39)
  CFB at Day 4: 0.25 H Postdose | -0.7 (1.16) | -0.2 (1.37)
  CFB at Day 4: 0.5 H Postdose | -0.5 (1.19) | 0.0 (1.42)
  CFB at Day 4: 1 H Postdose | -0.4 (1.19) | 0.0 (1.44)
  CFB at Day 4: 2 H Postdose | -0.3 (1.21) | 0.4 (1.53)
  CFB at Day 5: Predose | -1.0 (1.49) | -0.5 (1.32)
  CFB at Day 5: 0.25 H Postdose | -0.8 (1.41) | -0.3 (1.44)
  CFB at Day 5: 0.5 H Postdose | -0.8 (1.31) | -0.2 (1.29)
  CFB at Day 5: 1 H Postdose | -0.6 (1.35) | 0.2 (1.50)
  CFB at Day 5: 2 H Postdose | -0.3 (1.37) | 0.4 (1.49)
  CFB at Day 6: Predose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: Predose | -0.8 (1.15) | -0.5 (1.39)
  CFB at Day 6: 0.25 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.25 H Postdose | -0.7 (1.20) | -0.2 (1.40)
  CFB at Day 6: 0.5 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 0.5 H Postdose | -0.6 (1.18) | -0.2 (1.39)
  CFB at Day 6: 1 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 1 H Postdose | -0.4 (1.03) | 0.1 (1.45)
  CFB at Day 6: 2 H Postdose: number analyzed (Participants) | 43 | 45
  CFB at Day 6: 2 H Postdose | -0.2 (1.17) | 0.2 (1.49)
  CFB at Day 7: Predose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: Predose | -0.8 (1.26) | -0.6 (1.31)
  CFB at Day 7: 0.25 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 0.25 H Postdose | -0.8 (1.25) | -0.5 (1.47)
  CFB at Day 7: 0.5 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 0.5 H Postdose | -0.6 (1.23) | -0.3 (1.30)
  CFB at Day 7: 1 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 1 H Postdose | -0.4 (1.25) | -0.2 (1.36)
  CFB at Day 7: 2 H Postdose: number analyzed (Participants) | 42 | 44
  CFB at Day 7: 2 H Postdose | -0.2 (1.25) | 0.1 (1.40)
  CFB at Day 8: Predose: number analyzed (Participants) | 42 | 43
  CFB at Day 8: Predose | -0.8 (1.34) | -0.7 (1.36)
  CFB at Day 8: 1 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 8: 1 H Postdose | -0.6 (1.38) | -0.2 (1.65)
  CFB at Day 9: Predose: number analyzed (Participants) | 42 | 43
  CFB at Day 9: Predose | -0.9 (1.38) | -0.6 (1.35)
  CFB at Day 9: 1 H Postdose: number analyzed (Participants) | 42 | 43
  CFB at Day 9: 1 H Postdose | -0.6 (1.23) | -0.3 (1.42)
  CFB at Day 10: Predose: number analyzed (Participants) | 42 | 42
  CFB at Day 10: Predose | -1.0 (1.32) | -0.6 (1.38)
  CFB at Day 10: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 10: 1 H Postdose | -0.7 (1.28) | -0.3 (1.55)
  CFB at Day 11: Predose: number analyzed (Participants) | 42 | 42
  CFB at Day 11: Predose | -0.7 (1.23) | -0.6 (1.36)
  CFB at Day 11: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 11: 1 H Postdose | -0.6 (1.31) | -0.3 (1.68)
  CFB at Day 12: Predose: number analyzed (Participants) | 42 | 41
  CFB at Day 12: Predose | -0.9 (1.25) | -0.7 (1.44)
  CFB at Day 12: 1 H Postdose: number analyzed (Participants) | 42 | 41
  CFB at Day 12: 1 H Postdose | -0.7 (1.30) | -0.4 (1.76)
  CFB at Day 13: Predose: number analyzed (Participants) | 40 | 40
  CFB at Day 13: Predose | -0.8 (1.30) | -0.8 (1.50)
  CFB at Day 13: 1 H Postdose: number analyzed (Participants) | 40 | 40
  CFB at Day 13: 1 H Postdose | -0.6 (1.34) | -0.4 (1.50)
  CFB at Day 14: Predose: number analyzed (Participants) | 41 | 41
  CFB at Day 14: Predose | -0.7 (1.27) | -0.7 (1.35)
  CFB at Day 14: 1 H Postdose: number analyzed (Participants) | 41 | 41
  CFB at Day 14: 1 H Postdose | -0.5 (1.31) | -0.3 (1.46)
  CFB at Day 15: number analyzed (Participants) | 38 | 41
  CFB at Day 15 | -0.6 (1.50) | -0.8 (1.61)

119. Secondary Outcome: Change From Baseline in the 17-item HAM-D Total Score at All Time Points - Part B
Description: as for outcome 52
Time Frame: Baseline, Days 2, 3, 4, 5, 6, 7, 8, 15, 21, 28, 35 and 42
Population: as for outcome 52
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
score on a scale
  Change from Baseline at Day 2 | -3.5 (0.98) | -5.8 (0.97)
  Change from Baseline at Day 3 | -5.2 (1.09) | -9.3 (1.07)
  Change from Baseline at Day 4 | -7.7 (1.13) | -10.6 (1.11)
  Change from Baseline at Day 5 | -8.5 (1.19) | -12.3 (1.17)
  Change from Baseline at Day 6 | -9.1 (1.21) | -13.6 (1.19)
  Change from Baseline at Day 7 | -9.2 (1.29) | -13.7 (1.27)
  Change from Baseline at Day 8 | -11.0 (1.29) | -14.4 (1.27)
  Change from Baseline at Day 15 | -10.3 (1.33) | -17.4 (1.31)
  Change from Baseline at Day 21 | -11.3 (1.43) | -16.3 (1.40)
  Change from Baseline at Day 28 | -11.3 (1.44) | -15.4 (1.41)
  Change from Baseline at Day 35 | -12.6 (1.49) | -14.9 (1.47)
  Change from Baseline at Day 42 | -12.3 (1.49) | -14.6 (1.46)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 2; Test type: Superiority; p = 0.0223, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-D total score at each visit as the dependent variables; Least Squares Mean Difference = -2.3, 95% CI 2-sided [-4.3 to -0.3], Standard Error of Mean 0.99
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 3; Test type: Superiority; p = 0.0010, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-D total score at each visit as the dependent variables; Least Squares Mean Difference = -4.1, 95% CI 2-sided [-6.4 to -1.7], Standard Error of Mean 1.18
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 4; Test type: Superiority; p = 0.0233, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-D total score at each visit as the dependent variables; Least Squares Mean Difference = -2.9, 95% CI 2-sided [-5.5 to -0.4], Standard Error of Mean 1.27
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 5; Test type: Superiority; p = 0.0066, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-D total score at each visit as the dependent variables; Least Squares Mean Difference = -3.8, 95% CI 2-sided [-6.6 to -1.1], Standard Error of Mean 1.37
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 6; Test type: Superiority; p = 0.0019, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-D total score at each visit as the dependent variables; Least Squares Mean Difference = -4.5, 95% CI 2-sided [-7.3 to -1.7], Standard Error of Mean 1.40
Statistical Analysis 6: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 7; Test type: Superiority; p = 0.0043, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-D total score at each visit as the dependent variables; Least Squares Mean Difference = -4.5, 95% CI 2-sided [-7.6 to -1.5], Standard Error of Mean 1.53
Statistical Analysis 7: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 8; Test type: Superiority; p = 0.0318, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-D total score at each visit as the dependent variables; Least Squares Mean Difference = -3.4, 95% CI 2-sided [-6.4 to -0.3], Standard Error of Mean 1.54
Statistical Analysis 8: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 15; Test type: Superiority; p < 0.0001, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-D total score at each visit as the dependent variables; Least Squares Mean Difference = -7.0, 95% CI 2-sided [-10.2 to -3.9], Standard Error of Mean 1.60
Statistical Analysis 9: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 21; Test type: Superiority; p = 0.0064, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-D total score at each visit as the dependent variables; Least Squares Mean Difference = -4.9, 95% CI 2-sided [-8.4 to -1.4], Standard Error of Mean 1.76
Statistical Analysis 10: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 28; Test type: Superiority; p = 0.0243, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-D total score at each visit as the dependent variables; Least Squares Mean Difference = -4.1, 95% CI 2-sided [-7.6 to -0.5], Standard Error of Mean 1.77
Statistical Analysis 11: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 35; Test type: Superiority; p = 0.2285, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-D total score at each visit as the dependent variables; Least Squares Mean Difference = -2.3, 95% CI 2-sided [-6.0 to 1.4], Standard Error of Mean 1.86
Statistical Analysis 12: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 42; Test type: Superiority; p = 0.2120, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-D total score at each visit as the dependent variables; Least Squares Mean Difference = -2.3, 95% CI 2-sided [-6.0 to 1.4], Standard Error of Mean 1.86

120. Secondary Outcome: Percentage of Participants With HAM-D Response - Part B
Description: HAM-D response was defined as having a 50% or greater reduction from baseline in HAM-D total score. The HAM-D total score comprised a sum of 17 individual item scores. Items scored in a range of 0 to 2 included: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score could range from 0 to 52. Higher scores indicated a greater degree of depression. A negative change from baseline indicated less depression. A positive change from baseline indicated more depression. The analysis was performed in participants included in Part B of the study. Data is reported for participants who had HAM-D response.
Time Frame: Days 2, 8, 15, 21, 28, 35 and 42
Population: The efficacy set included all participants who were randomized and received at least 1 dose of the double-blind study drug and had a baseline and at least 1 post-baseline efficacy evaluation. Number analyzed: Number of participants in the efficacy set ith a non-missing value at the visit within each treatment group.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
percentage of participants
  Day 2 | 4.5 | 15.6
  Day 8: number analyzed (Participants) | 42 | 44
  Day 8 | 47.6 | 59.1
  Day 15: number analyzed (Participants) | 42 | 42
  Day 15 | 40.5 | 78.6
  Day 21: number analyzed (Participants) | 38 | 42
  Day 21 | 42.1 | 73.8
  Day 28: number analyzed (Participants) | 39 | 42
  Day 28 | 46.2 | 61.9
  Day 35: number analyzed (Participants) | 40 | 41
  Day 35 | 50.0 | 65.9
  Day 42: number analyzed (Participants) | 39 | 42
  Day 42 | 56.4 | 61.9
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 2; Test type: Superiority; p = 0.0884, Generalized Estimating Equation; Statistics are from a generalized estimating equation (GEE) method including the HAM-D response at each visit as the dependent variables; Odds Ratio (OR) = 4.4, 95% CI 2-sided [0.8 to 24.1] — For the model parameters estimation, the exchangeable working correlation structure was used
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 8; Test type: Superiority; p = 0.0732, Generalized Estimating Equation; Statistics are from a GEE method including the HAM-D response at each visit as the dependent variables; Odds Ratio (OR) = 2.4, 95% CI 2-sided [0.9 to 6.4] — For the model parameters estimation, the exchangeable working correlation structure was used
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 15; Test type: Superiority; p = 0.0002, Generalized Estimating Equation; Statistics are from a GEE method including the HAM-D response at each visit as the dependent variables; Odds Ratio (OR) = 9.6, 95% CI 2-sided [2.9 to 31.6] — For the model parameters estimation, the exchangeable working correlation structure was used
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 21; Test type: Superiority; p = 0.0006, Generalized Estimating Equation; Statistics are from a GEE method including the HAM-D response at each visit as the dependent variables; Odds Ratio (OR) = 6.7, 95% CI 2-sided [2.3 to 19.7] — For the model parameters estimation, the exchangeable working correlation structure was used
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 28; Test type: Superiority; p = 0.0379, Generalized Estimating Equation; Statistics are from a GEE method including the HAM-D response at each visit as the dependent variables; Odds Ratio (OR) = 3.1, 95% CI 2-sided [1.1 to 8.9] — For the model parameters estimation, the exchangeable working correlation structure was used
Statistical Analysis 6: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 35; Test type: Superiority; p = 0.0468, Generalized Estimating Equation; Statistics are from a GEE method including the HAM-D response at each visit as the dependent variables; Odds Ratio (OR) = 3.0, 95% CI 2-sided [1.0 to 9.0] — For the model parameters estimation, the exchangeable working correlation structure was used
Statistical Analysis 7: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 42; Test type: Superiority; p = 0.2208, Generalized Estimating Equation; Statistics are from a GEE method including the HAM-D response at each visit as the dependent variables; Odds Ratio (OR) = 1.9, 95% CI 2-sided [0.7 to 5.6] — For the model parameters estimation, the exchangeable working correlation structure was used

121. Secondary Outcome: Percentage of Participants With HAM-D Remission - Part B
Description: HAM-D remission was defined as having a HAM-D total score of ≤7. The HAM-D total score comprised a sum of the 17 individual item scores. Items scored in a range of 0 to 2 included: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score could range from 0 to 52. Higher scores indicated a greater degree of depression. A negative change from baseline indicated less depression. A positive change from baseline indicated more depression. The analysis was performed in participants included in Part B of the study.
Time Frame: Days 2, 8, 15, 21, 28, 35 and 42
Population: The efficacy set included all participants who were randomized and received at least 1 dose of the double-blind study drug and had a baseline and at least 1 post-baseline efficacy evaluation. Number analyzed: Number of participants in efficacy set with a non-missing value at both baseline and the visit within each treatment group.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
percentage of participants
  Day 2 | 0 | 2.2
  Day 8: number analyzed (Participants) | 42 | 44
  Day 8 | 28.6 | 36.4
  Day 15: number analyzed (Participants) | 42 | 42
  Day 15 | 26.2 | 64.3
  Day 21: number analyzed (Participants) | 38 | 42
  Day 21 | 26.3 | 52.4
  Day 28: number analyzed (Participants) | 39 | 42
  Day 28 | 28.2 | 52.4
  Day 35: number analyzed (Participants) | 40 | 41
  Day 35 | 35.0 | 43.9
  Day 42: number analyzed (Participants) | 39 | 42
  Day 42 | 33.3 | 45.2
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 8; Test type: Superiority; p = 0.4300, Generalized Estimating Equation; Statistics are from a GEE method including the HAM-D remission at each visit as the dependent variables; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.6 to 3.7] — For the model parameters estimation, the exchangeable working correlation structure was used
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 15; Test type: Superiority; p = 0.0005, Generalized Estimating Equation; Statistics are from a GEE method including the HAM-D remission at each visit as the dependent variables; Odds Ratio (OR) = 5.3, 95% CI 2-sided [2.1 to 13.3] — For the model parameters estimation, the exchangeable working correlation structure was used
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 21; Test type: Superiority; p = 0.0172, Generalized Estimating Equation; Statistics are from a GEE method including the HAM-D remission at each visit as the dependent variables; Odds Ratio (OR) = 3.1, 95% CI 2-sided [1.2 to 8.0] — For the model parameters estimation, the exchangeable working correlation structure was used
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 28; Test type: Superiority; p = 0.0221, Generalized Estimating Equation; Statistics are from a GEE method including the HAM-D remission at each visit as the dependent variables; Odds Ratio (OR) = 2.9, 95% CI 2-sided [1.2 to 7.3] — For the model parameters estimation, the exchangeable working correlation structure was used
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 35; Test type: Superiority; p = 0.4139, Generalized Estimating Equation; Statistics are from a GEE method including the HAM-D remission at each visit as the dependent variables; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.6 to 3.5] — For the model parameters estimation, the exchangeable working correlation structure was used
Statistical Analysis 6: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 42; Test type: Superiority; p = 0.2332, Generalized Estimating Equation; Statistics are from a GEE method including the HAM-D remission at each visit as the dependent variables; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.7 to 4.3] — For the model parameters estimation, the exchangeable working correlation structure was used

122. Secondary Outcome: Change From Baseline in the MADRS Total Score at Day 15 and All Other Time Points - Part B
Description: The MADRS was a ten-item diagnostic questionnaire which psychiatrists used to measure the severity of depressive episodes in participants with mood disorders. It was designed as an adjunct to the HAM-D, to be more sensitive than the Hamilton Scale to the changes brought on by antidepressants and other forms of treatment. Each item yielded a score of 0 to 6. The MADRS total score was calculated as the sum of the 10 individual item scores, which ranged from 0 to 60. Higher MADRS scores indicated more severe depression. A negative change from baseline indicated less severe depression. A positive change from baseline indicated more severe depression. The analysis was performed in participants included in Part B of the study.
Time Frame: Baseline, Days 2, 8, 15, 21, 28, 35 and 42
Population: as for outcome 52
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
score on a scale
  Change from Baseline at Day 2 | -4.5 (1.36) | -6.9 (1.35)
  Change from Baseline at Day 8 | -15.4 (1.90) | -19.4 (1.88)
  Change from Baseline at Day 15 | -15.0 (1.94) | -22.5 (1.92)
  Change from Baseline at Day 21 | -15.2 (2.14) | -21.9 (2.11)
  Change from Baseline at Day 28 | -14.8 (2.14) | -20.1 (2.11)
  Change from Baseline at Day 35 | -16.4 (2.25) | -19.4 (2.23)
  Change from Baseline at Day 42 | -17.2 (2.15) | -19.1 (2.11)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 2; Test type: Superiority; p = 0.0836, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in MADRS total score at each visit as the dependent variable; Least Squares Mean Difference = -2.4, 95% CI 2-sided [-5.1 to 0.3], Standard Error of Mean 1.38
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 8; Test type: Superiority; p = 0.0864, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in MADRS total score at each visit as the dependent variable; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-8.6 to 0.6], Standard Error of Mean 2.32
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 15; Test type: Superiority; p = 0.0021, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in MADRS total score at each visit as the dependent variable; Least Squares Mean Difference = -7.6, 95% CI 2-sided [-12.3 to -2.8], Standard Error of Mean 2.38
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 21; Test type: Superiority; p = 0.0157, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in MADRS total score at each visit as the dependent variable; Least Squares Mean Difference = -6.6, 95% CI 2-sided [-12.0 to -1.3], Standard Error of Mean 2.69
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 28; Test type: Superiority; p = 0.0533, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in MADRS total score at each visit as the dependent variable; Least Squares Mean Difference = -5.3, 95% CI 2-sided [-10.6 to 0.1], Standard Error of Mean 2.69
Statistical Analysis 6: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 35; Test type: Superiority; p = 0.2878, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in MADRS total score at each visit as the dependent variable; Least Squares Mean Difference = -3.1, 95% CI 2-sided [-8.8 to 2.6], Standard Error of Mean 2.87
Statistical Analysis 7: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 42; Test type: Superiority; p = 0.4664, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in MADRS total score at each visit as the dependent variable; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-7.4 to 3.4], Standard Error of Mean 2.70

123. Secondary Outcome: Change From Baseline in HAM-D Subscale Scores at All Time Points - Part B
Description: HAM-D subscales were: Core, symptoms: depressed mood (DM), feelings of guilt (FG), suicide, work and activities (WA), and retardation (RE); Anxiety, symptoms: anxiety (psychic and somatic), somatic symptoms (SS) (gastrointestinal and general), hypochondriasis, and loss of weight; Bech-6, symptoms: DM, FG, WA, RE, anxiety psychic (AP), and SS general; and Maier, symptoms: DM, FG, WA, RE, agitation, and AP. Each item was scored in a range of 0 to 2 or 0 to 4. Higher scores indicated a greater degree of depression. Subscale scores were calculated as sum of individual rating scores related to each subscale, divided by total possible score within subscale, multiplied by 100, and rounded to a whole number. Therefore, subscale scores would be within range of 0-100 and might be larger than total score. A negative change from baseline indicated less depression. A positive change from baseline indicated more depression. The analysis was performed in participants included in Part B of study.
Time Frame: Baseline, Days 2, 3, 4, 5, 6, 7, 8, 15, 21, 28, 35 and 42
Population: The efficacy set included all participants who were randomized and received at least 1 dose of the double-blind study drug and had a baseline and at least 1 post-baseline efficacy evaluation. Number analyzed: Number of participants in efficacy set with a non-missing value at both baseline and visit within each treatment group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
score on a scale
  Core: Baseline | 47.3 (6.86) | 46.9 (7.01)
  Core: Change from Baseline at Day 2 | -5.9 (6.84) | -7.2 (12.04)
  Core: Change from Baseline at Day 3 | -9.4 (9.16) | -14.1 (14.31)
  Core: Change from Baseline at Day 4: number analyzed (Participants) | 43 | 45
  Core: Change from Baseline at Day 4 | -13.3 (10.85) | -18.3 (14.92)
  Core: Change from Baseline at Day 5 | -15.8 (12.39) | -21.2 (15.45)
  Core: Change from Baseline at Day 6 | -17.5 (14.04) | -25.6 (15.20)
  Core: Change from Baseline at Day 7: number analyzed (Participants) | 43 | 45
  Core: Change from Baseline at Day 7 | -18.0 (15.97) | -24.8 (15.74)
  Core: Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Core: Change from Baseline at Day 8 | -22.5 (16.28) | -26.6 (16.35)
  Core: Change from Baseline at Day 15: number analyzed (Participants) | 42 | 42
  Core: Change from Baseline at Day 15 | -21.9 (17.94) | -33.1 (14.73)
  Core: Change from Baseline at Day 21: number analyzed (Participants) | 38 | 42
  Core: Change from Baseline at Day 21 | -22.9 (17.77) | -30.7 (16.10)
  Core: Change from Baseline at Day 28: number analyzed (Participants) | 39 | 42
  Core: Change from Baseline at Day 28 | -22.1 (17.42) | -29.3 (17.89)
  Core: Change from Baseline at Day 35: number analyzed (Participants) | 40 | 41
  Core: Change from Baseline at Day 35 | -24.3 (17.34) | -28.2 (17.20)
  Core: Change from Baseline at Day 42: number analyzed (Participants) | 39 | 42
  Core: Change from Baseline at Day 42 | -25.8 (17.79) | -28.0 (18.41)
  Anxiety: Baseline | 48.1 (13.28) | 48.8 (11.46)
  Anxiety: Change from Baseline at Day 2 | -8.4 (10.51) | -12.8 (12.63)
  Anxiety: Change from Baseline at Day 3 | -12.5 (10.21) | -18.9 (15.03)
  Anxiety: Change from Baseline at Day 4: number analyzed (Participants) | 43 | 45
  Anxiety: Change from Baseline at Day 4 | -17.5 (17.17) | -21.8 (16.33)
  Anxiety: Change from Baseline at Day 5 | -18.5 (18.72) | -24.1 (15.83)
  Anxiety: Change from Baseline at Day 6 | -18.8 (18.30) | -26.5 (17.21)
  Anxiety: Change from Baseline at Day 7: number analyzed (Participants) | 43 | 45
  Anxiety: Change from Baseline at Day 7 | -19.5 (17.65) | -25.4 (17.66)
  Anxiety: Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Anxiety: Change from Baseline at Day 8 | -21.5 (18.32) | -27.9 (17.96)
  Anxiety: Change from Baseline at Day 15: number analyzed (Participants) | 42 | 42
  Anxiety: Change from Baseline at Day 15 | -20.5 (17.11) | -34.1 (16.27)
  Anxiety: Change from Baseline at Day 21: number analyzed (Participants) | 38 | 42
  Anxiety: Change from Baseline at Day 21 | -23.6 (18.67) | -32.7 (17.85)
  Anxiety: Change from Baseline at Day 28: number analyzed (Participants) | 39 | 42
  Anxiety: Change from Baseline at Day 28 | -23.1 (20.34) | -30.8 (16.95)
  Anxiety: Change from Baseline at Day 35: number analyzed (Participants) | 40 | 41
  Anxiety: Change from Baseline at Day 35 | -24.9 (20.74) | -30.0 (17.75)
  Anxiety: Change from Baseline at Day 42: number analyzed (Participants) | 39 | 42
  Anxiety: Change from Baseline at Day 42 | -22.9 (21.60) | -29.7 (16.57)
  Bech-6: Baseline | 60.1 (7.12) | 59.8 (7.23)
  Bech-6: Change from Baseline at Day 2 | -6.8 (9.71) | -10.2 (14.55)
  Bech-6: Change from Baseline at Day 3 | -11.3 (9.38) | -18.8 (17.93)
  Bech-6: Change from Baseline at Day 4: number analyzed (Participants) | 43 | 45
  Bech-6: Change from Baseline at Day 4 | -17.0 (13.92) | -23.8 (19.11)
  Bech-6: Change from Baseline at Day 5 | -19.5 (16.61) | -26.8 (19.32)
  Bech-6: Change from Baseline at Day 6 | -21.4 (16.76) | -32.0 (20.13)
  Bech-6: Change from Baseline at Day 7: number analyzed (Participants) | 43 | 45
  Bech-6: Change from Baseline at Day 7 | -22.8 (18.88) | -31.4 (19.69)
  Bech-6: Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Bech-6: Change from Baseline at Day 8 | -27.5 (19.47) | -33.0 (20.08)
  Bech-6: Change from Baseline at Day 15: number analyzed (Participants) | 42 | 42
  Bech-6: Change from Baseline at Day 15 | -26.3 (21.07) | -41.8 (17.78)
  Bech-6: Change from Baseline at Day 21: number analyzed (Participants) | 38 | 42
  Bech-6: Change from Baseline at Day 21 | -27.9 (20.69) | -38.8 (20.80)
  Bech-6: Change from Baseline at Day 28: number analyzed (Participants) | 39 | 42
  Bech-6: Change from Baseline at Day 28 | -27.7 (21.02) | -36.1 (21.86)
  Bech-6: Change from Baseline at Day 35: number analyzed (Participants) | 40 | 41
  Bech-6: Change from Baseline at Day 35 | -29.3 (22.03) | -35.0 (21.51)
  Bech-6: Change from Baseline at Day 42: number analyzed (Participants) | 39 | 42
  Bech-6: Change from Baseline at Day 42 | -30.2 (22.34) | -34.7 (22.35)
  Meier: Baseline | 51.1 (6.56) | 49.4 (5.58)
  Meier: Change from Baseline at Day 2 | -6.3 (8.68) | -7.8 (12.10)
  Meier: Change from Baseline at Day 3 | -9.6 (8.54) | -16.0 (15.18)
  Meier: Change from Baseline at Day 4: number analyzed (Participants) | 43 | 45
  Meier: Change from Baseline at Day 4 | -14.1 (12.47) | -20.4 (16.38)
  Meier: Change from Baseline at Day 5 | -17.3 (13.74) | -23.2 (15.88)
  Meier: Change from Baseline at Day 6 | -18.2 (14.24) | -27.5 (16.95)
  Meier: Change from Baseline at Day 7: number analyzed (Participants) | 43 | 45
  Meier: Change from Baseline at Day 7 | -19.4 (16.85) | -26.3 (16.90)
  Meier: Change from Baseline at Day 8: number analyzed (Participants) | 42 | 44
  Meier: Change from Baseline at Day 8 | -24.6 (16.85) | -27.9 (16.72)
  Meier: Change from Baseline at Day 15: number analyzed (Participants) | 42 | 42
  Meier: Change from Baseline at Day 15 | -22.6 (17.15) | -35.1 (14.55)
  Meier: Change from Baseline at Day 21: number analyzed (Participants) | 38 | 42
  Meier: Change from Baseline at Day 21 | -23.8 (18.08) | -32.5 (16.88)
  Meier: Change from Baseline at Day 28: number analyzed (Participants) | 39 | 42
  Meier: Change from Baseline at Day 28 | -24.2 (17.57) | -30.8 (17.36)
  Meier: Change from Baseline at Day 35: number analyzed (Participants) | 40 | 41
  Meier: Change from Baseline at Day 35 | -25.5 (17.89) | -29.5 (18.24)
  Meier: Change from Baseline at Day 42: number analyzed (Participants) | 39 | 42
  Meier: Change from Baseline at Day 42 | -26.7 (18.21) | -29.1 (18.27)

124. Secondary Outcome: Change From Baseline (CFB) in HAM-D Individual Item Scores at All Time Points - Part B
Description: The HAM-D comprised individual ratings of the following symptoms scored in a range of 0 to 2: insomnia (early, middle, late), somatic symptoms (GI and general), genital symptoms, loss of weight, and insight. The following symptoms were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. Higher scores indicated a greater degree of depression. A negative change from baseline indicated less depression. A positive change from baseline indicated more depression. The analysis was performed in participants included in Part B of the study.
Time Frame: Baseline, Days 2, 3, 4, 5, 6, 7, 8, 15, 21, 28, 35 and 42
Population: as for outcome 121
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
score on a scale
  Depressed Mood: Baseline | 3.1 (0.56) | 3.1 (0.32)
  Depressed Mood: CFB at Day 2 | -0.3 (0.54) | -0.5 (0.84)
  Depressed Mood: CFB at Day 3 | -0.5 (0.63) | -0.8 (0.90)
  Depressed Mood: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Depressed Mood: CFB at Day 4 | -0.7 (0.77) | -1.2 (1.09)
  Depressed Mood: CFB at Day 5 | -1.0 (0.86) | -1.2 (1.10)
  Depressed Mood: CFB at Day 6 | -1.0 (0.99) | -1.6 (1.12)
  Depressed Mood: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Depressed Mood: CFB at Day 7 | -1.1 (1.14) | -1.4 (1.16)
  Depressed Mood: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Depressed Mood: CFB at Day 8 | -1.4 (1.25) | -1.7 (1.14)
  Depressed Mood: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Depressed Mood: CFB at Day 15 | -1.3 (1.23) | -2.0 (1.07)
  Depressed Mood: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Depressed Mood: CFB at Day 21 | -1.3 (1.34) | -1.8 (1.09)
  Depressed Mood: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Depressed Mood: CFB at Day 28 | -1.3 (1.31) | -1.7 (1.22)
  Depressed Mood: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Depressed Mood: CFB at Day 35 | -1.3 (1.31) | -1.7 (1.15)
  Depressed Mood: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Depressed Mood: CFB at Day 42 | -1.4 (1.29) | -1.7 (1.20)
  Work and Activities: Baseline | 3.1 (0.42) | 3.1 (0.33)
  Work and Activities: CFB at Day 2 | -0.3 (0.56) | -0.5 (0.89)
  Work and Activities: CFB at Day 3 | -0.5 (0.59) | -1.0 (1.18)
  Work and Activities: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Work and Activities: CFB at Day 4 | -0.9 (0.77) | -1.1 (1.12)
  Work and Activities: CFB at Day 5 | -1.0 (0.88) | -1.3 (1.28)
  Work and Activities: CFB at Day 6 | -1.2 (0.99) | -1.4 (1.27)
  Work and Activities: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Work and Activities: CFB at Day 7 | -1.1 (1.05) | -1.4 (1.20)
  Work and Activities: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Work and Activities: CFB at Day 8 | -1.4 (1.15) | -1.6 (1.22)
  Work and Activities: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Work and Activities: CFB at Day 15 | -1.5 (1.09) | -2.1 (1.18)
  Work and Activities: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Work and Activities: CFB at Day 21 | -1.5 (1.22) | -1.9 (1.09)
  Work and Activities: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Work and Activities: CFB at Day 28 | -1.6 (1.27) | -1.8 (1.22)
  Work and Activities: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Work and Activities: CFB at Day 35 | -1.7 (1.26) | -1.8 (1.31)
  Work and Activities: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Work and Activities: CFB at Day 42 | -1.8 (1.29) | -1.7 (1.29)
  Insomnia Early: Baseline | 1.7 (0.71) | 1.7 (0.65)
  Insomnia Early: CFB at Day 2 | 0.0 (0.82) | -0.5 (1.08)
  Insomnia Early: CFB at Day 3 | -0.2 (0.92) | -0.8 (1.07)
  Insomnia Early: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Insomnia Early: CFB at Day 4 | -0.3 (0.80) | -0.7 (1.16)
  Insomnia Early: CFB at Day 5 | -0.3 (0.88) | -1.0 (1.13)
  Insomnia Early: CFB at Day 6 | -0.5 (1.00) | -1.0 (1.02)
  Insomnia Early: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Insomnia Early: CFB at Day 7 | -0.3 (0.94) | -1.0 (1.02)
  Insomnia Early: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Insomnia Early: CFB at Day 8 | -0.4 (1.01) | -1.2 (0.90)
  Insomnia Early: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Insomnia Early: CFB at Day 15 | -0.2 (0.96) | -1.3 (1.00)
  Insomnia Early: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Insomnia Early: CFB at Day 21 | -0.3 (1.14) | -1.2 (0.94)
  Insomnia Early: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Insomnia Early: CFB at Day 28 | -0.5 (1.17) | -1.0 (0.96)
  Insomnia Early: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Insomnia Early: CFB at Day 35 | -0.5 (1.13) | -1.0 (1.04)
  Insomnia Early: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Insomnia Early: CFB at Day 42 | -0.7 (1.13) | -0.9 (0.98)
  Insomnia Middle: Baseline | 1.8 (0.51) | 1.7 (0.64)
  Insomnia Middle: CFB at Day 2 | -0.4 (0.87) | -0.5 (0.99)
  Insomnia Middle: CFB at Day 3 | -0.5 (0.79) | -1.0 (0.93)
  Insomnia Middle: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Insomnia Middle: CFB at Day 4 | -0.6 (0.95) | -0.9 (0.97)
  Insomnia Middle: CFB at Day 5 | -0.6 (0.87) | -0.9 (1.07)
  Insomnia Middle: CFB at Day 6 | -0.8 (1.05) | -0.9 (1.06)
  Insomnia Middle: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Insomnia Middle: CFB at Day 7 | -0.7 (0.99) | -1.0 (0.95)
  Insomnia Middle: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Insomnia Middle: CFB at Day 8 | -0.9 (1.01) | -1.1 (0.93)
  Insomnia Middle: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Insomnia Middle: CFB at Day 15 | -0.6 (0.99) | -1.2 (0.95)
  Insomnia Middle: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Insomnia Middle: CFB at Day 21 | -0.8 (0.90) | -1.2 (0.86)
  Insomnia Middle: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Insomnia Middle: CFB at Day 28 | -0.8 (0.98) | -0.9 (0.96)
  Insomnia Middle: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Insomnia Middle: CFB at Day 35 | -0.9 (1.00) | -0.9 (0.98)
  Insomnia Middle: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Insomnia Middle: CFB at Day 42 | -0.8 (0.94) | -1.0 (0.94)
  Insomnia Late: Baseline | 1.6 (0.70) | 1.5 (0.82)
  Insomnia Late: CFB at Day 2 | -0.5 (0.95) | -0.6 (1.05)
  Insomnia Late: CFB at Day 3 | -0.6 (1.00) | -0.7 (1.24)
  Insomnia Late: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Insomnia Late: CFB at Day 4 | -0.7 (1.09) | -0.7 (1.18)
  Insomnia Late: CFB at Day 5 | -0.8 (1.06) | -0.8 (1.24)
  Insomnia Late: CFB at Day 6 | -0.8 (1.06) | -0.9 (1.22)
  Insomnia Late: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Insomnia Late: CFB at Day 7 | -0.9 (1.10) | -0.8 (1.31)
  Insomnia Late: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Insomnia Late: CFB at Day 8 | -0.9 (1.05) | -0.9 (1.18)
  Insomnia Late: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Insomnia Late: CFB at Day 15 | -0.7 (1.04) | -1.1 (1.13)
  Insomnia Late: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Insomnia Late: CFB at Day 21 | -0.8 (1.05) | -1.0 (1.22)
  Insomnia Late: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Insomnia Late: CFB at Day 28 | -0.8 (1.14) | -1.0 (1.19)
  Insomnia Late: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Insomnia Late: CFB at Day 35 | -1.0 (1.11) | -0.9 (1.21)
  Insomnia Late: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Insomnia Late: CFB at Day 42 | -0.9 (1.09) | -1.1 (1.01)
  Genital Symptoms: Baseline | 1.7 (0.60) | 1.6 (0.68)
  Genital Symptoms: CFB at Day 2 | -0.1 (0.50) | -0.1 (0.50)
  Genital Symptoms: CFB at Day 3 | -0.1 (0.42) | -0.1 (0.42)
  Genital Symptoms: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Genital Symptoms: CFB at Day 4 | -0.2 (0.57) | -0.1 (0.67)
  Genital Symptoms: CFB at Day 5 | -0.2 (0.51) | -0.4 (0.69)
  Genital Symptoms: CFB at Day 6 | -0.3 (0.61) | -0.3 (0.56)
  Genital Symptoms: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Genital Symptoms: CFB at Day 7 | -0.3 (0.58) | -0.6 (0.72)
  Genital Symptoms: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Genital Symptoms: CFB at Day 8 | -0.4 (0.67) | -0.5 (0.66)
  Genital Symptoms: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Genital Symptoms: CFB at Day 15 | -0.6 (0.79) | -0.8 (0.78)
  Genital Symptoms: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Genital Symptoms: CFB at Day 21 | -0.6 (0.89) | -0.9 (0.80)
  Genital Symptoms: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Genital Symptoms: CFB at Day 28 | -0.6 (0.78) | -0.8 (0.87)
  Genital Symptoms: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Genital Symptoms: CFB at Day 35 | -0.7 (0.86) | -0.8 (0.90)
  Genital Symptoms: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Genital Symptoms: CFB at Day 42 | -0.6 (0.88) | -0.7 (0.86)
  Somatic Symptoms GI: Baseline | 1.3 (0.79) | 1.5 (0.76)
  Somatic Symptoms GI: CFB at Day 2 | -0.1 (0.69) | -0.4 (0.62)
  Somatic Symptoms GI: CFB at Day 3 | -0.2 (0.64) | -0.6 (0.77)
  Somatic Symptoms GI: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Somatic Symptoms GI: CFB at Day 4 | -0.4 (0.82) | -0.7 (0.73)
  Somatic Symptoms GI: CFB at Day 5 | -0.5 (0.98) | -0.8 (0.77)
  Somatic Symptoms GI: CFB at Day 6 | -0.5 (0.95) | -0.8 (0.85)
  Somatic Symptoms GI: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Somatic Symptoms GI: CFB at Day 7 | -0.4 (1.00) | -0.9 (0.89)
  Somatic Symptoms GI: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Somatic Symptoms GI: CFB at Day 8 | -0.5 (0.94) | -0.9 (0.95)
  Somatic Symptoms GI: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Somatic Symptoms GI: CFB at Day 15 | -0.4 (1.01) | -1.1 (0.86)
  Somatic Symptoms GI: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Somatic Symptoms GI: CFB at Day 21 | -0.6 (0.95) | -1.1 (0.89)
  Somatic Symptoms GI: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Somatic Symptoms GI: CFB at Day 28 | -0.6 (0.91) | -1.0 (0.92)
  Somatic Symptoms GI: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Somatic Symptoms GI: CFB at Day 35 | -0.7 (0.94) | -1.0 (0.89)
  Somatic Symptoms GI: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Somatic Symptoms GI: CFB at Day 42 | -0.7 (0.77) | -0.9 (0.84)
  Loss of Weight: Baseline | 0.9 (0.87) | 1.1 (0.86)
  Loss of Weight: CFB at Day 2 | -0.5 (0.73) | -0.5 (0.79)
  Loss of Weight: CFB at Day 3 | -0.5 (0.90) | -0.7 (0.88)
  Loss of Weight: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Loss of Weight: CFB at Day 4 | -0.5 (0.91) | -0.7 (1.00)
  Loss of Weight: CFB at Day 5 | -0.6 (0.97) | -0.7 (0.86)
  Loss of Weight: CFB at Day 6 | -0.6 (0.90) | -0.8 (0.93)
  Loss of Weight: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Loss of Weight: CFB at Day 7 | -0.7 (0.87) | -0.7 (0.94)
  Loss of Weight: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Loss of Weight: CFB at Day 8 | -0.6 (0.94) | -0.8 (0.91)
  Loss of Weight: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Loss of Weight: CFB at Day 15 | -0.7 (0.93) | -0.8 (0.88)
  Loss of Weight: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Loss of Weight: CFB at Day 21 | -0.7 (0.93) | -0.9 (0.88)
  Loss of Weight: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Loss of Weight: CFB at Day 28 | -0.6 (0.97) | -1.0 (0.88)
  Loss of Weight: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Loss of Weight: CFB at Day 35 | -0.7 (0.97) | -0.9 (0.90)
  Loss of Weight: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Loss of Weight: CFB at Day 42 | -0.6 (0.88) | -0.9 (0.95)
  Somatic Symptoms General: Baseline | 1.7 (0.50) | 1.7 (0.46)
  Somatic Symptoms General: CFB at Day 2 | -0.1 (0.55) | -0.3 (0.60)
  Somatic Symptoms General: CFB at Day 3 | -0.3 (0.47) | -0.4 (0.66)
  Somatic Symptoms General: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Somatic Symptoms General: CFB at Day 4 | -0.5 (0.74) | -0.5 (0.73)
  Somatic Symptoms General: CFB at Day 5 | -0.5 (0.85) | -0.5 (0.89)
  Somatic Symptoms General: CFB at Day 6 | -0.6 (0.70) | -0.7 (0.89)
  Somatic Symptoms General: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Somatic Symptoms General: CFB at Day 7 | -0.6 (0.72) | -0.9 (0.76)
  Somatic Symptoms General: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Somatic Symptoms General: CFB at Day 8 | -0.6 (0.79) | -0.8 (0.86)
  Somatic Symptoms General: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Somatic Symptoms General: CFB at Day 15 | -0.7 (0.91) | -1.1 (0.78)
  Somatic Symptoms General: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Somatic Symptoms General: CFB at Day 21 | -0.8 (0.88) | -1.0 (0.90)
  Somatic Symptoms General: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Somatic Symptoms General: CFB at Day 28 | -0.8 (0.96) | -0.9 (0.87)
  Somatic Symptoms General: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Somatic Symptoms General: CFB at Day 35 | -0.9 (0.94) | -1.0 (0.89)
  Somatic Symptoms General: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Somatic Symptoms General: CFB at Day 42 | -0.8 (0.92) | -0.9 (0.89)
  Feelings of Guilt: Baseline | 2.1 (0.70) | 1.9 (0.83)
  Feelings of Guilt: CFB at Day 2 | -0.3 (0.69) | -0.4 (0.68)
  Feelings of Guilt: CFB at Day 3 | -0.5 (0.73) | -0.5 (0.82)
  Feelings of Guilt: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Feelings of Guilt: CFB at Day 4 | -0.6 (0.87) | -0.7 (0.84)
  Feelings of Guilt: CFB at Day 5 | -0.7 (0.76) | -1.0 (0.93)
  Feelings of Guilt: CFB at Day 6 | -0.8 (0.97) | -1.2 (0.96)
  Feelings of Guilt: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Feelings of Guilt: CFB at Day 7 | -0.9 (0.99) | -1.2 (1.04)
  Feelings of Guilt: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Feelings of Guilt: CFB at Day 8 | -1.2 (0.91) | -1.2 (1.12)
  Feelings of Guilt: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Feelings of Guilt: CFB at Day 15 | -1.0 (1.15) | -1.4 (1.01)
  Feelings of Guilt: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Feelings of Guilt: CFB at Day 21 | -1.1 (1.04) | -1.2 (1.12)
  Feelings of Guilt: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Feelings of Guilt: CFB at Day 28 | -1.0 (1.03) | -1.3 (1.05)
  Feelings of Guilt: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Feelings of Guilt: CFB at Day 35 | -1.2 (1.00) | -1.1 (1.14)
  Feelings of Guilt: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Feelings of Guilt: CFB at Day 42 | -1.3 (0.95) | -1.2 (1.09)
  Suicide: Baseline | 0.3 (0.51) | 0.1 (0.29)
  Suicide: CFB at Day 2 | -0.2 (0.46) | 0.0 (0.15)
  Suicide: CFB at Day 3 | -0.2 (0.46) | 0.0 (0.15)
  Suicide: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Suicide: CFB at Day 4 | -0.2 (0.45) | 0.0 (0.21)
  Suicide: CFB at Day 5 | -0.2 (0.45) | 0.0 (0.26)
  Suicide: CFB at Day 6 | -0.2 (0.48) | 0.0 (0.21)
  Suicide: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Suicide: CFB at Day 7 | -0.2 (0.48) | -0.1 (0.25)
  Suicide: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Suicide: CFB at Day 8 | -0.2 (0.51) | -0.1 (0.29)
  Suicide: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Suicide: CFB at Day 15 | -0.2 (0.52) | -0.1 (0.30)
  Suicide: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Suicide: CFB at Day 21 | -0.2 (0.54) | -0.1 (0.30)
  Suicide: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Suicide: CFB at Day 28 | -0.2 (0.52) | -0.1 (0.30)
  Suicide: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Suicide: CFB at Day 35 | -0.2 (0.52) | -0.1 (0.26)
  Suicide: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Suicide: CFB at Day 42 | -0.2 (0.52) | -0.1 (0.30)
  Anxiety Psychic: Baseline | 2.3 (0.67) | 2.1 (0.49)
  Anxiety Psychic: CFB at Day 2 | -0.3 (0.78) | -0.4 (0.75)
  Anxiety Psychic: CFB at Day 3 | -0.5 (0.66) | -0.8 (0.94)
  Anxiety Psychic: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Anxiety Psychic: CFB at Day 4 | -0.7 (1.05) | -1.0 (1.16)
  Anxiety Psychic: CFB at Day 5 | -0.8 (1.05) | -1.1 (0.98)
  Anxiety Psychic: CFB at Day 6 | -0.8 (0.91) | -1.2 (1.13)
  Anxiety Psychic: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Anxiety Psychic: CFB at Day 7 | -0.9 (1.01) | -1.1 (1.25)
  Anxiety Psychic: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Anxiety Psychic: CFB at Day 8 | -1.1 (0.97) | -1.2 (1.01)
  Anxiety Psychic: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Anxiety Psychic: CFB at Day 15 | -0.9 (0.93) | -1.5 (0.86)
  Anxiety Psychic: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Anxiety Psychic: CFB at Day 21 | -1.0 (0.90) | -1.4 (0.97)
  Anxiety Psychic: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Anxiety Psychic: CFB at Day 28 | -1.0 (1.00) | -1.2 (0.92)
  Anxiety Psychic: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Anxiety Psychic: CFB at Day 35 | -0.9 (1.13) | -1.1 (1.04)
  Anxiety Psychic: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Anxiety Psychic: CFB at Day 42 | -0.9 (1.08) | -1.2 (0.83)
  Anxiety Somatic: Baseline | 1.4 (0.78) | 1.4 (0.75)
  Anxiety Somatic: CFB at Day 2 | -0.3 (0.61) | -0.4 (0.81)
  Anxiety Somatic: CFB at Day 3 | -0.4 (0.75) | -0.6 (0.84)
  Anxiety Somatic: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Anxiety Somatic: CFB at Day 4 | -0.5 (0.88) | -0.5 (0.84)
  Anxiety Somatic: CFB at Day 5 | -0.4 (0.87) | -0.6 (0.81)
  Anxiety Somatic: CFB at Day 6 | -0.4 (0.87) | -0.6 (0.69)
  Anxiety Somatic: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Anxiety Somatic: CFB at Day 7 | -0.4 (0.91) | -0.5 (0.87)
  Anxiety Somatic: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Anxiety Somatic: CFB at Day 8 | -0.6 (0.99) | -0.7 (0.87)
  Anxiety Somatic: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Anxiety Somatic: CFB at Day 15 | -0.6 (0.80) | -0.8 (0.83)
  Anxiety Somatic: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Anxiety Somatic: CFB at Day 21 | -0.7 (0.92) | -0.8 (0.87)
  Anxiety Somatic: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Anxiety Somatic: CFB at Day 28 | -0.7 (0.90) | -0.7 (0.94)
  Anxiety Somatic: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Anxiety Somatic: CFB at Day 35 | -0.8 (0.80) | -0.8 (0.86)
  Anxiety Somatic: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Anxiety Somatic: CFB at Day 42 | -0.6 (1.02) | -0.8 (0.85)
  Hypochondriasis: Baseline | 1.1 (0.85) | 1.0 (0.83)
  Hypochondriasis: CFB at Day 2 | -0.2 (0.76) | -0.2 (0.67)
  Hypochondriasis: CFB at Day 3 | -0.3 (0.74) | -0.3 (0.84)
  Hypochondriasis: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Hypochondriasis: CFB at Day 4 | -0.5 (0.83) | -0.5 (0.82)
  Hypochondriasis: CFB at Day 5 | -0.5 (0.90) | -0.6 (0.78)
  Hypochondriasis: CFB at Day 6 | -0.5 (1.02) | -0.6 (0.80)
  Hypochondriasis: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Hypochondriasis: CFB at Day 7 | -0.5 (1.03) | -0.5 (0.84)
  Hypochondriasis: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Hypochondriasis: CFB at Day 8 | -0.5 (1.02) | -0.6 (0.87)
  Hypochondriasis: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Hypochondriasis: CFB at Day 15 | -0.5 (0.77) | -0.7 (0.91)
  Hypochondriasis: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Hypochondriasis: CFB at Day 21 | -0.5 (0.73) | -0.7 (0.81)
  Hypochondriasis: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Hypochondriasis: CFB at Day 28 | -0.5 (0.91) | -0.7 (0.92)
  Hypochondriasis: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Hypochondriasis: CFB at Day 35 | -0.6 (0.87) | -0.7 (0.94)
  Hypochondriasis: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Hypochondriasis: CFB at Day 42 | -0.6 (0.96) | -0.7 (0.92)
  Insight: Baseline | 0.1 (0.25) | 0.1 (0.25)
  Insight: CFB at Day 2 | 0.0 (0.15) | 0.0 (0.21)
  Insight: CFB at Day 3 | 0.0 (0.21) | 0.0 (0.26)
  Insight: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Insight: CFB at Day 4 | 0.0 (0.21) | 0.0 (0.26)
  Insight: CFB at Day 5 | 0.0 (0.21) | 0.0 (0.26)
  Insight: CFB at Day 6 | 0.0 (0.21) | 0.0 (0.26)
  Insight: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Insight: CFB at Day 7 | 0.0 (0.21) | 0.0 (0.26)
  Insight: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Insight: CFB at Day 8 | 0.0 (0.22) | 0.0 (0.26)
  Insight: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Insight: CFB at Day 15 | 0.0 (0.22) | 0.0 (0.22)
  Insight: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Insight: CFB at Day 21 | -0.1 (0.23) | 0.0 (0.22)
  Insight: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Insight: CFB at Day 28 | -0.1 (0.22) | 0.0 (0.15)
  Insight: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Insight: CFB at Day 35 | -0.1 (0.22) | 0.0 (0.16)
  Insight: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Insight: CFB at Day 42 | -0.1 (0.22) | 0.0 (0.22)
  Agitation: Baseline | 0.8 (0.88) | 0.5 (0.63)
  Agitation: CFB at Day 2 | -0.2 (0.73) | 0.0 (0.52)
  Agitation: CFB at Day 3 | -0.2 (0.87) | -0.2 (0.53)
  Agitation: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Agitation: CFB at Day 4 | -0.2 (0.97) | -0.2 (0.53)
  Agitation: CFB at Day 5 | -0.4 (0.76) | -0.2 (0.61)
  Agitation: CFB at Day 6 | -0.3 (0.87) | -0.3 (0.60)
  Agitation: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Agitation: CFB at Day 7 | -0.3 (0.86) | -0.3 (0.60)
  Agitation: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Agitation: CFB at Day 8 | -0.5 (0.92) | -0.3 (0.64)
  Agitation: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Agitation: CFB at Day 15 | -0.4 (0.99) | -0.4 (0.66)
  Agitation: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Agitation: CFB at Day 21 | -0.4 (0.79) | -0.3 (0.65)
  Agitation: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Agitation: CFB at Day 28 | -0.6 (1.04) | -0.4 (0.59)
  Agitation: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Agitation: CFB at Day 35 | -0.6 (0.96) | -0.4 (0.63)
  Agitation: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Agitation: CFB at Day 42 | -0.6 (0.88) | -0.3 (0.68)
  Retardation: Baseline | 0.8 (0.89) | 1.2 (0.97)
  Retardation: CFB at Day 2 | -0.1 (0.63) | -0.2 (0.83)
  Retardation: CFB at Day 3 | -0.2 (0.67) | -0.5 (0.87)
  Retardation: CFB at Day 4: number analyzed (Participants) | 43 | 45
  Retardation: CFB at Day 4 | -0.3 (0.85) | -0.7 (0.95)
  Retardation: CFB at Day 5 | -0.3 (0.82) | -0.8 (0.96)
  Retardation: CFB at Day 6 | -0.3 (0.86) | -0.9 (0.99)
  Retardation: CFB at Day 7: number analyzed (Participants) | 43 | 45
  Retardation: CFB at Day 7 | -0.4 (0.88) | -0.8 (0.90)
  Retardation: CFB at Day 8: number analyzed (Participants) | 42 | 44
  Retardation: CFB at Day 8 | -0.4 (0.93) | -0.8 (0.93)
  Retardation: CFB at Day 15: number analyzed (Participants) | 42 | 42
  Retardation: CFB at Day 15 | -0.4 (0.96) | -1.0 (0.91)
  Retardation: CFB at Day 21: number analyzed (Participants) | 38 | 42
  Retardation: CFB at Day 21 | -0.4 (0.86) | -1.1 (0.93)
  Retardation: CFB at Day 28: number analyzed (Participants) | 39 | 42
  Retardation: CFB at Day 28 | -0.4 (0.75) | -1.0 (1.02)
  Retardation: CFB at Day 35: number analyzed (Participants) | 40 | 41
  Retardation: CFB at Day 35 | -0.5 (0.85) | -1.0 (0.94)
  Retardation: CFB at Day 42: number analyzed (Participants) | 39 | 42
  Retardation: CFB at Day 42 | -0.5 (0.79) | -0.9 (0.99)

125. Secondary Outcome: Change From Baseline in HAM-A Total Score at Day 15 and All Other Time Points - Part B
Description: The 14-item HAM-A was used to rate the severity of symptoms of anxiety. Each of the 14 items was defined by a series of symptoms, and measured both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Scoring for HAM-A was calculated by assigning scores of 0 (not present) to 4 (very severe), with a total score range of 0 to 56, where 0-13=Normal, 14-17 Mild Anxiety, 18-24 Moderate Anxiety, >=25 Severe Anxiety, per the Psych Congress Network. The HAM-A total score was calculated as the sum of the 14 individual item scores. A negative change from baseline indicated less anxiety. A positive change from baseline indicated more anxiety. The analysis was performed in participants included in Part B of the study.
Time Frame: Baseline, Days 2, 8, 15, 21, 28, 35 and 42
Population: as for outcome 52
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
score on a scale
  Change from Baseline at Day 2 | -3.7 (0.86) | -5.5 (0.83)
  Change from Baseline at Day 8 | -8.9 (1.09) | -11.4 (1.06)
  Change from Baseline at Day 15 | -8.6 (1.11) | -13.2 (1.08)
  Change from Baseline at Day 21 | -9.5 (1.25) | -12.9 (1.21)
  Change from Baseline at Day 28 | -10.0 (1.26) | -12.2 (1.22)
  Change from Baseline at Day 35 | -9.9 (1.38) | -12.0 (1.35)
  Change from Baseline at Day 42 | -9.6 (1.39) | -11.8 (1.35)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 2; Test type: Superiority; p = 0.0391, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-A total score at each visit as the dependent variable; Least Squares Mean Difference = -1.8, 95% CI 2-sided [-3.6 to -0.1], Standard Error of Mean 0.87
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 8; Test type: Superiority; p = 0.0516, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-A total score at each visit as the dependent variable; Least Squares Mean Difference = -2.5, 95% CI 2-sided [-5.1 to 0.0], Standard Error of Mean 1.29
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 15; Test type: Superiority; p = 0.0008, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-A total score at each visit as the dependent variable; Least Squares Mean Difference = -4.6, 95% CI 2-sided [-7.3 to -2.0], Standard Error of Mean 1.32
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 21; Test type: Superiority; p = 0.0282, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-A total score at each visit as the dependent variable; Least Squares Mean Difference = -3.4, 95% CI 2-sided [-6.5 to -0.4], Standard Error of Mean 1.54
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 28; Test type: Superiority; p = 0.1686, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-A total score at each visit as the dependent variable; Least Squares Mean Difference = -2.2, 95% CI 2-sided [-5.3 to 0.9], Standard Error of Mean 1.56
Statistical Analysis 6: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 35; Test type: Superiority; p = 0.2488, Mixed Effect Model for Repeated Measures; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-5.5 to 1.5], Standard Error of Mean 1.75
Statistical Analysis 7: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 42; Test type: Superiority; p = 0.2037, Mixed Effect Model for Repeated Measures; The MMRM included the change from baseline in HAM-A total score at each visit as the dependent variable; Least Squares Mean Difference = -2.3, 95% CI 2-sided [-5.7 to 1.2], Standard Error of Mean 1.76

126. Secondary Outcome: Percentage of Participants With CGI-I Response - Part B
Description: The CGI-I item employed a 7-point Likert scale to measure the overall improvement in the participant's condition post-treatment. The investigator rated the participant's total improvement whether or not it was due entirely to drug treatment. Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. The CGI-I was only rated at post-treatment assessments. By definition, all CGI-I assessments were evaluated against baseline conditions. CGI-I response was defined as having a score of 1 (very much improved) or 2 (much improved). The analysis was performed in participants included in Part B of the study. Data is reported for participants who had CGI-I response.
Time Frame: Days 2, 8, 15, 21, 28, 35 and 42
Population: as for outcome 121
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Placebo | Part B: SAGE-217
Number analyzed (Participants) | 44 | 45
percentage of participants
  Day 2 | 0 | 15.6
  Day 8: number analyzed (Participants) | 42 | 44
  Day 8 | 45.2 | 70.5
  Day 15: number analyzed (Participants) | 42 | 42
  Day 15 | 45.2 | 78.6
  Day 21: number analyzed (Participants) | 38 | 42
  Day 21 | 50.0 | 71.4
  Day 28: number analyzed (Participants) | 39 | 42
  Day 28 | 46.2 | 66.7
  Day 35: number analyzed (Participants) | 40 | 41
  Day 35 | 55.0 | 63.4
  Day 42: number analyzed (Participants) | 39 | 42
  Day 42 | 59.0 | 69.0
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 8; Test type: Superiority; p = 0.0048, Generalized Estimating Equation; Statistics are from a GEE method including the CGI-I response at each visit as the dependent variable; Odds Ratio (OR) = 5.5, 95% CI 2-sided [1.7 to 17.9] — For the model parameters estimation, the exchangeable working correlation structure was used
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 15; Test type: Superiority; p = 0.0007, Generalized Estimating Equation; Statistics are from a GEE method including the CGI-I response at each visit as the dependent variable; Odds Ratio (OR) = 8.6, 95% CI 2-sided [2.5 to 29.5] — For the model parameters estimation, the exchangeable working correlation structure was used
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 21; Test type: Superiority; p = 0.0113, Generalized Estimating Equation; Statistics are from a GEE method including the CGI-I response at each visit as the dependent variable; Odds Ratio (OR) = 4.4, 95% CI 2-sided [1.4 to 13.6] — For the model parameters estimation, the exchangeable working correlation structure was used
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 28; Test type: Superiority; p = 0.0227, Generalized Estimating Equation; Statistics are from a GEE method including the CGI-I response at each visit as the dependent variable; Odds Ratio (OR) = 3.9, 95% CI 2-sided [1.2 to 12.8] — For the model parameters estimation, the exchangeable working correlation structure was used
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 35; Test type: Superiority; p = 0.1516, Generalized Estimating Equation; Statistics are from a GEE method including the CGI-I response at each visit as the dependent variable; Odds Ratio (OR) = 2.3, 95% CI 2-sided [0.7 to 7.2] — For the model parameters estimation, the exchangeable working correlation structure was used
Statistical Analysis 6: Comparison: Part B: Placebo vs Part B: SAGE-217; Day 42; Test type: Superiority; p = 0.0793, Generalized Estimating Equation; Statistics are from a GEE method including the CGI-I response at each visit as the dependent variable; Odds Ratio (OR) = 2.7, 95% CI 2-sided [0.9 to 8.3] — For the model parameters estimation, the exchangeable working correlation structure was used

ADVERSE EVENTS:
Time Frame: Part A: Up to Day 21; Part B: Up to Day 21 and from Day 21 up to Day 42
Description: AEs included TEAEs and AEs that occurred during post-TEAE period. TEAE was defined as adverse event with onset after the start of study drug, or any worsening of a pre-existing medical condition/adverse event with onset after the start of study drug and until 7 days after the last dose. Post-TEAE period was defined as 7 days after final study drug dose through last follow-up. The safety set included all participants who received at least one dose of the study drug.
Arm/Group | Part A: SAGE-217 | Part B: Placebo | Part B: SAGE-217
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/44 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/44 | 0/45
Other Adverse Events (participants affected / at risk) | 12/13 | 12/44 | 15/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: SAGE-217 (N=13) | Part B: Placebo (N=44) | Part B: SAGE-217 (N=45)
Sedation (Nervous system disorders) | 6 | 2 | 2
Headache (Nervous system disorders) | 4 | 8 | 9
Somnolence (Nervous system disorders) | 3 | 1 | 3
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 0
Fatigue (General disorders) | 1 | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Euphoric mood (Psychiatric disorders) | 1 | 0 | 1
Libido increased (Psychiatric disorders) | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 3 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Hot flush (Vascular disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3 | 5
Chromaturia (Renal and urinary disorders) | 0 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2017-01-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT03000530/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT03000530/SAP_001.pdf